CLINICAL TRIAL: NCT01675427
Title: An International, Multi-Center Study Evaluating the Correlation of IL28B Genotypes With Patient Demographics and Disease Characteristics in Patients With Chronic Hepatitis C
Brief Title: A Study on the Correlation Between Interleukin 28B Genotypes With Clinical and Demographic Characteristics in Treatment-Naïve and Treatment-Experienced Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MV25600
Record Dates: First submitted 2012-08-24; First posted 2012-08-30 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (1):
- Chronic hepatitis C patients (Experimental)
  Interventions: Other: Interleukin 28B testing

INTERVENTIONS:
Other: Interleukin 28B testing — Blood sampling for ILB28 genotyping

SUMMARY:
This multicenter study will evaluate the correlation of interleukin 28B (IL28B) genotypes with disease characteristics and demographics in treatment-naïve and treatment-experienced chronic hepatitis C patients, including patients with HIV co-infection. There will be a single study visit for testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult (according to local legislation) male or female patient
* Chronic hepatitis C (CHC)
* Patients naïve to CHC treatment or patients who received prior interferon-based therapy for CHC for whom data on treatment received and treatment outcome is available; information on fibrosis stage prior to previous treatment is also required

Exclusion Criteria:

* Co-infection with hepatitis B
* History or evidence of decompensated liver disease
* History of major organ transplantation with an existing functional graft (including liver transplantation)
* End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4766 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (164):
- Alexandria, Virginia, United States
- Argentina (2):
  - Buenos Aires
  - Mar del Plata
- Belgium (13):
  - Antwerp
  - Bruges
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Hasselt
  - Heusy
  - Kortrijk
  - Leuven
  - Liège
  - Ostend
  - Roeselare
- Santiago, Chile
- Egypt (4):
  - Cairo
  - Giza
  - Menoufiya
  - Tanta
- Estonia (4):
  - Kohtla-Järve
  - Pärnu
  - Tallinn
  - Tartu
- France (14):
  - Avignon
  - Châteauroux
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Rouen
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (15):
  - Aachen
  - Berlin
  - Burghausen
  - Cologne
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt (Oder)
  - Kassel
  - Lübeck
  - Magdeburg
  - Mannheim
  - Rostock
  - Rottenburg
  - Tübingen
- Greece (7):
  - Alexandroupoli
  - Athens
  - Ioannina
  - Larissa
  - Nea Kifissia
  - Pátrai
  - Thessaloniki
- Italy (34):
  - Chieti, Abruzzo
  - Bari, Apulia
  - Bisceglie, Apulia
  - Castellana Grotte, Apulia
  - San Giovanni Rotondo, Apulia
  - Reggio Calabria, Calabria
  - Avellino, Campania
  - Gragnano, Campania
  - Marcianise, Campania
  - Napoli, Campania
  - Nocera Inferiore, Campania
  - Nola, Campania
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Savona, Liguria
  - Milan, Lombardy
  - Biella, Piedmont
  - Cuorgnè (TO), Piedmont
  - Omegna (VB), Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Torrette Di Ancona, The Marches
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Livorno, Tuscany
  - Padua, Veneto
- Safat, Kuwait
- Riga, Latvia
- Lebanon (4):
  - Baabda
  - Beirut
  - Nabatieh
  - Tripoli
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Mexico (3):
  - Culiacán
  - Mexico City
  - Tijuana
- Skopje, North Macedonia
- Muscat, Oman
- Pakistan (5):
  - Faisalabad
  - Gujranwala
  - Karachi
  - Lahore
  - Rawalpindi
- Peru (2):
  - La Victoria, Lima
  - Lima
- Portugal (6):
  - Almada
  - Amadora
  - Aveiro
  - Faro
  - Lisbon
  - Porto
- Doha, Qatar
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Iași
  - Timișoara
- Serbia (2):
  - Belgrade
  - Novi Sad
- Slovakia (4):
  - Banská Bystrica
  - Bratislava
  - Martin
  - Prešov
- Sweden (3):
  - Gävle
  - Karlstad
  - Uppsala
- Switzerland (2):
  - Lugano
  - Sankt Gallen
- Aleppo, Syria
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (14):
  - Adana
  - Adapazarı
  - Ankara
  - Eskişehir
  - Hatay
  - Istanbul
  - ISTANBULt
  - Izmir
  - Kayseri
  - Mersin
  - Samsun
  - Tokat Province
  - Trabzon
  - Zonguldak
- United Arab Emirates (2):
  - Dubai
  - Sharjah city
- Venezuela (2):
  - Caracas
  - Maracaibo

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Chronic Hepatitis C (CHC): Both treatment-naive and treatment-experienced participants with CHC were enrolled in this prospective, interventional Phase 4 study.
Period: Overall Study
Arm/Group | Participants With Chronic Hepatitis C (CHC)
Started | 4766
Completed | 4732
Not Completed | 34
Not completed — Withdrawal by Subject | 7
Not completed — Participant Refused Sample Collection | 18
Not completed — Sample not Collected by Mistake | 2
Not completed — Lost to Follow-up | 5
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Core Analysis Population: All participants enrolled who had a blood sample drawn for genotyping with available data for the primary variables, and who met all eligibility criteria for analysis.
Groups:
- Participants With CHC: Both treatment-naive and treatment-experienced participants with CHC were enrolled in this prospective, interventional Phase 4 study.
Arm/Group | Participants With CHC
Number analyzed (Participants) | 4616
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2043
  Male | 2573

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Interleukin 28B (IL28B) Genotype rs12979860 by Cirrhosis Status and Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype (Genotype 1 [G1], Genotype 2 [G2], Genotype 3 [G3], Genotype 4 [G4], and all other genotypes [Other]) and cirrhosis status ('Cirrhosis/transition to cirrhosis' or 'No cirrhosis') were obtained from medical records. Cirrhosis status was based upon previous biopsy or noninvasive assessment captured prior to treatment, if applicable.
Time Frame: Study Visit 1 (single study visit)
Population: Core Analysis Population (Treatment-Naive): Only participants who had not received prior treatment for CHC were included in the analysis; n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: IL28B rs12979860 Cysteine-Cysteine (CC): Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'CC' confirmed by blood sampling.
- Naive: IL28B rs12979860 Threonine-Cysteine (TC): Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'TC' confirmed by blood sampling.
- Naive: IL28B rs12979860 Threonine-Threonine (TT): Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'TT' confirmed by blood sampling.
Arm/Group | Naive: IL28B rs12979860 Cysteine-Cysteine (CC) | Naive: IL28B rs12979860 Threonine-Cysteine (TC) | Naive: IL28B rs12979860 Threonine-Threonine (TT)
Number analyzed (Participants) | 976 | 1511 | 415
participants
  G1, Cirrhosis (n=499,928,269) | 111 | 255 | 87
  G1, No cirrhosis (n=499,928,269) | 388 | 673 | 182
  G2, Cirrhosis (n=126,157,37) | 23 | 27 | 3
  G2, No cirrhosis (n=126,157,37) | 103 | 130 | 34
  G3, Cirrhosis (n=231,276,65) | 76 | 67 | 18
  G3, No cirrhosis (n=231,276,65) | 155 | 209 | 47
  G4, Cirrhosis (n=92,129,38) | 29 | 35 | 10
  G4, No cirrhosis (n=92,129,38) | 63 | 94 | 28
  Other, Cirrhosis (n=28,21,6) | 9 | 6 | 1
  Other, No cirrhosis (n=28,21,6) | 19 | 15 | 5
  Total, Cirrhosis (n=976,1511,415) | 248 | 390 | 119
  Total, No cirrhosis (n=976,1511,415) | 728 | 1121 | 296
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); G1; Test type: Superiority or Other; p = 0.0018, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); G2; Test type: Superiority or Other; p = 0.2289, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); G3; Test type: Superiority or Other; p = 0.1112, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); G4; Test type: Superiority or Other; p = 0.4681, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); Other genotypes; Test type: Superiority or Other; p = 0.4828, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 Cysteine-Cysteine (CC) vs Naive: IL28B rs12979860 Threonine-Cysteine (TC) vs Naive: IL28B rs12979860 Threonine-Threonine (TT); Total genotypes; Test type: Superiority or Other; p = 0.2702, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

2. Primary Outcome: Number of Participants With IL28B Genotype rs12979860 by Cirrhosis Status and HCV RNA Genotype: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and cirrhosis status were obtained from medical records. Cirrhosis status was based upon previous biopsy or noninvasive assessment captured prior to treatment, if applicable.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced): Only participants who had received prior treatment for CHC were included in the analysis; n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Experienced: IL28B rs12979860 CC: Treatment-experienced participants with CHC with IL28B polymorphism rs12979860 'CC' confirmed by blood sampling.
- Experienced: IL28B rs12979860 TC: Treatment-experienced participants with CHC with IL28B polymorphism rs12979860 'TC' confirmed by blood sampling.
- Experienced: IL28B rs12979860 TT: Treatment-experienced participants with CHC with IL28B polymorphism rs12979860 'TT' confirmed by blood sampling.
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 462 | 850 | 275
participants
  G1, Cirrhosis (n=281,653,226) | 93 | 208 | 67
  G1, No cirrhosis (n=281,653,226) | 188 | 445 | 159
  G2, Cirrhosis (n=89,36,9) | 30 | 8 | 3
  G2, No cirrhosis (n=89,36,9) | 59 | 28 | 6
  G3, Cirrhosis (n=55,75,19) | 19 | 26 | 6
  G3, No cirrhosis (n=55,75,19) | 36 | 49 | 13
  G4, Cirrhosis (n=25,66,19) | 4 | 15 | 5
  G4, No cirrhosis (n=25,66,19) | 21 | 51 | 14
  Other, Cirrhosis (n=12,20,2) | 6 | 7 | 0
  Other, No cirrhosis (n=12,20,2) | 6 | 13 | 2
  Total, Cirrhosis (n=462,850,275) | 152 | 264 | 81
  Total, No cirrhosis (n=462,850,275) | 310 | 586 | 194
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.4133, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.4400, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.8597, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.3975, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.1781, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.3159, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

3. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by Cirrhosis Status and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 2
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: IL28B rs8099917 TT: Treatment-naive participants with CHC with IL28B rs8099917 polymorphism 'TT' confirmed by blood sampling.
- Naive: IL28B rs8099917 Threonine-Glycine (TG): Treatment-naive participants with CHC with IL28B rs8099917 polymorphism 'TG' confirmed by blood sampling.
- Naive: IL28B rs8099917 Glycine-Glycine (GG): Treatment-naive participants with CHC with IL28B rs8099917 polymorphism 'GG' confirmed by blood sampling.
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 Threonine-Glycine (TG) | Naive: IL28B rs8099917 Glycine-Glycine (GG)
Number analyzed (Participants) | 1593 | 1141 | 168
participants
  G1, Cirrhosis (n=835,745,116) | 200 | 217 | 36
  G1, No cirrhosis (n=835,745,116) | 635 | 528 | 80
  G2, Cirrhosis (n=197,111,12) | 33 | 19 | 1
  G2, No cirrhosis (n=197,111,12) | 164 | 92 | 11
  G3, Cirrhosis (n=360,185,27) | 111 | 42 | 8
  G3, No cirrhosis (n=360,185,27) | 249 | 143 | 19
  G4, Cirrhosis (n=164,85,10) | 45 | 26 | 3
  G4, No cirrhosis (n=164,85,10) | 119 | 59 | 7
  Other, Cirrhosis (n=37,15,3) | 11 | 5 | 0
  Other, No cirrhosis (n=37,15,3) | 26 | 10 | 3
  Total, Cirrhosis (n=1593,1141,168) | 400 | 309 | 48
  Total, No cirrhosis (n=1593,1141,168) | 1193 | 832 | 120
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); G1; Test type: Superiority or Other; p = 0.0126, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); G2; Test type: Superiority or Other; p = 0.7174, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); G3; Test type: Superiority or Other; p = 0.1380, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); G4; Test type: Superiority or Other; p = 0.6258, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); Other genotypes; Test type: Superiority or Other; p = 0.5751, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 Threonine-Glycine (TG) vs Naive: IL28B rs8099917 Glycine-Glycine (GG); Total genotypes; Test type: Superiority or Other; p = 0.1681, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

4. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by Cirrhosis Status and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 2
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Experienced: IL28B rs8099917 TT: Treatment-experienced participants with CHC with IL28B rs8099917 polymorphism 'TT' confirmed by blood sampling.
- Experienced: IL28B rs8099917 TG: Treatment-experienced participants with CHC with IL28B rs8099917 polymorphism 'TG' confirmed by blood sampling.
- Experienced: IL28B rs8099917 GG: Treatment-experienced participants with CHC with IL28B rs8099917 polymorphism 'GG' confirmed by blood sampling.
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 796 | 682 | 109
participants
  G1, Cirrhosis (n=528,539,93) | 158 | 179 | 31
  G1, No cirrhosis (n=528,539,93) | 370 | 360 | 62
  G2, Cirrhosis (n=102,25,7) | 35 | 3 | 3
  G2, No cirrhosis (n=102,25,7) | 67 | 22 | 4
  G3, Cirrhosis (n=81,59,9) | 29 | 19 | 3
  G3, No cirrhosis (n=81,59,9) | 52 | 40 | 6
  G4, Cirrhosis (n=70,40,0) | 11 | 13 | 0
  G4, No cirrhosis (n=70,40,0) | 59 | 27 | 0
  Other, Cirrhosis (n=15,19,0) | 8 | 5 | 0
  Other, No cirrhosis (n=15,19,0) | 7 | 14 | 0
  Total, Cirrhosis (n=796,682,109) | 241 | 219 | 37
  Total, No cirrhosis (n=796,682,109) | 555 | 463 | 72
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.2693, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.3240, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.7006, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.0403, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.1075, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.3295, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

5. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by METAVIR Liver Inflammation Grade and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and liver inflammation grade (Grade A0, Grade A1, Grade A2, or Grade A3) were obtained from medical records. Liver inflammation grade was based upon previous biopsy using the METAVIR scoring system and captured prior to treatment, if applicable.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: IL28B rs12979860 CC: Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'CC' confirmed by blood sampling.
- Naive: IL28B rs12979860 TC: Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'TC' confirmed by blood sampling.
- Naive: IL28B rs12979860 TT: Treatment-naive participants with CHC with IL28B polymorphism rs12979860 'TT' confirmed by blood sampling.
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 127 | 184 | 61
participants
  G1, Grade A0 (n=76,132,46) | 1 | 4 | 2
  G1, Grade A1 (n=76,132,46) | 38 | 54 | 24
  G1, Grade A2 (n=76,132,46) | 27 | 57 | 11
  G1, Grade A3 (n=76,132,46) | 10 | 17 | 9
  G2, Grade A0 (n=8,4,0) | 0 | 1 | 0
  G2, Grade A1 (n=8,4,0) | 4 | 1 | 0
  G2, Grade A2 (n=8,4,0) | 4 | 2 | 0
  G2, Grade A3 (n=8,4,0) | 0 | 0 | 0
  G3, Grade A0 (n=18,14,5) | 1 | 1 | 0
  G3, Grade A1 (n=18,14,5) | 6 | 7 | 4
  G3, Grade A2 (n=18,14,5) | 7 | 5 | 1
  G3, Grade A3 (n=18,14,5) | 4 | 1 | 0
  G4, Grade A0 (n=21,34,8) | 0 | 5 | 1
  G4, Grade A1 (n=21,34,8) | 13 | 22 | 6
  G4, Grade A2 (n=21,34,8) | 7 | 3 | 0
  G4, Grade A3 (n=21,34,8) | 1 | 4 | 1
  Other, Grade A0 (n=4,0,2) | 0 | 0 | 0
  Other, Grade A1 (n=4,0,2) | 3 | 0 | 2
  Other, Grade A2 (n=4,0,2) | 1 | 0 | 0
  Other, Grade A3 (n=4,0,2) | 0 | 0 | 0
  Total, Grade A0 (n=127,184,61) | 2 | 11 | 3
  Total, Grade A1 (n=127,184,61) | 64 | 84 | 36
  Total, Grade A2 (n=127,184,61) | 46 | 67 | 12
  Total, Grade A3 (n=127,184,61) | 15 | 22 | 10
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.9859, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.7055, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0920, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0781, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.4795, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.3069, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

6. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by METAVIR Liver Inflammation Grade and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 5
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 149 | 249 | 73
participants
  G1, Grade A0 (n=102,203,60) | 3 | 5 | 2
  G1, Grade A1 (n=102,203,60) | 33 | 79 | 19
  G1, Grade A2 (n=102,203,60) | 48 | 90 | 32
  G1, Grade A3 (n=102,203,60) | 18 | 29 | 7
  G2, Grade A0 (n=28,7,1) | 0 | 1 | 0
  G2, Grade A1 (n=28,7,1) | 13 | 4 | 0
  G2, Grade A2 (n=28,7,1) | 15 | 2 | 1
  G2, Grade A3 (n=28,7,1) | 0 | 0 | 0
  G3, Grade A0 (n=11,7,4) | 1 | 0 | 0
  G3, Grade A1 (n=11,7,4) | 3 | 3 | 2
  G3, Grade A2 (n=11,7,4) | 6 | 3 | 2
  G3, Grade A3 (n=11,7,4) | 1 | 1 | 0
  G4, Grade A0 (n=5,29,8) | 0 | 0 | 0
  G4, Grade A1 (n=5,29,8) | 1 | 15 | 5
  G4, Grade A2 (n=5,29,8) | 3 | 10 | 3
  G4, Grade A3 (n=5,29,8) | 1 | 4 | 0
  Other, Grade A0 (n=3,3,0) | 0 | 0 | 0
  Other, Grade A1 (n=3,3,0) | 1 | 2 | 0
  Other, Grade A2 (n=3,3,0) | 0 | 1 | 0
  Other, Grade A3 (n=3,3,0) | 2 | 0 | 0
  Total, Grade A0 (n=149,249,73) | 4 | 6 | 2
  Total, Grade A1 (n=149,249,73) | 51 | 103 | 26
  Total, Grade A2 (n=149,249,73) | 72 | 106 | 38
  Total, Grade A3 (n=149,249,73) | 22 | 34 | 7
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.5216, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.3419, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.7586, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.1351, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.2386, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.3921, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

7. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by METAVIR Liver Inflammation Grade and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 5
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: IL28B rs8099917 TG: Treatment-naive participants with CHC with IL28B rs8099917 polymorphism 'TG' confirmed by blood sampling.
- Naive: IL28B rs8099917 GG: Treatment-naive participants with CHC with IL28B rs8099917 polymorphism 'GG' confirmed by blood sampling.
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 207 | 143 | 22
participants
  G1, Grade A0 (n=127,109,18) | 1 | 4 | 2
  G1, Grade A1 (n=127,109,18) | 63 | 45 | 8
  G1, Grade A2 (n=127,109,18) | 46 | 45 | 4
  G1, Grade A3 (n=127,109,18) | 17 | 15 | 4
  G2, Grade A0 (n=11,1,0) | 0 | 1 | 0
  G2, Grade A1 (n=11,1,0) | 5 | 0 | 0
  G2, Grade A2 (n=11,1,0) | 6 | 0 | 0
  G2, Grade A3 (n=11,1,0) | 0 | 0 | 0
  G3, Grade A0 (n=22,13,2) | 1 | 1 | 0
  G3, Grade A1 (n=22,13,2) | 9 | 6 | 2
  G3, Grade A2 (n=22,13,2) | 8 | 5 | 0
  G3, Grade A3 (n=22,13,2) | 4 | 1 | 0
  G4, Grade A0 (n=43,19,1) | 4 | 2 | 0
  G4, Grade A1 (n=43,19,1) | 29 | 12 | 0
  G4, Grade A2 (n=43,19,1) | 8 | 2 | 0
  G4, Grade A3 (n=43,19,1) | 2 | 3 | 1
  Other, Grade A0 (n=4,1,1) | 0 | 0 | 0
  Other, Grade A1 (n=4,1,1) | 3 | 1 | 1
  Other, Grade A2 (n=4,1,1) | 1 | 0 | 0
  Other, Grade A3 (n=4,1,1) | 0 | 0 | 0
  Total, Grade A0 (n=207,143,22) | 6 | 8 | 2
  Total, Grade A1 (n=207,143,22) | 109 | 64 | 11
  Total, Grade A2 (n=207,143,22) | 69 | 52 | 4
  Total, Grade A3 (n=207,143,22) | 23 | 19 | 5
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.8537, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0763, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.2432, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.4247, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.4884, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.6119, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

8. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by METAVIR Liver Inflammation Grade and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 5
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 235 | 205 | 31
participants
  G1, Grade A0 (n=160,177,28) | 4 | 5 | 1
  G1, Grade A1 (n=160,177,28) | 52 | 70 | 9
  G1, Grade A2 (n=160,177,28) | 77 | 79 | 14
  G1, Grade A3 (n=160,177,28) | 27 | 23 | 4
  G2, Grade A0 (n=30,5,1) | 0 | 1 | 0
  G2, Grade A1 (n=30,5,1) | 14 | 3 | 0
  G2, Grade A2 (n=30,5,1) | 16 | 1 | 1
  G2, Grade A3 (n=30,5,1) | 0 | 0 | 0
  G3, Grade A0 (n=14,6,2) | 1 | 0 | 0
  G3, Grade A1 (n=14,6,2) | 4 | 3 | 1
  G3, Grade A2 (n=14,6,2) | 7 | 3 | 1
  G3, Grade A3 (n=14,6,2) | 2 | 0 | 0
  G4, Grade A0 (n=28,14,0) | 0 | 0 | 0
  G4, Grade A1 (n=28,14,0) | 14 | 7 | 0
  G4, Grade A2 (n=28,14,0) | 10 | 6 | 0
  G4, Grade A3 (n=28,14,0) | 4 | 1 | 0
  Other, Grade A0 (n=3,3,0) | 0 | 0 | 0
  Other, Grade A1 (n=3,3,0) | 1 | 2 | 0
  Other, Grade A2 (n=3,3,0) | 0 | 1 | 0
  Other, Grade A3 (n=3,3,0) | 2 | 0 | 0
  Total, Grade A0 (n=235,205,31) | 5 | 6 | 1
  Total, Grade A1 (n=235,205,31) | 85 | 85 | 10
  Total, Grade A2 (n=235,205,31) | 110 | 90 | 16
  Total, Grade A3 (n=235,205,31) | 35 | 24 | 4
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.2416, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.2671, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.4619, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.8364, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.2386, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.2887, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

9. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Gender: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including gender, were obtained from medical records and/or participant interview at the Study Visit.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  Male | 582 | 802 | 224
  Female | 396 | 716 | 196
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.0049, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

10. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Gender: Treatment-Experienced
Description: as for outcome 9
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  Male | 287 | 509 | 169
  Female | 203 | 405 | 127
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.5651, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

11. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Gender: Treatment-Naive
Description: as for outcome 9
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1598 | 1147 | 171
participants
  Male | 910 | 608 | 90
  Female | 688 | 539 | 81
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.0420, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

12. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Gender: Treatment-Experienced
Description: as for outcome 9
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 851 | 730 | 119
participants
  Male | 489 | 412 | 64
  Female | 362 | 318 | 55
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.4545, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

13. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Ethnic Origin: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including self-reported ethnic origin, were obtained from medical records and/or participant interview at the Study Visit.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  Caucasian/white | 860 | 1349 | 373
  Black | 5 | 24 | 19
  Asian/Oriental | 89 | 83 | 9
  Native American/American Indian | 0 | 1 | 1
  Other | 24 | 61 | 18
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

14. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Ethnic Origin: Treatment-Experienced
Description: as for outcome 13
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  Caucasian/white | 314 | 807 | 259
  Black | 3 | 20 | 15
  Asian/Oriental | 161 | 42 | 5
  Native American/American Indian | 0 | 2 | 0
  Other | 12 | 43 | 17
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

15. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Ethnic Origin: Treatment-Naive
Description: as for outcome 13
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1598 | 1147 | 171
participants
  Caucasian/white | 1402 | 1030 | 150
  Black | 34 | 12 | 2
  Asian/Oriental | 123 | 53 | 5
  Native American/American Indian | 1 | 0 | 1
  Other | 38 | 52 | 13
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

16. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Ethnic Origin: Treatment-Experienced
Description: as for outcome 13
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 851 | 730 | 119
participants
  Caucasian/white | 628 | 651 | 101
  Black | 31 | 6 | 1
  Asian/Oriental | 172 | 31 | 5
  Native American/American Indian | 0 | 2 | 0
  Other | 20 | 40 | 12
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

17. Secondary Outcome: Mean Body Weight by IL28B Genotype rs12979860: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including pre-treatment body weight, were obtained from medical records and/or participant interview at the Study Visit. Mean body weight was calculated by averaging the values of all participants within each arm and expressed in kilograms (kg).
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 975 | 1516 | 419
kg | 74.6 [73.7 to 75.6] | 74.4 [73.6 to 75.1] | 74.2 [72.7 to 75.6]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.5468, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

18. Secondary Outcome: Mean Body Weight by IL28B Genotype rs12979860: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including pre-treatment body weight, were obtained from medical records and/or participant interview at the Study Visit. Mean body weight was calculated by averaging the values of all participants within each arm and expressed in kg.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 489 | 913 | 296
kg | 72.7 [71.4 to 73.9] | 75.0 [74.1 to 75.9] | 75.1 [73.5 to 76.7]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.0020, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

19. Secondary Outcome: Mean Body Weight by IL28B Genotype rs8099917: Treatment-Naive
Description: as for outcome 18
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1594 | 1145 | 171
kg | 74.8 [74.0 to 75.5] | 74.2 [73.4 to 75.0] | 72.8 [70.5 to 75.2]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.1623, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

20. Secondary Outcome: Mean Body Weight by IL28B Genotype rs8099917: Treatment-Experienced
Description: as for outcome 18
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 850 | 729 | 119
kg | 73.7 [72.7 to 74.6] | 75.2 [74.2 to 76.2] | 73.8 [71.2 to 76.4]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.0663, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

21. Secondary Outcome: Mean Body Mass Index (BMI) by IL28B Genotype rs12979860: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including height and pre-treatment body weight, were obtained from medical records and/or participant interview at the Study Visit. Each participant's BMI was calculated as weight divided by height-squared, expressed in kilograms per meter-squared (kg/m^2), and mean BMI was calculated by averaging the values of all participants within each arm.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 975 | 1511 | 418
kg/m^2 | 25.8 [25.5 to 26.1] | 26.0 [25.8 to 26.3] | 26.0 [25.6 to 26.5]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.2617, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

22. Secondary Outcome: BMI by IL28B Genotype rs12979860: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Demographic characteristics, including height and pre-treatment body weight, were obtained from medical records and/or participant interview at the Study Visit. Each participant's BMI was calculated as weight divided by height-squared, expressed in kg/m^2, and mean BMI was calculated by averaging the values of all participants within each arm.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 488 | 912 | 293
kg/m^2 | 25.8 [25.5 to 26.2] | 26.4 [26.1 to 26.7] | 26.3 [25.8 to 26.8]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p = 0.0526, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

23. Secondary Outcome: BMI by IL28B Genotype rs8099917: Treatment-Naive
Description: as for outcome 22
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1592 | 1141 | 171
kg/m^2 | 26.0 [25.7 to 26.2] | 26.0 [25.7 to 26.3] | 25.4 [24.8 to 26.1]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.7918, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

24. Secondary Outcome: BMI by IL28B Genotype rs8099917: Treatment-Experienced
Description: as for outcome 22
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 848 | 727 | 118
kg/m^2 | 26.0 [25.7 to 26.3] | 26.4 [26.1 to 26.7] | 26.4 [25.6 to 27.2]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Test type: Superiority or Other; p = 0.0842, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

25. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype was obtained from medical records.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 950 | 1496 | 413
participants
  G1 | 500 | 930 | 272
  G2 | 126 | 160 | 37
  G3 | 232 | 277 | 65
  G4 | 92 | 129 | 39
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

26. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 25
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 476 | 892 | 291
participants
  G1 | 295 | 703 | 239
  G2 | 92 | 38 | 11
  G3 | 63 | 84 | 20
  G4 | 26 | 67 | 21
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

27. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype: Treatment-Naive
Description: as for outcome 25
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1561 | 1131 | 167
participants
  G1 | 837 | 747 | 118
  G2 | 198 | 113 | 12
  G3 | 361 | 186 | 27
  G4 | 165 | 85 | 10
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

28. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 25
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 834 | 709 | 116
participants
  G1 | 563 | 574 | 100
  G2 | 107 | 27 | 7
  G3 | 93 | 65 | 9
  G4 | 71 | 43 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

29. Secondary Outcome: Mean HCV RNA Level by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA level was obtained from medical records. Mean HCV RNA level was calculated by averaging the values of all participants within each arm and expressed in log10 international units per milliliter (log10 IU/mL).
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 928 | 1467 | 407
log10 IU/mL
  G1 (n=481,903,263) | 5.96 [5.87 to 6.06] | 5.89 [5.84 to 5.94] | 5.72 [5.63 to 5.82]
  G2 (n=121,157,36) | 5.95 [5.80 to 6.11] | 5.76 [5.61 to 5.92] | 5.92 [5.62 to 6.21]
  G3 (n=226,268,63) | 6.02 [5.89 to 6.15] | 5.81 [5.71 to 5.91] | 5.51 [5.30 to 5.71]
  G4 (n=84,123,38) | 5.68 [5.50 to 5.86] | 5.59 [5.46 to 5.73] | 5.45 [5.16 to 5.74]
  Other (n=16,16,7) | 5.46 [4.66 to 6.26] | 5.48 [4.87 to 6.08] | 5.58 [4.29 to 6.87]
  Total (n=928,1467,407) | 5.94 [5.88 to 6.01] | 5.83 [5.79 to 5.87] | 5.68 [5.60 to 5.76]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.2887, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.1634, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.8956, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

30. Secondary Outcome: Mean HCV RNA Level by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA level was obtained from medical records. Mean HCV RNA level was calculated by averaging the values of all participants within each arm and expressed in log10 IU/mL.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 382 | 744 | 240
log10 IU/mL
  G1 (n=244,591,196) | 6.06 [5.95 to 6.17] | 5.98 [5.92 to 6.03] | 5.84 [5.75 to 5.93]
  G2 (n=68,30,10) | 5.39 [5.13 to 5.65] | 6.07 [5.79 to 6.35] | 5.64 [5.00 to 6.29]
  G3 (n=38,53,12) | 5.97 [5.64 to 6.30] | 5.78 [5.52 to 6.05] | 5.60 [5.15 to 6.04]
  G4 (n=22,56,20) | 5.49 [5.12 to 5.87] | 5.58 [5.39 to 5.77] | 5.66 [5.31 to 6.00]
  Other (n=10,14,2) | 5.59 [4.57 to 6.61] | 5.63 [5.17 to 6.10] | 4.90 [4.50 to 5.30]
  Total (n=382,744,240) | 5.89 [5.79 to 5.98] | 5.93 [5.88 to 5.98] | 5.80 [5.71 to 5.88]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0145, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.1027, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.5998, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.2935, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.0039, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

31. Primary Outcome: Number of Participants With IL28B Genotype rs12979860 by Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and liver fibrosis stage ('Cirrhotic,' 'Transition to cirrhosis,' 'Advanced fibrosis noncirrhotic,' 'Mild/minimal fibrosis,' and 'No fibrosis') were obtained from medical records. Liver fibrosis stage was based upon previous biopsy using these five categories and captured prior to treatment, if applicable.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 331 | 465 | 126
participants
  G1, Cirrhotic (n=207,324,91) | 10 | 17 | 14
  G1, Transition (n=207,324,91) | 28 | 40 | 17
  G1, Advanced (n=207,324,91) | 51 | 88 | 16
  G1, Mild (n=207,324,91) | 101 | 140 | 34
  G1, No fibrosis (n=207,324,91) | 17 | 39 | 10
  G2, Cirrhotic (n=24,25,5) | 1 | 0 | 0
  G2, Transition (n=24,25,5) | 3 | 5 | 0
  G2, Advanced (n=24,25,5) | 9 | 5 | 1
  G2, Mild (n=24,25,5) | 11 | 13 | 4
  G2, No fibrosis (n=24,25,5) | 0 | 2 | 0
  G3, Cirrhotic (n=67,65,16) | 8 | 6 | 1
  G3, Transition (n=67,65,16) | 12 | 3 | 5
  G3, Advanced (n=67,65,16) | 13 | 12 | 3
  G3, Mild (n=67,65,16) | 28 | 32 | 3
  G3, No fibrosis (n=67,65,16) | 6 | 12 | 4
  G4, Cirrhotic (n=28,48,12) | 1 | 2 | 0
  G4, Transition (n=28,48,12) | 4 | 4 | 1
  G4, Advanced (n=28,48,12) | 6 | 14 | 2
  G4, Mild (n=28,48,12) | 15 | 21 | 8
  G4, No fibrosis (n=28,48,12) | 2 | 7 | 1
  Other, Cirrhotic (n=5,3,2) | 1 | 0 | 0
  Other, Transition (n=5,3,2) | 1 | 0 | 0
  Other, Advanced (n=5,3,2) | 2 | 0 | 0
  Other, Mild (n=5,3,2) | 0 | 2 | 2
  Other, No fibrosis (n=5,3,2) | 1 | 1 | 0
  Total, Cirrhotic (n=331,465,126) | 21 | 25 | 15
  Total, Transition (n=331,465,126) | 48 | 52 | 23
  Total, Advanced (n=331,465,126) | 81 | 119 | 22
  Total, Mild (n=331,465,126) | 155 | 208 | 51
  Total, No fibrosis (n=331,465,126) | 26 | 61 | 15
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.1981, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.1616, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.1192, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.4485, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.1525, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.7262, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

32. Primary Outcome: Number of Participants With IL28B Genotype rs12979860 by Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 31
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 277 | 511 | 164
participants
  G1, Cirrhotic (n=186,422,141) | 20 | 41 | 10
  G1, Transition (n=186,422,141) | 35 | 86 | 26
  G1, Advanced (n=186,422,141) | 63 | 111 | 40
  G1, Mild (n=186,422,141) | 55 | 141 | 50
  G1, No fibrosis (n=186,422,141) | 13 | 43 | 15
  G2, Cirrhotic (n=49,11,5) | 5 | 1 | 0
  G2, Transition (n=49,11,5) | 9 | 2 | 1
  G2, Advanced (n=49,11,5) | 15 | 3 | 1
  G2, Mild (n=49,11,5) | 15 | 5 | 1
  G2, No fibrosis (n=49,11,5) | 5 | 0 | 2
  G3, Cirrhotic (n=26,31,7) | 5 | 5 | 0
  G3, Transition (n=26,31,7) | 3 | 4 | 1
  G3, Advanced (n=26,31,7) | 8 | 5 | 2
  G3, Mild (n=26,31,7) | 8 | 13 | 2
  G3, No fibrosis (n=26,31,7) | 2 | 4 | 2
  G4, Cirrhotic (n=9,35,10) | 0 | 6 | 2
  G4, Transition (n=9,35,10) | 2 | 2 | 0
  G4, Advanced (n=9,35,10) | 2 | 17 | 4
  G4, Mild (n=9,35,10) | 4 | 9 | 3
  G4, No fibrosis (n=9,35,10) | 1 | 1 | 1
  Other, Cirrhotic (n=7,12,1) | 2 | 1 | 0
  Other, Transition (n=7,12,1) | 2 | 2 | 0
  Other, Advanced (n=7,12,1) | 0 | 4 | 0
  Other, Mild (n=7,12,1) | 2 | 5 | 1
  Other, No fibrosis (n=7,12,1) | 1 | 0 | 0
  Total, Cirrhotic (n=277,511,164) | 32 | 54 | 12
  Total, Transition (n=277,511,164) | 51 | 96 | 28
  Total, Advanced (n=277,511,164) | 88 | 140 | 47
  Total, Mild (n=277,511,164) | 84 | 173 | 57
  Total, No fibrosis (n=277,511,164) | 22 | 48 | 20
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0911, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.4674, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.1604, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.5937, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.3830, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.0507, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

33. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 31
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 527 | 343 | 52
participants
  G1, Cirrhotic (n=331,252,39) | 20 | 16 | 5
  G1, Transition (n=331,252,39) | 44 | 34 | 7
  G1, Advanced (n=331,252,39) | 89 | 62 | 4
  G1, Mild (n=331,252,39) | 145 | 110 | 20
  G1, No fibrosis (n=331,252,39) | 33 | 30 | 3
  G2, Cirrhotic (n=33,19,2) | 1 | 0 | 0
  G2, Transition (n=33,19,2) | 5 | 3 | 0
  G2, Advanced (n=33,19,2) | 10 | 4 | 1
  G2, Mild (n=33,19,2) | 17 | 10 | 1
  G2, No fibrosis (n=33,19,2) | 0 | 2 | 0
  G3, Cirrhotic (n=98,42,8) | 13 | 1 | 1
  G3, Transition (n=98,42,8) | 15 | 2 | 3
  G3, Advanced (n=98,42,8) | 18 | 10 | 0
  G3, Mild (n=98,42,8) | 40 | 22 | 1
  G3, No fibrosis (n=98,42,8) | 12 | 7 | 3
  G4, Cirrhotic (n=59,27,2) | 2 | 1 | 0
  G4, Transition (n=59,27,2) | 5 | 4 | 0
  G4, Advanced (n=59,27,2) | 14 | 7 | 1
  G4, Mild (n=59,27,2) | 32 | 11 | 1
  G4, No fibrosis (n=59,27,2) | 6 | 4 | 0
  Other, Cirrhotic (n=6,3,1) | 1 | 0 | 0
  Other, Transition (n=6,3,1) | 1 | 0 | 0
  Other, Advanced (n=6,3,1) | 2 | 0 | 0
  Other, Mild (n=6,3,1) | 1 | 2 | 1
  Other, No fibrosis (n=6,3,1) | 1 | 1 | 0
  Total, Cirrhotic (n=527,343,52) | 37 | 18 | 6
  Total, Transition (n=527,343,52) | 70 | 43 | 10
  Total, Advanced (n=527,343,52) | 133 | 83 | 6
  Total, Mild (n=527,343,52) | 235 | 155 | 24
  Total, No fibrosis (n=527,343,52) | 52 | 44 | 6
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.8686, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.3135, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0578, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.5833, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.1610, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.2925, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

34. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 31
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 468 | 415 | 69
participants
  G1, Cirrhotic (n=332,356,61) | 34 | 32 | 5
  G1, Transition (n=332,356,61) | 58 | 74 | 15
  G1, Advanced (n=332,356,61) | 109 | 92 | 13
  G1, Mild (n=332,356,61) | 106 | 119 | 21
  G1, No fibrosis (n=332,356,61) | 25 | 39 | 7
  G2, Cirrhotic (n=52,9,4) | 6 | 0 | 0
  G2, Transition (n=52,9,4) | 10 | 1 | 1
  G2, Advanced (n=52,9,4) | 15 | 3 | 1
  G2, Mild (n=52,9,4) | 16 | 5 | 0
  G2, No fibrosis (n=52,9,4) | 5 | 0 | 2
  G3, Cirrhotic (n=38,22,4) | 6 | 4 | 0
  G3, Transition (n=38,22,4) | 5 | 2 | 1
  G3, Advanced (n=38,22,4) | 9 | 5 | 1
  G3, Mild (n=38,22,4) | 13 | 9 | 1
  G3, No fibrosis (n=38,22,4) | 5 | 2 | 1
  G4, Cirrhotic (n=37,17,0) | 4 | 4 | 0
  G4, Transition (n=37,17,0) | 2 | 2 | 0
  G4, Advanced (n=37,17,0) | 18 | 5 | 0
  G4, Mild (n=37,17,0) | 10 | 6 | 0
  G4, No fibrosis (n=37,17,0) | 3 | 0 | 0
  Other, Cirrhotic (n=9,11,0) | 2 | 1 | 0
  Other, Transition (n=9,11,0) | 3 | 1 | 0
  Other, Advanced (n=9,11,0) | 1 | 3 | 0
  Other, Mild (n=9,11,0) | 2 | 6 | 0
  Other, No fibrosis (n=9,11,0) | 1 | 0 | 0
  Total, Cirrhotic (n=468,415,69) | 52 | 41 | 5
  Total, Transition (n=468,415,69) | 78 | 80 | 17
  Total, Advanced (n=468,415,69) | 152 | 108 | 15
  Total, Mild (n=468,415,69) | 147 | 145 | 22
  Total, No fibrosis (n=468,415,69) | 39 | 41 | 10
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.3709, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.2054, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.8457, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.3492, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.2846, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.2646, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

35. Primary Outcome: Number of Participants With IL28B Genotype rs12979860 by METAVIR Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and liver fibrosis stage (Stage F0, Stage F1, Stage F2, Stage F3, or Stage F4) were obtained from medical records. Liver fibrosis stage was based upon previous biopsy using the METAVIR scoring system and captured prior to treatment, if applicable.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 166 | 249 | 77
participants
  G1, Stage F0 (n=95,177,56) | 6 | 20 | 5
  G1, Stage F1 (n=95,177,56) | 33 | 63 | 16
  G1, Stage F2 (n=95,177,56) | 34 | 57 | 15
  G1, Stage F3 (n=95,177,56) | 16 | 23 | 9
  G1, Stage F4 (n=95,177,56) | 6 | 14 | 11
  G2, Stage F0 (n=15,11,2) | 0 | 0 | 0
  G2, Stage F1 (n=15,11,2) | 6 | 5 | 2
  G2, Stage F2 (n=15,11,2) | 6 | 2 | 0
  G2, Stage F3 (n=15,11,2) | 2 | 4 | 0
  G2, Stage F4 (n=15,11,2) | 1 | 0 | 0
  G3, Stage F0 (n=31,26,9) | 0 | 3 | 2
  G3, Stage F1 (n=31,26,9) | 8 | 10 | 2
  G3, Stage F2 (n=31,26,9) | 9 | 7 | 1
  G3, Stage F3 (n=31,26,9) | 7 | 2 | 4
  G3, Stage F4 (n=31,26,9) | 7 | 4 | 0
  G4, Stage F0 (n=21,35,8) | 2 | 6 | 1
  G4, Stage F1 (n=21,35,8) | 12 | 12 | 5
  G4, Stage F2 (n=21,35,8) | 4 | 13 | 1
  G4, Stage F3 (n=21,35,8) | 3 | 3 | 1
  G4, Stage F4 (n=21,35,8) | 0 | 1 | 0
  Other, Stage F0 (n=4,0,2) | 1 | 0 | 0
  Other, Stage F1 (n=4,0,2) | 0 | 0 | 2
  Other, Stage F2 (n=4,0,2) | 2 | 0 | 0
  Other, Stage F3 (n=4,0,2) | 1 | 0 | 0
  Other, Stage F4 (n=4,0,2) | 0 | 0 | 0
  Total, Stage F0 (n=166,249,77) | 9 | 29 | 8
  Total, Stage F1 (n=166,249,77) | 59 | 90 | 27
  Total, Stage F2 (n=166,249,77) | 55 | 79 | 17
  Total, Stage F3 (n=166,249,77) | 29 | 32 | 14
  Total, Stage F4 (n=166,249,77) | 14 | 19 | 11
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.5348, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.5469, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0463, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.9393, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.3404, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.4237, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

36. Primary Outcome: Number of Participants With IL28B Genotype rs12979860 by METAVIR Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 35
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 174 | 322 | 86
participants
  G1, Stage F0 (n=119,259,70) | 7 | 20 | 8
  G1, Stage F1 (n=119,259,70) | 28 | 61 | 15
  G1, Stage F2 (n=119,259,70) | 44 | 83 | 31
  G1, Stage F3 (n=119,259,70) | 26 | 62 | 12
  G1, Stage F4 (n=119,259,70) | 14 | 33 | 4
  G2, Stage F0 (n=31,7,1) | 1 | 0 | 1
  G2, Stage F1 (n=31,7,1) | 11 | 3 | 0
  G2, Stage F2 (n=31,7,1) | 9 | 3 | 0
  G2, Stage F3 (n=31,7,1) | 6 | 0 | 0
  G2, Stage F4 (n=31,7,1) | 4 | 1 | 0
  G3, Stage F0 (n=16,23,5) | 1 | 3 | 2
  G3, Stage F1 (n=16,23,5) | 3 | 8 | 1
  G3, Stage F2 (n=16,23,5) | 6 | 5 | 2
  G3, Stage F3 (n=16,23,5) | 1 | 3 | 0
  G3, Stage F4 (n=16,23,5) | 5 | 4 | 0
  G4, Stage F0 (n=5,30,9) | 0 | 0 | 1
  G4, Stage F1 (n=5,30,9) | 1 | 7 | 2
  G4, Stage F2 (n=5,30,9) | 2 | 16 | 4
  G4, Stage F3 (n=5,30,9) | 2 | 2 | 0
  G4, Stage F4 (n=5,30,9) | 0 | 5 | 2
  Other, Stage F0 (n=3,3,1) | 0 | 0 | 0
  Other, Stage F1 (n=3,3,1) | 1 | 1 | 1
  Other, Stage F2 (n=3,3,1) | 0 | 1 | 0
  Other, Stage F3 (n=3,3,1) | 1 | 0 | 0
  Other, Stage F4 (n=3,3,1) | 1 | 1 | 0
  Total, Stage F0 (n=174,322,86) | 9 | 23 | 12
  Total, Stage F1 (n=174,322,86) | 44 | 80 | 19
  Total, Stage F2 (n=174,322,86) | 61 | 108 | 37
  Total, Stage F3 (n=174,322,86) | 36 | 67 | 12
  Total, Stage F4 (n=174,322,86) | 24 | 44 | 6
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.2510, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.2943, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0478, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.5387, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.3878, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.0748, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

37. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by METAVIR Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 35
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 277 | 187 | 28
participants
  G1, Stage F0 (n=168,139,21) | 13 | 16 | 2
  G1, Stage F1 (n=168,139,21) | 59 | 45 | 8
  G1, Stage F2 (n=168,139,21) | 59 | 43 | 4
  G1, Stage F3 (n=168,139,21) | 22 | 22 | 4
  G1, Stage F4 (n=168,139,21) | 15 | 13 | 3
  G2, Stage F0 (n=20,7,1) | 0 | 0 | 0
  G2, Stage F1 (n=20,7,1) | 10 | 2 | 1
  G2, Stage F2 (n=20,7,1) | 6 | 2 | 0
  G2, Stage F3 (n=20,7,1) | 3 | 3 | 0
  G2, Stage F4 (n=20,7,1) | 1 | 0 | 0
  G3, Stage F0 (n=42,20,4) | 2 | 2 | 1
  G3, Stage F1 (n=42,20,4) | 10 | 9 | 1
  G3, Stage F2 (n=42,20,4) | 11 | 6 | 0
  G3, Stage F3 (n=42,20,4) | 9 | 2 | 2
  G3, Stage F4 (n=42,20,4) | 10 | 1 | 0
  G4, Stage F0 (n=43,20,1) | 6 | 3 | 0
  G4, Stage F1 (n=43,20,1) | 22 | 7 | 0
  G4, Stage F2 (n=43,20,1) | 11 | 6 | 1
  G4, Stage F3 (n=43,20,1) | 4 | 3 | 0
  G4, Stage F4 (n=43,20,1) | 0 | 1 | 0
  Other, Stage F0 (n=4,1,1) | 1 | 0 | 0
  Other, Stage F1 (n=4,1,1) | 0 | 1 | 1
  Other, Stage F2 (n=4,1,1) | 2 | 0 | 0
  Other, Stage F3 (n=4,1,1) | 1 | 0 | 0
  Other, Stage F4 (n=4,1,1) | 0 | 0 | 0
  Total, Stage F0 (n=277,187,28) | 22 | 21 | 3
  Total, Stage F1 (n=277,187,28) | 101 | 64 | 11
  Total, Stage F2 (n=277,187,28) | 89 | 57 | 5
  Total, Stage F3 (n=277,187,28) | 39 | 30 | 6
  Total, Stage F4 (n=277,187,28) | 26 | 15 | 3
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.9887, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.5507, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0175, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.2246, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.3519, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.7140, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

38. Primary Outcome: Number of Participants With IL28B Genotype rs8099917 by METAVIR Liver Fibrosis Stage and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 35
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 291 | 256 | 35
participants
  G1, Stage F0 (n=200,217,31) | 14 | 18 | 3
  G1, Stage F1 (n=200,217,31) | 46 | 50 | 8
  G1, Stage F2 (n=200,217,31) | 74 | 74 | 10
  G1, Stage F3 (n=200,217,31) | 45 | 48 | 7
  G1, Stage F4 (n=200,217,31) | 21 | 27 | 3
  G2, Stage F0 (n=33,5,1) | 1 | 0 | 1
  G2, Stage F1 (n=33,5,1) | 12 | 2 | 0
  G2, Stage F2 (n=33,5,1) | 9 | 3 | 0
  G2, Stage F3 (n=33,5,1) | 6 | 0 | 0
  G2, Stage F4 (n=33,5,1) | 5 | 0 | 0
  G3, Stage F0 (n=25,16,3) | 3 | 2 | 1
  G3, Stage F1 (n=25,16,3) | 6 | 5 | 1
  G3, Stage F2 (n=25,16,3) | 7 | 5 | 1
  G3, Stage F3 (n=25,16,3) | 3 | 1 | 0
  G3, Stage F4 (n=25,16,3) | 6 | 3 | 0
  G4, Stage F0 (n=30,14,0) | 1 | 0 | 0
  G4, Stage F1 (n=30,14,0) | 7 | 3 | 0
  G4, Stage F2 (n=30,14,0) | 17 | 5 | 0
  G4, Stage F3 (n=30,14,0) | 2 | 2 | 0
  G4, Stage F4 (n=30,14,0) | 3 | 4 | 0
  Other, Stage F0 (n=3,4,0) | 0 | 0 | 0
  Other, Stage F1 (n=3,4,0) | 1 | 2 | 0
  Other, Stage F2 (n=3,4,0) | 0 | 1 | 0
  Other, Stage F3 (n=3,4,0) | 1 | 0 | 0
  Other, Stage F4 (n=3,4,0) | 1 | 1 | 0
  Total, Stage F0 (n=291,256,35) | 19 | 20 | 5
  Total, Stage F1 (n=291,256,35) | 72 | 62 | 9
  Total, Stage F2 (n=291,256,35) | 107 | 88 | 11
  Total, Stage F3 (n=291,256,35) | 57 | 51 | 7
  Total, Stage F4 (n=291,256,35) | 36 | 35 | 3
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.8622, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.1622, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.2566, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.1574, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.5784, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.6603, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

39. Primary Outcome: Mean FibroScan Values by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and liver elastography (FibroScan) were obtained from medical records. FibroScan values were based upon previous noninvasive assessment captured prior to treatment, if applicable. Mean FibroScan values were determined by averaging the values of all participants within each arm and expressed in kilopascals (kPa).
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 324 | 517 | 140
kPa
  G1 (n=177,316,82) | 9.61 [8.51 to 10.7] | 10.2 [9.22 to 11.1] | 12.6 [10.3 to 15.0]
  G2 (n=40,55,15) | 11.1 [7.26 to 14.9] | 7.69 [6.65 to 8.72] | 7.15 [4.35 to 9.94]
  G3 (n=60,83,24) | 11.7 [9.45 to 14.0] | 9.3 [7.82 to 10.8] | 8.99 [6.14 to 11.8]
  G4 (n=43,59,18) | 11.4 [7.54 to 15.3] | 13.4 [10.4 to 16.5] | 11.1 [5.85 to 16.4]
  Other (n=4,4,1) | 12.1 [4.65 to 19.6] | 21.9 [-34.4 to 78.2] | 4.00 [NA to NA] — Confidence interval not presented because the analysis only included 1 participant.
  Total (n=324,517,140) | 10.5 [9.45 to 11.4] | 10.2 [9.46 to 11.0] | 11.2 [9.53 to 12.8]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0605, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0899, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0634, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.6165, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.1649, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.9159, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

40. Primary Outcome: Mean FibroScan Values by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and liver elastography (FibroScan) were obtained from medical records. FibroScan values were based upon previous noninvasive assessment captured prior to treatment, if applicable. Mean FibroScan values were determined by averaging the values of all participants within each arm and expressed in kPa.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 54 | 122 | 39
kPa
  G1 (n=27,84,32) | 11.7 [8.4 to 14.9] | 13.2 [10.3 to 16.2] | 13.5 [9.69 to 17.4]
  G2 (n=6,10,0) | 13.3 [6.37 to 20.2] | 5.11 [4.06 to 6.16] | 8.17 [5.14 to 11.2]
  G3 (n=15,14,4) | 12.3 [6.57 to 18.1] | 8.64 [5.22 to 12.1] | 9.48 [0.708 to 18.2]
  G4 (n=6,14,3) | 10.7 [-2.17 to 23.5] | 10.6 [6.16 to 15.0] | 8.9 [-0.589 to 18.4]
  Other (n=0,0,0) | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0. | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0. | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Total (n=54,122,39) | 11.9 [9.46 to 14.4] | 11.7 [9.61 to 13.9] | 12.8 [9.54 to 16.0]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.7454, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0016, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.5261, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.3422, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.9026, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

41. Primary Outcome: Mean FibroScan Values by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 40
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 528 | 404 | 49
kPa
  G1 (n=287,259,29) | 9.46 [8.61 to 10.3] | 10.9 [9.78 to 12.1] | 13.7 [9.77 to 17.6]
  G2 (n=63,42,5) | 9.44 [6.96 to 11.9] | 7.95 [6.73 to 9.18] | 8.76 [-1.92 to 19.4]
  G3 (n=100,57,10) | 11.4 [9.67 to 13.2] | 8.45 [7.30 to 9.60] | 6.51 [2.86 to 10.2]
  G4 (n=72,44,4) | 11.2 [8.63 to 13.8] | 14.2 [10.2 to 18.2] | 13.7 [-9.32 to 36.6]
  Other (n=6,2,1) | 9.32 [3.40 to 15.2] | 40.1 [-403 to 484] | 4.00 [NA to NA] — Confidence interval not presented because the analysis only included 1 participant.
  Total (n=528,404,49) | 10.1 [9.34 to 10.8] | 10.8 [9.83 to 11.7] | 11.5 [8.70 to 14.3]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0017, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.8864, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0291, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.5472, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 1.000, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.1148, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

42. Primary Outcome: Mean FibroScan Values by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 40
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 97 | 103 | 15
kPa
  G1 (n=53,77,13) | 12.7 [9.89 to 15.5] | 13.7 [10.6 to 16.9] | 10.2 [7.00 to 13.4]
  G2 (n=9,7,0) | 10.5 [5.31 to 15.6] | 5.21 [3.71 to 6.72] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  G3 (n=21,10,2) | 12.1 [7.70 to 16.4] | 7.82 [5.00 to 10.6] | 5.95 [-8.66 to 20.6]
  G4 (n=14,9,0) | 9.74 [4.76 to 14.7] | 11.4 [4.95 to 17.8] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Other (n=0,0,0) | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0. | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0. | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Total (n=97,103,15) | 11.9 [10.0 to 13.8] | 12.4 [9.91 to 14.8] | 9.62 [6.79 to 12.5]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.4207, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0566, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.1211, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.3772, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.4023, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

43. Secondary Outcome: Mean HCV RNA Level by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 30
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1529 | 1108 | 165
log10 IU/mL
  G1 (n=809,723,115) | 5.99 [5.92 to 6.05] | 5.82 [5.76 to 5.87] | 5.61 [5.47 to 5.75]
  G2 (n=191,111,12) | 5.90 [5.76 to 6.03] | 5.74 [5.57 to 5.92] | 6.20 [5.80 to 6.59]
  G3 (n=350,181,26) | 5.99 [5.88 to 6.09] | 5.69 [5.57 to 5.80] | 5.39 [5.10 to 5.68]
  G4 (n=155,82,8) | 5.64 [5.51 to 5.77] | 5.53 [5.35 to 5.71] | 5.53 [4.98 to 6.07]
  Other (n=24,11,4) | 5.53 [4.95 to 6.10] | 5.13 [4.24 to 6.01] | 6.27 [5.13 to 7.42]
  Total (n=1529,1108,165) | 5.93 [5.89 to 5.98] | 5.76 [5.71 to 5.81] | 5.63 [5.51 to 5.75]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.2132, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.3031, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.9550, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

44. Secondary Outcome: Mean HCV RNA Level by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 30
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 679 | 594 | 93
log10 IU/mL
  G1 (n=469,480,82) | 6.04 [5.97 to 6.12] | 5.92 [5.86 to 5.97] | 5.85 [5.71 to 5.99]
  G2 (n=81,21,6) | 5.52 [5.29 to 5.75] | 5.97 [5.60 to 6.33] | 5.49 [4.39 to 6.58]
  G3 (n=59,39,5) | 5.87 [5.61 to 6.13] | 5.78 [5.47 to 6.10] | 5.73 [5.14 to 6.32]
  G4 (n=59,39,0) | 5.67 [5.49 to 5.85] | 5.43 [5.18 to 5.69] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Other (n=11,15,0) | 5.59 [4.68 to 6.49] | 5.54 [5.09 to 5.99] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Total (n=679,594,93) | 5.93 [5.86 to 5.99] | 5.87 [5.81 to 5.92] | 5.82 [5.68 to 5.96]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.1890, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.5793, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.0847, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.5506, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0020, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

45. Secondary Outcome: Mean Alanine Aminotransferase (ALT) Ratio by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. ALT level was obtained from medical records captured prior to treatment, if applicable. Each participant's ALT ratio was calculated as ALT level divided by the upper limit of normal (55 international units per liter [IU/L] for males and 30 IU/L for females). Mean ALT ratio was calculated by averaging the values of all participants within each arm.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 955 | 1480 | 416
ratio
  G1 (n=488,914,269) | 2.09 [1.92 to 2.27] | 1.77 [1.68 to 1.86] | 1.63 [1.47 to 1.79]
  G2 (n=123,152,37) | 2.42 [1.96 to 2.88] | 1.96 [1.64 to 2.27] | 1.21 [0.932 to 1.48]
  G3 (n=228,272,65) | 2.80 [2.52 to 3.08] | 2.32 [2.09 to 2.55] | 2.05 [1.64 to 2.45]
  G4 (n=88,121,38) | 2.00 [1.63 to 2.37] | 1.66 [1.46 to 1.86] | 1.65 [1.29 to 2.01]
  Other (n=28,21,7) | 1.46 [0.964 to 1.96] | 1.72 [1.13 to 2.31] | 1.33 [0.686 to 1.98]
  Total (n=955,1480,416) | 2.28 [2.14 to 2.41] | 1.88 [1.80 to 1.96] | 1.65 [1.53 to 1.78]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0007, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0061, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.3885, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.3597, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

46. Secondary Outcome: Mean ALT Ratio by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. ALT level was obtained from medical records captured prior to treatment, if applicable. Each participant's ALT ratio was calculated as ALT level divided by the upper limit of normal (55 IU/L for males and 30 IU/L for females). Mean ALT ratio was calculated by averaging the values of all participants within each arm.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 398 | 686 | 229
ratio
  G1 (n=241,528,184) | 3.00 [2.69 to 3.32] | 2.14 [2.00 to 2.29] | 2.00 [1.75 to 2.25]
  G2 (n=80,32,9) | 3.45 [2.73 to 4.18] | 1.84 [1.24 to 2.43] | 2.02 [0.934 to 3.10]
  G3 (n=45,66,17) | 3.06 [2.55 to 3.58] | 2.49 [2.03 to 2.96] | 2.27 [1.38 to 3.16]
  G4 (n=23,47,17) | 1.65 [1.20 to 2.11] | 1.79 [1.42 to 2.16] | 1.23 [0.768 to 1.70]
  Other (n=9,13,2) | 2.99 [1.03 to 4.95] | 1.82 [1.06 to 2.57] | 2.17 [-12.4 to 16.8]
  Total (n=398,686,229) | 3.02 [2.77 to 3.27] | 2.13 [2.01 to 2.26] | 1.96 [1.75 to 2.18]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0005, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0110, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0980, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.2264, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

47. Secondary Outcome: Mean ALT Ratio by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 46
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1557 | 1126 | 168
ratio
  G1 (n=818,737,116) | 2.02 [1.90 to 2.15] | 1.67 [1.58 to 1.75] | 1.67 [1.42 to 1.92]
  G2 (n=192,108,12) | 2.09 [1.77 to 2.41] | 2.06 [1.65 to 2.46] | 1.31 [0.622 to 2.01]
  G3 (n=355,183,27) | 2.72 [2.49 to 2.96] | 2.08 [1.88 to 2.28] | 2.03 [1.49 to 2.57]
  G4 (n=155,83,9) | 1.78 [1.55 to 2.02] | 1.84 [1.57 to 2.10] | 1.20 [1.04 to 1.35]
  Other (n=37,15,4) | 1.66 [1.20 to 2.12] | 1.25 [0.803 to 1.69] | 1.56 [0.139 to 2.99]
  Total (n=1557,1126,168) | 2.16 [2.06 to 2.26] | 1.78 [1.70 to 1.86] | 1.67 [1.47 to 1.87]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0098, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.6291, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0013, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.5588, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.9932, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

48. Secondary Outcome: Mean ALT Ratio by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 46
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 667 | 556 | 90
ratio
  G1 (n=442,437,74) | 2.60 [2.39 to 2.82] | 2.11 [1.96 to 2.27] | 2.00 [1.71 to 2.29]
  G2 (n=92,23,6) | 3.26 [2.61 to 3.91] | 1.79 [1.06 to 2.53] | 2.04 [0.297 to 3.78]
  G3 (n=68,51,9) | 3.04 [2.62 to 3.47] | 2.29 [1.75 to 2.83] | 1.90 [1.28 to 2.52]
  G4 (n=54,33,0) | 1.58 [1.32 to 1.84] | 1.76 [1.25 to 2.27] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Other (n=11,12,1) | 2.78 [1.18 to 4.38] | 1.75 [0.949 to 2.54] | 3.32 [NA to NA] — Confidence interval not presented because the analysis only included 1 participant.
  Total (n=667,556,90) | 2.66 [2.48 to 2.84] | 2.09 [1.95 to 2.23] | 2.01 [1.75 to 2.27]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0007, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0020, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0013, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.7166, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.3217, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

49. Secondary Outcome: Mean Aspartate Aminotransferase (AST) Ratio by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. AST level was obtained from medical records captured prior to treatment, if applicable. Each participant's AST ratio was calculated as AST level divided by the upper limit of normal (40 IU/L for males and 25 IU/L for females). Mean AST ratio was calculated by averaging the values of all participants within each arm.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 940 | 1444 | 405
ratio
  G1 (n=480,891,264) | 1.62 [1.51 to 1.73] | 1.59 [1.51 to 1.66] | 1.46 [1.34 to 1.58]
  G2 (n=122,151,37) | 1.93 [1.61 to 2.26] | 1.63 [1.38 to 1.87] | 1.06 [0.827 to 1.29]
  G3 (n=227,266,64) | 2.17 [2.00 to 2.35] | 1.88 [1.69 to 2.07] | 1.44 [1.21 to 1.67]
  G4 (n=83,118,33) | 1.71 [1.39 to 2.03] | 1.54 [1.33 to 1.75] | 1.41 [1.12 to 1.70]
  Other (n=28,18,7) | 1.41 [0.899 to 1.92] | 1.63 [0.952 to 2.31] | 1.29 [0.605 to 1.97]
  Total (n=940,1444,405) | 1.80 [1.71 to 1.89] | 1.64 [1.57 to 1.71] | 1.41 [1.32 to 1.50]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.1894, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0054, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.5360, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.2185, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

50. Secondary Outcome: Mean AST Ratio by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 49
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 391 | 655 | 218
ratio
  G1 (n=234,501,173) | 2.27 [2.02 to 2.51] | 1.78 [1.66 to 1.90] | 1.65 [1.48 to 1.83]
  G2 (n=80,32,9) | 2.49 [2.08 to 2.90] | 1.33 [0.966 to 1.70] | 1.58 [0.802 to 2.36]
  G3 (n=45,63,17) | 2.42 [1.98 to 2.87] | 2.07 [1.65 to 2.50] | 1.71 [1.09 to 2.32]
  G4 (n=23,46,17) | 1.31 [0.985 to 1.63] | 1.52 [1.23 to 1.81] | 1.36 [0.856 to 1.86]
  Other (n=9,13,2) | 1.86 [1.00 to 2.71] | 1.47 [1.03 to 1.92] | 1.09 [-3.50 to 5.68]
  Total (n=391,655,218) | 2.27 [2.09 to 2.44] | 1.76 [1.66 to 1.86] | 1.63 [1.48 to 1.78]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0002, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0003, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0106, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.7821, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.2372, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

51. Secondary Outcome: Mean AST Ratio by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 49
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1524 | 1105 | 160
ratio
  G1 (n=800,724,111) | 1.65 [1.56 to 1.73] | 1.51 [1.43 to 1.59] | 1.49 [1.30 to 1.69]
  G2 (n=190,108,12) | 1.71 [1.48 to 1.94] | 1.66 [1.35 to 1.98] | 1.37 [0.725 to 2.02]
  G3 (n=350,181,26) | 2.13 [1.96 to 2.29] | 1.68 [1.51 to 1.85] | 1.42 [1.07 to 1.77]
  G4 (n=148,79,7) | 1.54 [1.33 to 1.75] | 1.69 [1.42 to 1.96] | 1.14 [0.708 to 1.58]
  Other (n=36,13,4) | 1.41 [0.996 to 1.82] | 1.62 [0.707 to 2.54] | 1.51 [0.0157 to 3.00]
  Total (n=1524,1105,160) | 1.75 [1.68 to 1.82] | 1.57 [1.50 to 1.64] | 1.46 [1.30 to 1.61]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0688, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.4367, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.1951, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.2927, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0013, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

52. Secondary Outcome: Mean AST Ratio by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 49
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 647 | 531 | 86
ratio
  G1 (n=423,415,70) | 2.01 [1.86 to 2.17] | 1.78 [1.65 to 1.92] | 1.66 [1.40 to 1.92]
  G2 (n=92,23,6) | 2.34 [1.97 to 2.71] | 1.36 [0.874 to 1.85] | 1.61 [0.494 to 2.73]
  G3 (n=67,49,9) | 2.36 [2.02 to 2.69] | 1.96 [1.44 to 2.49] | 1.63 [0.697 to 2.56]
  G4 (n=54,32,0) | 1.30 [1.13 to 1.48] | 1.65 [1.21 to 2.10] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Other (n=11,12,1) | 1.79 [1.11 to 2.47] | 1.41 [0.905 to 1.91] | 1.45 [NA to NA] — Confidence interval not presented because the analysis only included 1 participant.
  Total (n=647,531,86) | 2.03 [1.91 to 2.16] | 1.77 [1.65 to 1.88] | 1.65 [1.42 to 1.88]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0247, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0034, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0017, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.3346, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.3215, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0003, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

53. Secondary Outcome: Mean Platelet Count by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Platelet count was obtained from medical records captured prior to treatment, if applicable. Mean platelet count was calculated by averaging the values of all participants within each arm and expressed in 10^9 cells per liter (10^9 cells/L).
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 939 | 1458 | 415
10^9 cells/L
  G1 (n=483,900,269) | 200 [195 to 205] | 204 [200 to 208] | 201 [194 to 208]
  G2 (n=121,147,37) | 190 [180 to 200] | 212 [201 to 222] | 203 [189 to 218]
  G3 (n=225,268,64) | 186 [180 to 193] | 201 [194 to 207] | 193 [182 to 204]
  G4 (n=85,124,38) | 198 [185 to 211] | 191 [182 to 200] | 189 [177 to 201]
  Other (n=25,19,7) | 216 [169 to 263] | 203 [172 to 234] | 195 [165 to 225]
  Total (n=939,1458,415) | 196 [192 to 199] | 203 [200 to 206] | 199 [194 to 204]
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.3609, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0018, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0356, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.7044, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.8578, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p = 0.0076, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

54. Secondary Outcome: Mean Platelet Count by IL28B Genotype rs12979860 and HCV RNA Genotype: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. Platelet count was obtained from medical records captured prior to treatment, if applicable. Mean platelet count was calculated by averaging the values of all participants within each arm and expressed in 10^9 cells/L.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 383 | 651 | 210
10^9 cells/L
  G1 (n=233,501,167) | 180 [173 to 186] | 196 [191 to 202] | 197 [189 to 205]
  G2 (n=74,29,8) | 166 [154 to 178] | 181 [167 to 195] | 165 [102 to 228]
  G3 (n=46,65,17) | 182 [167 to 197] | 191 [176 to 206] | 191 [161 to 221]
  G4 (n=22,43,17) | 194 [180 to 208] | 184 [171 to 197] | 185 [161 to 209]
  Other (n=8,13,1) | 173. [142 to 204] | 202 [150 to 255] | 209 [NA to NA] — Confidence interval not presented because the analysis only included 1 participant.
  Total (n=383,651,210) | 178 [173 to 183] | 194 [190 to 199] | 194 [187 to 202]
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0002, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.2017, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.5878, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.4144, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.4492, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

55. Secondary Outcome: Mean Platelet Count by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Naive
Description: as for outcome 54
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1538 | 1106 | 168
10^9 cells/L
  G1 (n=810,727,115) | 200 [196 to 203] | 205 [200 to 210] | 203 [191 to 215]
  G2 (n=188,105,12) | 199 [190 to 207] | 209 [198 to 219] | 194 [158 to 229]
  G3 (n=351,179,27) | 191 [185 to 196] | 201 [193 to 208] | 196 [178 to 214]
  G4 (n=156,81,10) | 195 [187 to 204] | 190 [178 to 202] | 185 [159 to 211]
  Other (n=33,14,4) | 216 [180 to 252] | 193 [157 to 229] | 199 [139 to 258]
  Total (n=1538,1106,168) | 197 [194 to 200] | 203 [200 to 207] | 200 [191 to 209]
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0671, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.1009, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.0635, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.4162, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.9305, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0041, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

56. Secondary Outcome: Mean Platelet Count by IL28B Genotype rs8099917 and HCV RNA Genotype: Treatment-Experienced
Description: as for outcome 54
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 641 | 519 | 84
10^9 cells/L
  G1 (n=426,406,69) | 186 [181 to 192] | 199 [192 to 205] | 190 [180 to 200]
  G2 (n=84,21,6) | 167 [156 to 178] | 184 [157 to 210] | 162 [126 to 197]
  G3 (n=68,51,9) | 180 [168 to 191] | 199 [180 to 219] | 182 [149 to 214]
  G4 (n=53,29,0) | 189 [178 to 200] | 182 [167 to 197] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Other (n=10,12,0) | 194 [131 to 257] | 190 [155 to 226] | NA [NA to NA] — The total number of participants analyzed in this arm/group by category was 0.
  Total (n=641,519,64) | 183 [179 to 188] | 197 [192 to 202] | 187 [178 to 196]
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0059, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.2808, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.2401, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.2993, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.5529, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0005, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of a continuous variable across the three IL28B genotype categories

57. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Region: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype was obtained from medical records, and geographic region of study site was documented during intake/enrollment.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  G1, Asia (n=500,930,272) | 16 | 9 | 0
  G1, Europe (n=500,930,272) | 388 | 680 | 183
  G1, Middle East (n=500,930,272) | 65 | 167 | 57
  G1, Latin America (n=500,930,272) | 31 | 74 | 32
  G2, Asia (n=126,160,37) | 4 | 2 | 0
  G2, Europe (n=126,160,37) | 111 | 144 | 36
  G2, Middle East (n=126,160,37) | 7 | 12 | 0
  G2, Latin America (n=126,160,37) | 4 | 2 | 1
  G3, Asia (n=232,277,65) | 45 | 52 | 8
  G3, Europe (n=232,277,65) | 177 | 200 | 55
  G3, Middle East (n=232,277,65) | 8 | 20 | 2
  G3, Latin America (n=232,277,65) | 2 | 5 | 0
  G4, Asia (n=92,129,39) | 0 | 0 | 0
  G4, Europe (n=92,129,39) | 37 | 64 | 27
  G4, Middle East (n=92,129,39) | 53 | 62 | 12
  G4, Latin America (n=92,129,39) | 2 | 3 | 0
  Other, Asia (n=28,22,7) | 13 | 3 | 0
  Other, Europe (n=28,22,7) | 8 | 7 | 2
  Other, Middle East (n=28,22,7) | 5 | 11 | 4
  Other, Latin America (n=28,22,7) | 2 | 1 | 1
  Total, Asia (n=978,1518,420) | 78 | 66 | 8
  Total, Europe (n=978,1518,420) | 721 | 1095 | 303
  Total, Middle East (n=978,1518,420) | 138 | 272 | 75
  Total, Latin America (n=978,1518,420) | 41 | 85 | 34
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.3572, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.2041, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0467, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.0525, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

58. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Region: Treatment-Experienced
Description: as for outcome 57
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  G1, Asia (n=295,703,239) | 83 | 13 | 0
  G1, Europe (n=295,703,239) | 174 | 534 | 186
  G1, Middle East (n=295,703,239) | 17 | 87 | 30
  G1, Latin America (n=295,703,239) | 21 | 69 | 23
  G2, Asia (n=92,38,11) | 59 | 8 | 1
  G2, Europe (n=92,38,11) | 29 | 28 | 6
  G2, Middle East (n=92,38,11) | 2 | 1 | 2
  G2, Latin America (n=92,38,11) | 2 | 1 | 2
  G3, Asia (n=63,84,20) | 9 | 14 | 3
  G3, Europe (n=63,84,20) | 52 | 61 | 15
  G3, Middle East (n=63,84,20) | 0 | 3 | 0
  G3, Latin America (n=63,84,20) | 2 | 6 | 2
  G4, Asia (n=26,67,21) | 0 | 0 | 0
  G4, Europe (n=26,67,21) | 14 | 36 | 14
  G4, Middle East (n=26,67,21) | 12 | 29 | 7
  G4, Latin America (n=26,67,21) | 0 | 2 | 0
  Other, Asia (n=14,22,5) | 4 | 1 | 0
  Other, Europe (n=14,22,5) | 6 | 5 | 1
  Other, Middle East (n=14,22,5) | 2 | 15 | 4
  Other, Latin America (n=14,22,5) | 2 | 1 | 0
  Total, Asia (n=490,914,296) | 155 | 36 | 4
  Total, Europe (n=490,914,296) | 275 | 664 | 222
  Total, Middle East (n=490,914,296) | 33 | 135 | 43
  Total, Latin America (n=490,914,296) | 27 | 79 | 27
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.5275, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.6593, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.0372, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

59. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Region: Treatment-Naive
Description: as for outcome 57
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1598 | 1147 | 171
participants
  G1, Asia (n=837,747,118) | 19 | 6 | 0
  G1, Europe (n=837,747,118) | 632 | 543 | 76
  G1, Middle East (n=837,747,118) | 138 | 130 | 21
  G1, Latin America (n=837,747,118) | 48 | 68 | 21
  G2, Asia (n=198,113,12) | 4 | 2 | 0
  G2, Europe (n=198,113,12) | 174 | 106 | 11
  G2, Middle East (n=198,113,12) | 15 | 4 | 0
  G2, Latin America (n=198,113,12) | 5 | 1 | 1
  G3, Asia (n=361,186,27) | 67 | 33 | 5
  G3, Europe (n=361,186,27) | 275 | 135 | 22
  G3, Middle East (n=361,186,27) | 17 | 13 | 0
  G3, Latin America (n=361,186,27) | 2 | 5 | 0
  G4, Asia (n=165,85,10) | 0 | 0 | 0
  G4, Europe (n=165,85,10) | 77 | 46 | 5
  G4, Middle East (n=165,85,10) | 85 | 37 | 5
  G4, Latin America (n=165,85,10) | 3 | 2 | 0
  Other, Asia (n=37,16,4) | 14 | 2 | 0
  Other, Europe (n=37,16,4) | 11 | 4 | 2
  Other, Middle East (n=37,16,4) | 9 | 9 | 2
  Other, Latin America (n=37,16,4) | 3 | 1 | 0
  Total, Asia (n=1598,1147,171) | 104 | 43 | 5
  Total, Europe (n=1598,1147,171) | 1169 | 834 | 116
  Total, Middle East (n=1598,1147,171) | 264 | 193 | 28
  Total, Latin America (n=1598,1147,171) | 61 | 77 | 22
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.3857, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.2356, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.7993, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.2164, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

60. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Region: Treatment-Experienced
Description: as for outcome 57
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 851 | 730 | 119
participants
  G1, Asia (n=563,574,100) | 87 | 9 | 0
  G1, Europe (n=563,574,100) | 378 | 442 | 74
  G1, Middle East (n=563,574,100) | 59 | 62 | 13
  G1, Latin America (n=563,574,100) | 39 | 61 | 13
  G2, Asia (n=107,27,7) | 61 | 6 | 1
  G2, Europe (n=107,27,7) | 40 | 19 | 4
  G2, Middle East (n=107,27,7) | 3 | 2 | 0
  G2, Latin America (n=107,27,7) | 3 | 0 | 2
  G3, Asia (n=93,65,9) | 12 | 11 | 3
  G3, Europe (n=93,65,9) | 76 | 47 | 5
  G3, Middle East (n=93,65,9) | 1 | 2 | 0
  G3, Latin America (n=93,65,9) | 4 | 5 | 1
  G4, Asia (n=71,43,0) | 0 | 0 | 0
  G4, Europe (n=71,43,0) | 41 | 23 | 0
  G4, Middle East (n=71,43,0) | 29 | 19 | 0
  G4, Latin America (n=71,43,0) | 1 | 1 | 0
  Other, Asia (n=17,21,3) | 4 | 1 | 0
  Other, Europe (n=17,21,3) | 6 | 6 | 0
  Other, Middle East (n=17,21,3) | 5 | 13 | 3
  Other, Latin America (n=17,21,3) | 2 | 1 | 0
  Total, Asia (n=851,730,119) | 164 | 27 | 4
  Total, Europe (n=851,730,119) | 541 | 537 | 83
  Total, Middle East (n=851,730,119) | 97 | 98 | 16
  Total, Latin America (n=851,730,119) | 49 | 68 | 16
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.4820, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.8668, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.2032, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

61. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Country: Treatment-Naive (Table 1 of 2 [G1, G2, G3])
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype was obtained from medical records, and country of study site was documented during intake/enrollment.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category. The table below (G1, G2, G3) is continued onto the subsequent table; thus, the overall number of participants analyzed reflects the total number analyzed among all genotypes (G1, G2, G3, G4, and Other).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  G1, Argentina (n=500,930,272) | 5 | 7 | 4
  G1, Belgium (n=500,930,272) | 15 | 41 | 13
  G1, Chile (n=500,930,272) | 4 | 10 | 4
  G1, Egypt (n=500,930,272) | 0 | 0 | 0
  G1, Estonia (n=500,930,272) | 44 | 70 | 11
  G1, France (n=500,930,272) | 48 | 76 | 16
  G1, Germany (n=500,930,272) | 30 | 54 | 16
  G1, Greece (n=500,930,272) | 22 | 35 | 11
  G1, Italy (n=500,930,272) | 101 | 167 | 59
  G1, Kuwait (n=500,930,272) | 1 | 0 | 0
  G1, Latvia (n=500,930,272) | 5 | 3 | 2
  G1, Lebanon (n=500,930,272) | 4 | 16 | 2
  G1, Lithuania (n=500,930,272) | 16 | 46 | 9
  G1, Macedonia (n=500,930,272) | 12 | 15 | 4
  G1, Mexico (n=500,930,272) | 5 | 13 | 2
  G1, Oman (n=500,930,272) | 2 | 5 | 1
  G1, Pakistan (n=500,930,272) | 4 | 5 | 0
  G1, Peru (n=500,930,272) | 14 | 35 | 12
  G1, Portugal (n=500,930,272) | 11 | 13 | 2
  G1, Qatar (n=500,930,272) | 1 | 1 | 1
  G1, Romania (n=500,930,272) | 60 | 121 | 34
  G1, Taiwan (n=500,930,272) | 12 | 4 | 0
  G1, Turkey (n=500,930,272) | 54 | 138 | 51
  G1, Slovakia (n=500,930,272) | 12 | 13 | 3
  G1, Serbia (n=500,930,272) | 2 | 9 | 2
  G1, Sweden (n=500,930,272) | 5 | 9 | 0
  G1, Switzerland (n=500,930,272) | 5 | 8 | 1
  G1, Syria (n=500,930,272) | 1 | 1 | 0
  G1, United Arab Emirates (n=500,930,272) | 2 | 6 | 2
  G1, Venezuela (n=500,930,272) | 3 | 9 | 10
  G2, Argentina (n=126,160,37) | 0 | 0 | 0
  G2, Belgium (n=126,160,37) | 4 | 4 | 0
  G2, Chile (n=126,160,37) | 0 | 0 | 0
  G2, Egypt (n=126,160,37) | 0 | 0 | 0
  G2, Estonia (n=126,160,37) | 3 | 7 | 1
  G2, France (n=126,160,37) | 4 | 3 | 2
  G2, Germany (n=126,160,37) | 3 | 2 | 0
  G2, Greece (n=126,160,37) | 3 | 3 | 1
  G2, Italy (n=126,160,37) | 81 | 117 | 30
  G2, Kuwait (n=126,160,37) | 0 | 0 | 0
  G2, Latvia (n=126,160,37) | 0 | 1 | 0
  G2, Lebanon (n=126,160,37) | 1 | 1 | 0
  G2, Lithuania (n=126,160,37) | 7 | 6 | 2
  G2, Macedonia (n=126,160,37) | 0 | 0 | 0
  G2, Mexico (n=126,160,37) | 1 | 1 | 1
  G2, Oman (n=126,160,37) | 0 | 0 | 0
  G2, Pakistan (n=126,160,37) | 1 | 1 | 0
  G2, Peru (n=126,160,37) | 0 | 0 | 0
  G2, Portugal (n=126,160,37) | 1 | 0 | 0
  G2, Qatar (n=126,160,37) | 0 | 0 | 0
  G2, Romania (n=126,160,37) | 0 | 0 | 0
  G2, Taiwan (n=126,160,37) | 3 | 1 | 0
  G2, Turkey (n=126,160,37) | 6 | 11 | 0
  G2, Slovakia (n=126,160,37) | 0 | 0 | 0
  G2, Serbia (n=126,160,37) | 0 | 0 | 0
  G2, Sweden (n=126,160,37) | 3 | 1 | 0
  G2, Switzerland (n=126,160,37) | 2 | 0 | 0
  G2, Syria (n=126,160,37) | 0 | 0 | 0
  G2, United Arab Emirates (n=126,160,37) | 0 | 0 | 0
  G2, Venezuela (n=126,160,37) | 3 | 1 | 0
  G3, Argentina (n=232,277,65) | 1 | 0 | 0
  G3, Belgium (n=232,277,65) | 9 | 6 | 1
  G3, Chile (n=232,277,65) | 0 | 0 | 0
  G3, Egypt (n=232,277,65) | 0 | 0 | 0
  G3, Estonia (n=232,277,65) | 27 | 25 | 6
  G3, France (n=232,277,65) | 4 | 14 | 1
  G3, Germany (n=232,277,65) | 7 | 14 | 2
  G3, Greece (n=232,277,65) | 22 | 26 | 10
  G3, Italy (n=232,277,65) | 70 | 70 | 22
  G3, Kuwait (n=232,277,65) | 0 | 1 | 0
  G3, Latvia (n=232,277,65) | 0 | 0 | 0
  G3, Lebanon (n=232,277,65) | 2 | 7 | 0
  G3, Lithuania (n=232,277,65) | 15 | 12 | 4
  G3, Macedonia (n=232,277,65) | 6 | 9 | 0
  G3, Mexico (n=232,277,65) | 0 | 4 | 0
  G3, Oman (n=232,277,65) | 0 | 3 | 2
  G3, Pakistan (n=232,277,65) | 45 | 52 | 8
  G3, Peru (n=232,277,65) | 1 | 0 | 0
  G3, Portugal (n=232,277,65) | 4 | 3 | 2
  G3, Qatar (n=232,277,65) | 0 | 0 | 0
  G3, Romania (n=232,277,65) | 1 | 1 | 0
  G3, Taiwan (n=232,277,65) | 0 | 0 | 0
  G3, Turkey (n=232,277,65) | 5 | 8 | 0
  G3, Slovakia (n=232,277,65) | 2 | 6 | 3
  G3, Serbia (n=232,277,65) | 5 | 5 | 3
  G3, Sweden (n=232,277,65) | 4 | 7 | 0
  G3, Switzerland (n=232,277,65) | 1 | 2 | 1
  G3, Syria (n=232,277,65) | 0 | 0 | 0
  G3, United Arab Emirates (n=232,277,65) | 1 | 1 | 0
  G3, Venezuela (n=232,277,65) | 0 | 1 | 0
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p = 0.0103, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.8373, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.3672, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

62. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Country: Treatment-Naive (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category. The table below (G4, Other, Total) is a continuation of the preceding table; thus, the overall number of participants analyzed reflects the total number analyzed among all genotypes (G1, G2, G3, G4, and Other).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  G4, Argentina (n=92,129,39) | 1 | 3 | 0
  G4, Belgium (n=92,129,39) | 1 | 8 | 4
  G4, Chile (n=92,129,39) | 0 | 0 | 0
  G4, Egypt (n=92,129,39) | 28 | 28 | 2
  G4, Estonia (n=92,129,39) | 0 | 0 | 1
  G4, France (n=92,129,39) | 4 | 11 | 4
  G4, Germany (n=92,129,39) | 0 | 1 | 0
  G4, Greece (n=92,129,39) | 5 | 6 | 1
  G4, Italy (n=92,129,39) | 25 | 33 | 13
  G4, Kuwait (n=92,129,39) | 1 | 4 | 2
  G4, Latvia (n=92,129,39) | 0 | 0 | 0
  G4, Lebanon (n=92,129,39) | 7 | 15 | 2
  G4, Lithuania (n=92,129,39) | 0 | 0 | 0
  G4, Macedonia (n=92,129,39) | 0 | 0 | 0
  G4, Mexico (n=92,129,39) | 0 | 0 | 0
  G4, Oman (n=92,129,39) | 0 | 0 | 0
  G4, Pakistan (n=92,129,39) | 0 | 0 | 0
  G4, Peru (n=92,129,39) | 0 | 0 | 0
  G4, Portugal (n=92,129,39) | 1 | 3 | 2
  G4, Qatar (n=92,129,39) | 0 | 0 | 0
  G4, Romania (n=92,129,39) | 0 | 0 | 0
  G4, Taiwan (n=92,129,39) | 0 | 0 | 0
  G4, Turkey (n=92,129,39) | 4 | 5 | 1
  G4, Slovakia (n=92,129,39) | 0 | 0 | 0
  G4, Serbia (n=92,129,39) | 0 | 2 | 1
  G4, Sweden (n=92,129,39) | 0 | 0 | 0
  G4, Switzerland (n=92,129,39) | 1 | 0 | 1
  G4, Syria (n=92,129,39) | 10 | 7 | 1
  G4, United Arab Emirates (n=92,129,39) | 3 | 3 | 4
  G4, Venezuela (n=92,129,39) | 1 | 0 | 0
  Other, Argentina (n=28,22,7) | 0 | 0 | 0
  Other, Belgium (n=28,22,7) | 4 | 1 | 0
  Other, Chile (n=28,22,7) | 0 | 0 | 0
  Other, Egypt (n=28,22,7) | 0 | 0 | 0
  Other, Estonia (n=28,22,7) | 0 | 0 | 0
  Other, France (n=28,22,7) | 2 | 4 | 1
  Other, Germany (n=28,22,7) | 1 | 0 | 0
  Other, Greece (n=28,22,7) | 0 | 0 | 0
  Other, Italy (n=28,22,7) | 0 | 2 | 1
  Other, Kuwait (n=28,22,7) | 0 | 0 | 0
  Other, Latvia (n=28,22,7) | 0 | 0 | 0
  Other, Lebanon (n=28,22,7) | 0 | 1 | 0
  Other, Lithuania (n=28,22,7) | 0 | 0 | 0
  Other, Macedonia (n=28,22,7) | 0 | 0 | 0
  Other, Mexico (n=28,22,7) | 0 | 0 | 0
  Other, Oman (n=28,22,7) | 0 | 0 | 0
  Other, Pakistan (n=28,22,7) | 0 | 2 | 0
  Other, Peru (n=28,22,7) | 1 | 1 | 0
  Other, Portugal (n=28,22,7) | 0 | 0 | 0
  Other, Qatar (n=28,22,7) | 0 | 0 | 0
  Other, Romania (n=28,22,7) | 0 | 0 | 0
  Other, Taiwan (n=28,22,7) | 13 | 1 | 0
  Other, Turkey (n=28,22,7) | 5 | 10 | 4
  Other, Slovakia (n=28,22,7) | 0 | 0 | 0
  Other, Serbia (n=28,22,7) | 0 | 0 | 0
  Other, Sweden (n=28,22,7) | 0 | 0 | 0
  Other, Switzerland (n=28,22,7) | 1 | 0 | 0
  Other, Syria (n=28,22,7) | 0 | 0 | 0
  Other, United Arab Emirates (n=28,22,7) | 0 | 0 | 0
  Other, Venezuela (n=28,22,7) | 1 | 0 | 1
  Total, Argentina (n=978,1518,420) | 7 | 10 | 4
  Total, Belgium (n=978,1518,420) | 33 | 60 | 18
  Total, Chile (n=978,1518,420) | 4 | 10 | 4
  Total, Egypt (n=978,1518,420) | 28 | 28 | 2
  Total, Estonia (n=978,1518,420) | 74 | 102 | 19
  Total, France (n=978,1518,420) | 62 | 108 | 24
  Total, Germany (n=978,1518,420) | 41 | 71 | 18
  Total, Greece (n=978,1518,420) | 52 | 70 | 23
  Total, Italy (n=978,1518,420) | 277 | 389 | 125
  Total, Kuwait (n=978,1518,420) | 2 | 5 | 2
  Total, Latvia (n=978,1518,420) | 5 | 4 | 2
  Total, Lebanon (n=978,1518,420) | 14 | 40 | 4
  Total, Lithuania (n=978,1518,420) | 38 | 64 | 15
  Total, Macedonia (n=978,1518,420) | 18 | 24 | 4
  Total, Mexico (n=978,1518,420) | 6 | 18 | 3
  Total, Oman (n=978,1518,420) | 2 | 8 | 3
  Total, Pakistan (n=978,1518,420) | 50 | 60 | 8
  Total, Peru (n=978,1518,420) | 16 | 36 | 12
  Total, Portugal (n=978,1518,420) | 17 | 19 | 6
  Total, Qatar (n=978,1518,420) | 1 | 1 | 1
  Total, Romania (n=978,1518,420) | 61 | 122 | 34
  Total, Taiwan (n=978,1518,420) | 28 | 6 | 0
  Total, Turkey (n=978,1518,420) | 74 | 172 | 56
  Total, Slovakia (n=978,1518,420) | 14 | 19 | 6
  Total, Serbia (n=978,1518,420) | 7 | 16 | 6
  Total, Sweden (n=978,1518,420) | 12 | 17 | 0
  Total, Switzerland (n=978,1518,420) | 10 | 10 | 3
  Total, Syria (n=978,1518,420) | 11 | 8 | 1
  Total, United Arab Emirates (n=978,1518,420) | 6 | 10 | 6
  Total, Venezuela (n=978,1518,420) | 8 | 11 | 11
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0637, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.0474, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

63. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Country: Treatment-Experienced (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced); n = number of participants analyzed within each HCV RNA genotype category. The table below (G1, G2, G3) is continued onto the subsequent table; thus, the overall number of participants analyzed reflects the total number analyzed among all genotypes (G1, G2, G3, G4, and Other).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  G1, Argentina (n=295,703,239) | 4 | 9 | 0
  G1, Belgium (n=295,703,239) | 14 | 37 | 9
  G1, Chile (n=295,703,239) | 7 | 16 | 3
  G1, Egypt (n=295,703,239) | 0 | 1 | 0
  G1, Estonia (n=295,703,239) | 3 | 2 | 2
  G1, France (n=295,703,239) | 41 | 125 | 44
  G1, Germany (n=295,703,239) | 16 | 36 | 17
  G1, Greece (n=295,703,239) | 4 | 18 | 7
  G1, Italy (n=295,703,239) | 40 | 117 | 46
  G1, Kuwait (n=295,703,239) | 0 | 0 | 0
  G1, Latvia (n=295,703,239) | 6 | 41 | 15
  G1, Lebanon (n=295,703,239) | 2 | 14 | 4
  G1, Lithuania (n=295,703,239) | 8 | 43 | 9
  G1, Macedonia (n=295,703,239) | 0 | 0 | 0
  G1, Mexico (n=295,703,239) | 3 | 18 | 6
  G1, Oman (n=295,703,239) | 1 | 5 | 0
  G1, Pakistan (n=295,703,239) | 2 | 2 | 0
  G1, Peru (n=295,703,239) | 5 | 18 | 7
  G1, Portugal (n=295,703,239) | 13 | 17 | 8
  G1, Qatar (n=295,703,239) | 2 | 3 | 2
  G1, Romania (n=295,703,239) | 23 | 80 | 25
  G1, Taiwan (n=295,703,239) | 81 | 11 | 0
  G1, Turkey (n=295,703,239) | 12 | 59 | 23
  G1, Slovakia (n=295,703,239) | 2 | 13 | 2
  G1, Serbia (n=295,703,239) | 0 | 0 | 0
  G1, Sweden (n=295,703,239) | 2 | 1 | 0
  G1, Switzerland (n=295,703,239) | 2 | 4 | 2
  G1, Syria (n=295,703,239) | 0 | 0 | 0
  G1, United Arab Emirates (n=295,703,239) | 0 | 5 | 1
  G1, Venezuela (n=295,703,239) | 2 | 8 | 7
  G2, Argentina (n=92,38,11) | 0 | 0 | 0
  G2, Belgium (n=92,38,11) | 0 | 0 | 0
  G2, Chile (n=92,38,11) | 0 | 0 | 0
  G2, Egypt (n=92,38,11) | 0 | 0 | 0
  G2, Estonia (n=92,38,11) | 0 | 0 | 0
  G2, France (n=92,38,11) | 9 | 9 | 2
  G2, Germany (n=92,38,11) | 0 | 0 | 0
  G2, Greece (n=92,38,11) | 0 | 1 | 0
  G2, Italy (n=92,38,11) | 18 | 16 | 3
  G2, Kuwait (n=92,38,11) | 0 | 0 | 0
  G2, Latvia (n=92,38,11) | 0 | 2 | 0
  G2, Lebanon (n=92,38,11) | 0 | 0 | 0
  G2, Lithuania (n=92,38,11) | 2 | 0 | 1
  G2, Macedonia (n=92,38,11) | 0 | 0 | 0
  G2, Mexico (n=92,38,11) | 1 | 1 | 1
  G2, Oman (n=92,38,11) | 0 | 0 | 0
  G2, Pakistan (n=92,38,11) | 0 | 0 | 0
  G2, Peru (n=92,38,11) | 0 | 0 | 0
  G2, Portugal (n=92,38,11) | 0 | 0 | 0
  G2, Qatar (n=92,38,11) | 0 | 0 | 0
  G2, Romania (n=92,38,11) | 0 | 0 | 0
  G2, Taiwan (n=92,38,11) | 59 | 8 | 1
  G2, Turkey (n=92,38,11) | 2 | 1 | 2
  G2, Slovakia (n=92,38,11) | 0 | 0 | 0
  G2, Serbia (n=92,38,11) | 0 | 0 | 0
  G2, Sweden (n=92,38,11) | 0 | 0 | 0
  G2, Switzerland (n=92,38,11) | 0 | 0 | 0
  G2, Syria (n=92,38,11) | 0 | 0 | 0
  G2, United Arab Emirates (n=92,38,11) | 0 | 0 | 0
  G2, Venezuela (n=92,38,11) | 1 | 0 | 1
  G3, Argentina (n=63,84,20) | 1 | 3 | 0
  G3, Belgium (n=63,84,20) | 3 | 4 | 2
  G3, Chile (n=63,84,20) | 1 | 2 | 1
  G3, Egypt (n=63,84,20) | 0 | 0 | 0
  G3, Estonia (n=63,84,20) | 0 | 0 | 0
  G3, France (n=63,84,20) | 12 | 13 | 2
  G3, Germany (n=63,84,20) | 3 | 4 | 0
  G3, Greece (n=63,84,20) | 2 | 5 | 1
  G3, Italy (n=63,84,20) | 15 | 14 | 5
  G3, Kuwait (n=63,84,20) | 0 | 0 | 0
  G3, Latvia (n=63,84,20) | 0 | 0 | 0
  G3, Lebanon (n=63,84,20) | 0 | 1 | 0
  G3, Lithuania (n=63,84,20) | 5 | 14 | 1
  G3, Macedonia (n=63,84,20) | 0 | 1 | 0
  G3, Mexico (n=63,84,20) | 0 | 1 | 0
  G3, Oman (n=63,84,20) | 0 | 0 | 0
  G3, Pakistan (n=63,84,20) | 8 | 14 | 3
  G3, Peru (n=63,84,20) | 0 | 0 | 0
  G3, Portugal (n=63,84,20) | 11 | 4 | 3
  G3, Qatar (n=63,84,20) | 0 | 0 | 0
  G3, Romania (n=63,84,20) | 0 | 0 | 0
  G3, Taiwan (n=63,84,20) | 1 | 0 | 0
  G3, Turkey (n=63,84,20) | 0 | 1 | 0
  G3, Slovakia (n=63,84,20) | 1 | 2 | 0
  G3, Serbia (n=63,84,20) | 0 | 0 | 0
  G3, Sweden (n=63,84,20) | 0 | 0 | 1
  G3, Switzerland (n=63,84,20) | 0 | 0 | 0
  G3, Syria (n=63,84,20) | 0 | 0 | 0
  G3, United Arab Emirates (n=63,84,20) | 0 | 1 | 0
  G3, Venezuela (n=63,84,20) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.5522, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

64. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by HCV RNA Genotype and Country: Treatment-Experienced (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced); n = number of participants analyzed within each HCV RNA genotype category. The table below (G4, Other, Total) is a continuation of the preceding table; thus, the overall number of participants analyzed reflects the total number analyzed among all genotypes (G1, G2, G3, G4, and Other).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  G4, Argentina (n=26,67,21) | 0 | 1 | 0
  G4, Belgium (n=26,67,21) | 1 | 4 | 6
  G4, Chile (n=26,67,21) | 0 | 1 | 0
  G4, Egypt (n=26,67,21) | 10 | 25 | 6
  G4, Estonia (n=26,67,21) | 0 | 0 | 0
  G4, France (n=26,67,21) | 4 | 13 | 5
  G4, Germany (n=26,67,21) | 2 | 1 | 0
  G4, Greece (n=26,67,21) | 1 | 3 | 0
  G4, Italy (n=26,67,21) | 3 | 9 | 2
  G4, Kuwait (n=26,67,21) | 0 | 0 | 0
  G4, Latvia (n=26,67,21) | 0 | 0 | 0
  G4, Lebanon (n=26,67,21) | 1 | 3 | 1
  G4, Lithuania (n=26,67,21) | 0 | 0 | 0
  G4, Macedonia (n=26,67,21) | 0 | 0 | 0
  G4, Mexico (n=26,67,21) | 0 | 0 | 0
  G4, Oman (n=26,67,21) | 0 | 0 | 0
  G4, Pakistan (n=26,67,21) | 0 | 0 | 0
  G4, Peru (n=26,67,21) | 0 | 0 | 0
  G4, Portugal (n=26,67,21) | 3 | 6 | 1
  G4, Qatar (n=26,67,21) | 0 | 0 | 0
  G4, Romania (n=26,67,21) | 0 | 0 | 0
  G4, Taiwan (n=26,67,21) | 0 | 0 | 0
  G4, Turkey (n=26,67,21) | 1 | 0 | 0
  G4, Slovakia (n=26,67,21) | 0 | 0 | 0
  G4, Serbia (n=26,67,21) | 0 | 0 | 0
  G4, Sweden (n=26,67,21) | 0 | 0 | 0
  G4, Switzerland (n=26,67,21) | 0 | 0 | 0
  G4, Syria (n=26,67,21) | 0 | 0 | 0
  G4, United Arab Emirates (n=26,67,21) | 0 | 1 | 0
  G4, Venezuela (n=26,67,21) | 0 | 0 | 0
  Other, Argentina (n=14,22,5) | 0 | 0 | 0
  Other, Belgium (n=14,22,5) | 3 | 2 | 0
  Other, Chile (n=14,22,5) | 0 | 0 | 0
  Other, Egypt (n=14,22,5) | 0 | 0 | 0
  Other, Estonia (n=14,22,5) | 0 | 0 | 0
  Other, France (n=14,22,5) | 2 | 2 | 1
  Other, Germany (n=14,22,5) | 0 | 0 | 0
  Other, Greece (n=14,22,5) | 0 | 0 | 0
  Other, Italy (n=14,22,5) | 0 | 1 | 0
  Other, Kuwait (n=14,22,5) | 0 | 0 | 0
  Other, Latvia (n=14,22,5) | 0 | 0 | 0
  Other, Lebanon (n=14,22,5) | 0 | 0 | 0
  Other, Lithuania (n=14,22,5) | 0 | 0 | 0
  Other, Macedonia (n=14,22,5) | 0 | 0 | 0
  Other, Mexico (n=14,22,5) | 0 | 0 | 0
  Other, Oman (n=14,22,5) | 0 | 1 | 0
  Other, Pakistan (n=14,22,5) | 1 | 1 | 0
  Other, Peru (n=14,22,5) | 1 | 1 | 0
  Other, Portugal (n=14,22,5) | 1 | 0 | 0
  Other, Qatar (n=14,22,5) | 0 | 0 | 0
  Other, Romania (n=14,22,5) | 0 | 0 | 0
  Other, Taiwan (n=14,22,5) | 3 | 0 | 0
  Other, Turkey (n=14,22,5) | 2 | 14 | 4
  Other, Slovakia (n=14,22,5) | 0 | 0 | 0
  Other, Serbia (n=14,22,5) | 0 | 0 | 0
  Other, Sweden (n=14,22,5) | 0 | 0 | 0
  Other, Switzerland (n=14,22,5) | 0 | 0 | 0
  Other, Syria (n=14,22,5) | 0 | 0 | 0
  Other, United Arab Emirates (n=14,22,5) | 0 | 0 | 0
  Other, Venezuela (n=14,22,5) | 1 | 0 | 0
  Total, Argentina (n=490,914,296) | 5 | 13 | 0
  Total, Belgium (n=490,914,296) | 21 | 47 | 17
  Total, Chile (n=490,914,296) | 8 | 19 | 4
  Total, Egypt (n=490,914,296) | 10 | 26 | 6
  Total, Estonia (n=490,914,296) | 3 | 2 | 2
  Total, France (n=490,914,296) | 68 | 162 | 54
  Total, Germany (n=490,914,296) | 21 | 41 | 17
  Total, Greece (n=490,914,296) | 7 | 27 | 8
  Total, Italy (n=490,914,296) | 76 | 157 | 56
  Total, Kuwait (n=490,914,296) | 0 | 0 | 0
  Total, Latvia (n=490,914,296) | 6 | 43 | 15
  Total, Lebanon (n=490,914,296) | 3 | 18 | 5
  Total, Lithuania (n=490,914,296) | 15 | 57 | 11
  Total, Macedonia (n=490,914,296) | 0 | 1 | 0
  Total, Mexico (n=490,914,296) | 4 | 20 | 8
  Total, Oman (n=490,914,296) | 1 | 6 | 0
  Total, Pakistan (n=490,914,296) | 11 | 17 | 3
  Total, Peru (n=490,914,296) | 6 | 19 | 7
  Total, Portugal (n=490,914,296) | 28 | 27 | 12
  Total, Qatar (n=490,914,296) | 2 | 3 | 2
  Total, Romania (n=490,914,296) | 23 | 80 | 25
  Total, Taiwan (n=490,914,296) | 144 | 19 | 1
  Total, Turkey (n=490,914,296) | 17 | 75 | 29
  Total, Slovakia (n=490,914,296) | 3 | 15 | 2
  Total, Serbia (n=490,914,296) | 0 | 0 | 0
  Total, Sweden (n=490,914,296) | 2 | 1 | 1
  Total, Switzerland (n=490,914,296) | 2 | 4 | 2
  Total, Syria (n=490,914,296) | 0 | 0 | 0
  Total, United Arab Emirates (n=490,914,296) | 0 | 7 | 1
  Total, Venezuela (n=490,914,296) | 4 | 8 | 8
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.5117, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Other genotypes; Test type: Superiority or Other; p = 0.3437, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

65. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Country: Treatment-Naive (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: as for outcome 61
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1598 | 1147 | 171
participants
  G1, Argentina (n=837,747,118) | 7 | 7 | 2
  G1, Belgium (n=837,747,118) | 32 | 32 | 5
  G1, Chile (n=837,747,118) | 9 | 8 | 1
  G1, Egypt (n=837,747,118) | 0 | 0 | 0
  G1, Estonia (n=837,747,118) | 62 | 58 | 5
  G1, France (n=837,747,118) | 82 | 53 | 5
  G1, Germany (n=837,747,118) | 50 | 45 | 5
  G1, Greece (n=837,747,118) | 35 | 29 | 4
  G1, Italy (n=837,747,118) | 160 | 139 | 28
  G1, Kuwait (n=837,747,118) | 1 | 0 | 0
  G1, Latvia (n=837,747,118) | 6 | 4 | 0
  G1, Lebanon (n=837,747,118) | 13 | 8 | 1
  G1, Lithuania (n=837,747,118) | 37 | 32 | 2
  G1, Macedonia (n=837,747,118) | 18 | 10 | 3
  G1, Mexico (n=837,747,118) | 5 | 13 | 2
  G1, Oman (n=837,747,118) | 5 | 3 | 0
  G1, Pakistan (n=837,747,118) | 7 | 2 | 0
  G1, Peru (n=837,747,118) | 20 | 31 | 10
  G1, Portugal (n=837,747,118) | 19 | 6 | 1
  G1, Qatar (n=837,747,118) | 2 | 0 | 1
  G1, Romania (n=837,747,118) | 97 | 102 | 16
  G1, Taiwan (n=837,747,118) | 12 | 4 | 0
  G1, Turkey (n=837,747,118) | 110 | 115 | 18
  G1, Slovakia (n=837,747,118) | 15 | 12 | 1
  G1, Serbia (n=837,747,118) | 6 | 6 | 1
  G1, Sweden (n=837,747,118) | 8 | 6 | 0
  G1, Switzerland (n=837,747,118) | 5 | 9 | 0
  G1, Syria (n=837,747,118) | 1 | 1 | 0
  G1, United Arab Emirates (n=837,747,118) | 6 | 3 | 1
  G1, Venezuela (n=837,747,118) | 7 | 9 | 6
  G2, Argentina (n=198,113,12) | 0 | 0 | 0
  G2, Belgium (n=198,113,12) | 6 | 2 | 0
  G2, Chile (n=198,113,12) | 0 | 0 | 0
  G2, Egypt (n=198,113,12) | 0 | 0 | 0
  G2, Estonia (n=198,113,12) | 7 | 4 | 0
  G2, France (n=198,113,12) | 7 | 1 | 1
  G2, Germany (n=198,113,12) | 5 | 0 | 0
  G2, Greece (n=198,113,12) | 5 | 2 | 0
  G2, Italy (n=198,113,12) | 128 | 91 | 9
  G2, Kuwait (n=198,113,12) | 0 | 0 | 0
  G2, Latvia (n=198,113,12) | 1 | 0 | 0
  G2, Lebanon (n=198,113,12) | 2 | 0 | 0
  G2, Lithuania (n=198,113,12) | 9 | 5 | 1
  G2, Macedonia (n=198,113,12) | 0 | 0 | 0
  G2, Mexico (n=198,113,12) | 1 | 1 | 1
  G2, Oman (n=198,113,12) | 0 | 0 | 0
  G2, Pakistan (n=198,113,12) | 1 | 1 | 0
  G2, Peru (n=198,113,12) | 0 | 0 | 0
  G2, Portugal (n=198,113,12) | 1 | 0 | 0
  G2, Qatar (n=198,113,12) | 0 | 0 | 0
  G2, Romania (n=198,113,12) | 0 | 0 | 0
  G2, Taiwan (n=198,113,12) | 3 | 1 | 0
  G2, Turkey (n=198,113,12) | 13 | 4 | 0
  G2, Slovakia (n=198,113,12) | 0 | 0 | 0
  G2, Serbia (n=198,113,12) | 0 | 0 | 0
  G2, Sweden (n=198,113,12) | 3 | 1 | 0
  G2, Switzerland (n=198,113,12) | 2 | 0 | 0
  G2, Syria (n=198,113,12) | 0 | 0 | 0
  G2, United Arab Emirates (n=198,113,12) | 0 | 0 | 0
  G2, Venezuela (n=198,113,12) | 4 | 0 | 0
  G3, Argentina (n=361,186,27) | 1 | 0 | 0
  G3, Belgium (n=361,186,27) | 10 | 6 | 0
  G3, Chile (n=361,186,27) | 0 | 0 | 0
  G3, Egypt (n=361,186,27) | 0 | 0 | 0
  G3, Estonia (n=361,186,27) | 36 | 22 | 0
  G3, France (n=361,186,27) | 8 | 10 | 1
  G3, Germany (n=361,186,27) | 13 | 10 | 0
  G3, Greece (n=361,186,27) | 34 | 21 | 3
  G3, Italy (n=361,186,27) | 109 | 43 | 10
  G3, Kuwait (n=361,186,27) | 0 | 1 | 0
  G3, Latvia (n=361,186,27) | 0 | 0 | 0
  G3, Lebanon (n=361,186,27) | 4 | 5 | 0
  G3, Lithuania (n=361,186,27) | 22 | 7 | 2
  G3, Macedonia (n=361,186,27) | 12 | 3 | 0
  G3, Mexico (n=361,186,27) | 0 | 4 | 0
  G3, Oman (n=361,186,27) | 2 | 3 | 0
  G3, Pakistan (n=361,186,27) | 67 | 33 | 5
  G3, Peru (n=361,186,27) | 1 | 0 | 0
  G3, Portugal (n=361,186,27) | 4 | 4 | 1
  G3, Qatar (n=361,186,27) | 0 | 0 | 0
  G3, Romania (n=361,186,27) | 2 | 0 | 0
  G3, Taiwan (n=361,186,27) | 0 | 0 | 0
  G3, Turkey (n=361,186,27) | 9 | 4 | 0
  G3, Slovakia (n=361,186,27) | 4 | 5 | 2
  G3, Serbia (n=361,186,27) | 9 | 2 | 2
  G3, Sweden (n=361,186,27) | 10 | 1 | 0
  G3, Switzerland (n=361,186,27) | 2 | 1 | 1
  G3, Syria (n=361,186,27) | 0 | 0 | 0
  G3, United Arab Emirates (n=361,186,27) | 2 | 0 | 0
  G3, Venezuela (n=361,186,27) | 0 | 1 | 0
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p = 0.0381, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.6852, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.1185, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

66. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Country: Treatment-Naive (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: as for outcome 62
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs8099917 TT | Naive: IL28B rs8099917 TG | Naive: IL28B rs8099917 GG
Number analyzed (Participants) | 1598 | 1147 | 171
participants
  G4, Argentina (n=165,85,10) | 2 | 2 | 0
  G4, Belgium (n=165,85,10) | 9 | 4 | 0
  G4, Chile (n=165,85,10) | 0 | 0 | 0
  G4, Egypt (n=165,85,10) | 41 | 16 | 1
  G4, Estonia (n=165,85,10) | 0 | 1 | 0
  G4, France (n=165,85,10) | 10 | 9 | 0
  G4, Germany (n=165,85,10) | 1 | 0 | 0
  G4, Greece (n=165,85,10) | 6 | 4 | 2
  G4, Italy (n=165,85,10) | 47 | 21 | 3
  G4, Kuwait (n=165,85,10) | 4 | 3 | 0
  G4, Latvia (n=165,85,10) | 0 | 0 | 0
  G4, Lebanon (n=165,85,10) | 13 | 9 | 2
  G4, Lithuania (n=165,85,10) | 0 | 0 | 0
  G4, Macedonia (n=165,85,10) | 0 | 0 | 0
  G4, Mexico (n=165,85,10) | 0 | 0 | 0
  G4, Oman (n=165,85,10) | 0 | 0 | 0
  G4, Pakistan (n=165,85,10) | 0 | 0 | 0
  G4, Peru (n=165,85,10) | 0 | 0 | 0
  G4, Portugal (n=165,85,10) | 3 | 3 | 0
  G4, Qatar (n=165,85,10) | 0 | 0 | 0
  G4, Romania (n=165,85,10) | 0 | 0 | 0
  G4, Taiwan (n=165,85,10) | 0 | 0 | 0
  G4, Turkey (n=165,85,10) | 9 | 1 | 0
  G4, Slovakia (n=165,85,10) | 0 | 0 | 0
  G4, Serbia (n=165,85,10) | 0 | 3 | 0
  G4, Sweden (n=165,85,10) | 0 | 0 | 0
  G4, Switzerland (n=165,85,10) | 1 | 1 | 0
  G4, Syria (n=165,85,10) | 14 | 4 | 0
  G4, United Arab Emirates (n=165,85,10) | 4 | 4 | 2
  G4, Venezuela (n=165,85,10) | 1 | 0 | 0
  Other, Argentina (n=37,16,4) | 0 | 0 | 0
  Other, Belgium (n=37,16,4) | 4 | 1 | 0
  Other, Chile (n=37,16,4) | 0 | 0 | 0
  Other, Egypt (n=37,16,4) | 0 | 0 | 0
  Other, Estonia (n=37,16,4) | 0 | 0 | 0
  Other, France (n=37,16,4) | 4 | 2 | 1
  Other, Germany (n=37,16,4) | 1 | 0 | 0
  Other, Greece (n=37,16,4) | 0 | 0 | 0
  Other, Italy (n=37,16,4) | 1 | 1 | 1
  Other, Kuwait (n=37,16,4) | 0 | 0 | 0
  Other, Latvia (n=37,16,4) | 0 | 0 | 0
  Other, Lebanon (n=37,16,4) | 1 | 0 | 0
  Other, Lithuania (n=37,16,4) | 0 | 0 | 0
  Other, Macedonia (n=37,16,4) | 0 | 0 | 0
  Other, Mexico (n=37,16,4) | 0 | 0 | 0
  Other, Oman (n=37,16,4) | 0 | 0 | 0
  Other, Pakistan (n=37,16,4) | 1 | 1 | 0
  Other, Peru (n=37,16,4) | 2 | 0 | 0
  Other, Portugal (n=37,16,4) | 0 | 0 | 0
  Other, Qatar (n=37,16,4) | 0 | 0 | 0
  Other, Romania (n=37,16,4) | 0 | 0 | 0
  Other, Taiwan (n=37,16,4) | 13 | 1 | 0
  Other, Turkey (n=37,16,4) | 8 | 9 | 2
  Other, Slovakia (n=37,16,4) | 0 | 0 | 0
  Other, Serbia (n=37,16,4) | 0 | 0 | 0
  Other, Sweden (n=37,16,4) | 0 | 0 | 0
  Other, Switzerland (n=37,16,4) | 1 | 0 | 0
  Other, Syria (n=37,16,4) | 0 | 0 | 0
  Other, United Arab Emirates (n=37,16,4) | 0 | 0 | 0
  Other, Venezuela (n=37,16,4) | 1 | 1 | 0
  Total, Argentina (n=1598,1147,171) | 10 | 9 | 2
  Total, Belgium (n=1598,1147,171) | 61 | 45 | 5
  Total, Chile (n=1598,1147,171) | 9 | 8 | 1
  Total, Egypt (n=1598,1147,171) | 41 | 16 | 1
  Total, Estonia (n=1598,1147,171) | 105 | 85 | 5
  Total, France (n=1598,1147,171) | 111 | 75 | 8
  Total, Germany (n=1598,1147,171) | 70 | 55 | 5
  Total, Greece (n=1598,1147,171) | 80 | 56 | 9
  Total, Italy (n=1598,1147,171) | 445 | 295 | 51
  Total, Kuwait (n=1598,1147,171) | 5 | 4 | 0
  Total, Latvia (n=1598,1147,171) | 7 | 4 | 0
  Total, Lebanon (n=1598,1147,171) | 33 | 22 | 3
  Total, Lithuania (n=1598,1147,171) | 68 | 44 | 5
  Total, Macedonia (n=1598,1147,171) | 30 | 13 | 3
  Total, Mexico (n=1598,1147,171) | 6 | 18 | 3
  Total, Oman (n=1598,1147,171) | 7 | 6 | 0
  Total, Pakistan (n=1598,1147,171) | 76 | 37 | 5
  Total, Peru (n=1598,1147,171) | 23 | 31 | 10
  Total, Portugal (n=1598,1147,171) | 27 | 13 | 2
  Total, Qatar (n=1598,1147,171) | 2 | 0 | 1
  Total, Romania (n=1598,1147,171) | 99 | 102 | 16
  Total, Taiwan (n=1598,1147,171) | 28 | 6 | 0
  Total, Turkey (n=1598,1147,171) | 149 | 133 | 20
  Total, Slovakia (n=1598,1147,171) | 19 | 17 | 3
  Total, Serbia (n=1598,1147,171) | 15 | 11 | 3
  Total, Sweden (n=1598,1147,171) | 21 | 8 | 0
  Total, Switzerland (n=1598,1147,171) | 11 | 11 | 1
  Total, Syria (n=1598,1147,171) | 15 | 5 | 0
  Total, United Arab Emirates (n=1598,1147,171) | 12 | 7 | 3
  Total, Venezuela (n=1598,1147,171) | 13 | 11 | 6
Statistical Analysis 1: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.2611, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.6059, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: IL28B rs8099917 TT vs Naive: IL28B rs8099917 TG vs Naive: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p = 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

67. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Country: Treatment-Experienced (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: as for outcome 63
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 851 | 730 | 119
participants
  G1, Argentina (n=563,574,100) | 6 | 7 | 0
  G1, Belgium (n=563,574,100) | 28 | 27 | 5
  G1, Chile (n=563,574,100) | 11 | 13 | 2
  G1, Egypt (n=563,574,100) | 0 | 1 | 0
  G1, Estonia (n=563,574,100) | 4 | 2 | 1
  G1, France (n=563,574,100) | 80 | 117 | 13
  G1, Germany (n=563,574,100) | 33 | 29 | 7
  G1, Greece (n=563,574,100) | 11 | 14 | 4
  G1, Italy (n=563,574,100) | 88 | 98 | 17
  G1, Kuwait (n=563,574,100) | 0 | 0 | 0
  G1, Latvia (n=563,574,100) | 22 | 33 | 7
  G1, Lebanon (n=563,574,100) | 9 | 9 | 2
  G1, Lithuania (n=563,574,100) | 27 | 30 | 3
  G1, Macedonia (n=563,574,100) | 0 | 0 | 0
  G1, Mexico (n=563,574,100) | 6 | 17 | 4
  G1, Oman (n=563,574,100) | 5 | 1 | 0
  G1, Pakistan (n=563,574,100) | 3 | 1 | 0
  G1, Peru (n=563,574,100) | 8 | 16 | 6
  G1, Portugal (n=563,574,100) | 23 | 11 | 4
  G1, Qatar (n=563,574,100) | 5 | 2 | 0
  G1, Romania (n=563,574,100) | 51 | 66 | 11
  G1, Taiwan (n=563,574,100) | 84 | 8 | 0
  G1, Turkey (n=563,574,100) | 37 | 46 | 11
  G1, Slovakia (n=563,574,100) | 7 | 9 | 1
  G1, Serbia (n=563,574,100) | 0 | 0 | 0
  G1, Sweden (n=563,574,100) | 2 | 1 | 0
  G1, Switzerland (n=563,574,100) | 2 | 5 | 1
  G1, Syria (n=563,574,100) | 0 | 0 | 0
  G1, United Arab Emirates (n=563,574,100) | 3 | 3 | 0
  G1, Venezuela (n=563,574,100) | 8 | 8 | 1
  G2, Argentina (n=107,27,7) | 0 | 0 | 0
  G2, Belgium (n=107,27,7) | 0 | 0 | 0
  G2, Chile (n=107,27,7) | 0 | 0 | 0
  G2, Egypt (n=107,27,7) | 0 | 0 | 0
  G2, Estonia (n=107,27,7) | 0 | 0 | 0
  G2, France (n=107,27,7) | 15 | 4 | 1
  G2, Germany (n=107,27,7) | 0 | 0 | 0
  G2, Greece (n=107,27,7) | 0 | 1 | 0
  G2, Italy (n=107,27,7) | 22 | 12 | 3
  G2, Kuwait (n=107,27,7) | 0 | 0 | 0
  G2, Latvia (n=107,27,7) | 1 | 1 | 0
  G2, Lebanon (n=107,27,7) | 0 | 0 | 0
  G2, Lithuania (n=107,27,7) | 2 | 1 | 0
  G2, Macedonia (n=107,27,7) | 0 | 0 | 0
  G2, Mexico (n=107,27,7) | 2 | 0 | 1
  G2, Oman (n=107,27,7) | 0 | 0 | 0
  G2, Pakistan (n=107,27,7) | 0 | 0 | 0
  G2, Peru (n=107,27,7) | 0 | 0 | 0
  G2, Portugal (n=107,27,7) | 0 | 0 | 0
  G2, Qatar (n=107,27,7) | 0 | 0 | 0
  G2, Romania (n=107,27,7) | 0 | 0 | 0
  G2, Taiwan (n=107,27,7) | 61 | 6 | 1
  G2, Turkey (n=107,27,7) | 3 | 2 | 0
  G2, Slovakia (n=107,27,7) | 0 | 0 | 0
  G2, Serbia (n=107,27,7) | 0 | 0 | 0
  G2, Sweden (n=107,27,7) | 0 | 0 | 0
  G2, Switzerland (n=107,27,7) | 0 | 0 | 0
  G2, Syria (n=107,27,7) | 0 | 0 | 0
  G2, United Arab Emirates (n=107,27,7) | 0 | 0 | 0
  G2, Venezuela (n=107,27,7) | 1 | 0 | 1
  G3, Argentina (n=93,65,9) | 2 | 2 | 0
  G3, Belgium (n=93,65,9) | 4 | 3 | 2
  G3, Chile (n=93,65,9) | 2 | 1 | 1
  G3, Egypt (n=93,65,9) | 0 | 0 | 0
  G3, Estonia (n=93,65,9) | 0 | 0 | 0
  G3, France (n=93,65,9) | 18 | 9 | 0
  G3, Germany (n=93,65,9) | 4 | 3 | 0
  G3, Greece (n=93,65,9) | 2 | 6 | 0
  G3, Italy (n=93,65,9) | 22 | 11 | 1
  G3, Kuwait (n=93,65,9) | 0 | 0 | 0
  G3, Latvia (n=93,65,9) | 0 | 0 | 0
  G3, Lebanon (n=93,65,9) | 0 | 1 | 0
  G3, Lithuania (n=93,65,9) | 11 | 8 | 1
  G3, Macedonia (n=93,65,9) | 1 | 0 | 0
  G3, Mexico (n=93,65,9) | 0 | 2 | 0
  G3, Oman (n=93,65,9) | 0 | 0 | 0
  G3, Pakistan (n=93,65,9) | 11 | 11 | 3
  G3, Peru (n=93,65,9) | 0 | 0 | 0
  G3, Portugal (n=93,65,9) | 13 | 4 | 1
  G3, Qatar (n=93,65,9) | 0 | 0 | 0
  G3, Romania (n=93,65,9) | 0 | 0 | 0
  G3, Taiwan (n=93,65,9) | 1 | 0 | 0
  G3, Turkey (n=93,65,9) | 1 | 0 | 0
  G3, Slovakia (n=93,65,9) | 1 | 2 | 0
  G3, Serbia (n=93,65,9) | 0 | 0 | 0
  G3, Sweden (n=93,65,9) | 0 | 1 | 0
  G3, Switzerland (n=93,65,9) | 0 | 0 | 0
  G3, Syria (n=93,65,9) | 0 | 0 | 0
  G3, United Arab Emirates (n=93,65,9) | 0 | 1 | 0
  G3, Venezuela (n=93,65,9) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0048, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.5127, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

68. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by HCV RNA Genotype and Country: Treatment-Experienced (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 61
Time Frame: Study Visit 1
Population: as for outcome 64
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 851 | 730 | 119
participants
  G4, Argentina (n=71,43,0) | 1 | 0 | 0
  G4, Belgium (n=71,43,0) | 10 | 1 | 0
  G4, Chile (n=71,43,0) | 0 | 1 | 0
  G4, Egypt (n=71,43,0) | 26 | 15 | 0
  G4, Estonia (n=71,43,0) | 0 | 0 | 0
  G4, France (n=71,43,0) | 14 | 8 | 0
  G4, Germany (n=71,43,0) | 2 | 1 | 0
  G4, Greece (n=71,43,0) | 2 | 2 | 0
  G4, Italy (n=71,43,0) | 8 | 6 | 0
  G4, Kuwait (n=71,43,0) | 0 | 0 | 0
  G4, Latvia (n=71,43,0) | 0 | 0 | 0
  G4, Lebanon (n=71,43,0) | 1 | 4 | 0
  G4, Lithuania (n=71,43,0) | 0 | 0 | 0
  G4, Macedonia (n=71,43,0) | 0 | 0 | 0
  G4, Mexico (n=71,43,0) | 0 | 0 | 0
  G4, Oman (n=71,43,0) | 0 | 0 | 0
  G4, Pakistan (n=71,43,0) | 0 | 0 | 0
  G4, Peru (n=71,43,0) | 0 | 0 | 0
  G4, Portugal (n=71,43,0) | 5 | 5 | 0
  G4, Qatar (n=71,43,0) | 0 | 0 | 0
  G4, Romania (n=71,43,0) | 0 | 0 | 0
  G4, Taiwan (n=71,43,0) | 0 | 0 | 0
  G4, Turkey (n=71,43,0) | 1 | 0 | 0
  G4, Slovakia (n=71,43,0) | 0 | 0 | 0
  G4, Serbia (n=71,43,0) | 0 | 0 | 0
  G4, Sweden (n=71,43,0) | 0 | 0 | 0
  G4, Switzerland (n=71,43,0) | 0 | 0 | 0
  G4, Syria (n=71,43,0) | 0 | 0 | 0
  G4, United Arab Emirates (n=71,43,0) | 1 | 0 | 0
  G4, Venezuela (n=71,43,0) | 0 | 0 | 0
  Other, Argentina (n=17,21,3) | 0 | 0 | 0
  Other, Belgium (n=17,21,3) | 3 | 2 | 0
  Other, Chile (n=17,21,3) | 0 | 0 | 0
  Other, Egypt (n=17,21,3) | 0 | 0 | 0
  Other, Estonia (n=17,21,3) | 0 | 0 | 0
  Other, France (n=17,21,3) | 2 | 3 | 0
  Other, Germany (n=17,21,3) | 0 | 0 | 0
  Other, Greece (n=17,21,3) | 0 | 0 | 0
  Other, Italy (n=17,21,3) | 0 | 1 | 0
  Other, Kuwait (n=17,21,3) | 0 | 0 | 0
  Other, Latvia (n=17,21,3) | 0 | 0 | 0
  Other, Lebanon (n=17,21,3) | 0 | 0 | 0
  Other, Lithuania (n=17,21,3) | 0 | 0 | 0
  Other, Macedonia (n=17,21,3) | 0 | 0 | 0
  Other, Mexico (n=17,21,3) | 0 | 0 | 0
  Other, Oman (n=17,21,3) | 0 | 1 | 0
  Other, Pakistan (n=17,21,3) | 1 | 1 | 0
  Other, Peru (n=17,21,3) | 1 | 1 | 0
  Other, Portugal (n=17,21,3) | 1 | 0 | 0
  Other, Qatar (n=17,21,3) | 0 | 0 | 0
  Other, Romania (n=17,21,3) | 0 | 0 | 0
  Other, Taiwan (n=17,21,3) | 3 | 0 | 0
  Other, Turkey (n=17,21,3) | 5 | 12 | 3
  Other, Slovakia (n=17,21,3) | 0 | 0 | 0
  Other, Serbia (n=17,21,3) | 0 | 0 | 0
  Other, Sweden (n=17,21,3) | 0 | 0 | 0
  Other, Switzerland (n=17,21,3) | 0 | 0 | 0
  Other, Syria (n=17,21,3) | 0 | 0 | 0
  Other, United Arab Emirates (n=17,21,3) | 0 | 0 | 0
  Other, Venezuela (n=17,21,3) | 1 | 0 | 0
  Total, Argentina (n=851,730,119) | 9 | 9 | 0
  Total, Belgium (n=851,730,119) | 45 | 33 | 7
  Total, Chile (n=851,730,119) | 13 | 15 | 3
  Total, Egypt (n=851,730,119) | 26 | 16 | 0
  Total, Estonia (n=851,730,119) | 4 | 2 | 1
  Total, France (n=851,730,119) | 129 | 141 | 14
  Total, Germany (n=851,730,119) | 39 | 33 | 7
  Total, Greece (n=851,730,119) | 15 | 23 | 4
  Total, Italy (n=851,730,119) | 140 | 128 | 21
  Total, Kuwait (n=851,730,119) | 0 | 0 | 0
  Total, Latvia (n=851,730,119) | 23 | 34 | 7
  Total, Lebanon (n=851,730,119) | 10 | 14 | 2
  Total, Lithuania (n=851,730,119) | 40 | 39 | 4
  Total, Macedonia (n=851,730,119) | 1 | 0 | 0
  Total, Mexico (n=851,730,119) | 8 | 19 | 5
  Total, Oman (n=851,730,119) | 5 | 2 | 0
  Total, Pakistan (n=851,730,119) | 15 | 13 | 3
  Total, Peru (n=851,730,119) | 9 | 17 | 6
  Total, Portugal (n=851,730,119) | 42 | 20 | 5
  Total, Qatar (n=851,730,119) | 5 | 2 | 0
  Total, Romania (n=851,730,119) | 51 | 66 | 11
  Total, Taiwan (n=851,730,119) | 149 | 14 | 1
  Total, Turkey (n=851,730,119) | 47 | 60 | 14
  Total, Slovakia (n=851,730,119) | 8 | 11 | 1
  Total, Serbia (n=851,730,119) | 0 | 0 | 0
  Total, Sweden (n=851,730,119) | 2 | 2 | 0
  Total, Switzerland (n=851,730,119) | 2 | 5 | 1
  Total, Syria (n=851,730,119) | 0 | 0 | 0
  Total, United Arab Emirates (n=851,730,119) | 4 | 4 | 0
  Total, Venezuela (n=851,730,119) | 10 | 8 | 2
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.3465, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Other genotypes; Test type: Superiority or Other; p = 0.7358, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the IL28B distribution between the nominal categories of interest

69. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by IL28B Genotype rs8099917 Category: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Arm/Group | Naive: IL28B rs12979860 CC | Naive: IL28B rs12979860 TC | Naive: IL28B rs12979860 TT
Number analyzed (Participants) | 978 | 1518 | 420
participants
  Naive: IL28B rs8099917 TT | 974 | 550 | 74
  Naive: IL28B rs8099917 TG | 4 | 965 | 178
  Naive: IL28B rs8099917 GG | 0 | 3 | 168
Statistical Analysis 1: Comparison: Naive: IL28B rs12979860 CC vs Naive: IL28B rs12979860 TC vs Naive: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

70. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by IL28B Genotype rs8099917 Category: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 490 | 914 | 296
participants
  Experienced: IL28B rs8099917 TT | 489 | 314 | 48
  Experienced: IL28B rs8099917 TG | 1 | 597 | 132
  Experienced: IL28B rs8099917 GG | 0 | 3 | 116
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

71. Secondary Outcome: Number of Participants With Inosine Triphosphatase (ITPA) Genotype rs7270101 by ITPA Genotype rs1127354 Category: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive).
Measure: Number; unit: participants
Groups:
- Naive: ITPA rs7270101 CC: Treatment-naive participants with CHC with ITPA rs7270101 polymorphism 'CC' confirmed by blood sampling.
- Naive: ITPA rs7270101 Alanine-Cysteine (AC): Treatment-naive participants with CHC with ITPA rs7270101 polymorphism 'AC' confirmed by blood sampling.
- Naive: ITPA rs7270101 Alanine-Alanine (AA): Treatment-naive participants with CHC with ITPA rs7270101 polymorphism 'AA' confirmed by blood sampling.
Arm/Group | Naive: ITPA rs7270101 CC | Naive: ITPA rs7270101 Alanine-Cysteine (AC) | Naive: ITPA rs7270101 Alanine-Alanine (AA)
Number analyzed (Participants) | 36 | 491 | 2389
participants
  Naive: ITPA rs1127354 AA | 0 | 0 | 11
  Naive: ITPA rs1127354 Cysteine-Alanine (CA) | 0 | 34 | 343
  Naive: ITPA rs1127354 CC | 36 | 457 | 2035
Statistical Analysis 1: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 Alanine-Cysteine (AC) vs Naive: ITPA rs7270101 Alanine-Alanine (AA); Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Tests for association between the two variables

72. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by ITPA Genotype rs1127354 Category: Treatment-Experienced
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Experienced).
Measure: Number; unit: participants
Groups:
- Experienced: ITPA rs7270101 CC: Treatment-experienced participants with CHC with ITPA rs7270101 polymorphism 'CC' confirmed by blood sampling.
- Experienced: ITPA rs7270101 AC: Treatment-experienced participants with CHC with ITPA rs7270101 polymorphism 'AC' confirmed by blood sampling.
- Experienced: ITPA rs7270101 AA: Treatment-experienced participants with CHC with ITPA rs7270101 polymorphism 'AA' confirmed by blood sampling.
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 18 | 269 | 1411
participants
  Experienced: ITPA rs1127354 AA | 0 | 0 | 15
  Experienced: ITPA rs1127354 CA | 0 | 23 | 211
  Experienced: ITPA rs1127354 CC | 18 | 246 | 1185
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Test type: Superiority or Other; p = 0.0066, Chi-squared — Pearson Chi-Square Tests for association between the two variables

73. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Region: Treatment-Naive
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype. HCV RNA genotype was obtained from medical records, and geographic region of study site was documented during intake/enrollment.
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: ITPA rs1127354 AA: Treatment-naive participants with CHC with ITPA rs1127354 polymorphism 'AA' confirmed by blood sampling.
- Naive: ITPA rs1127354 CA: Treatment-naive participants with CHC with ITPA rs1127354 polymorphism 'CA' confirmed by blood sampling.
- Naive: ITPA rs1127354 CC: Treatment-naive participants with CHC with ITPA rs1127354 polymorphism 'CC' confirmed by blood sampling.
Arm/Group | Naive: ITPA rs1127354 AA | Naive: ITPA rs1127354 CA | Naive: ITPA rs1127354 CC
Number analyzed (Participants) | 11 | 377 | 2528
participants
  G1, Asia (n=9,212,1481) | 0 | 8 | 17
  G1, Europe (n=9,212,1481) | 7 | 167 | 1077
  G1, Middle East (n=9,212,1481) | 2 | 32 | 255
  G1, Latin America (n=9,212,1481) | 0 | 5 | 132
  G2, Asia (n=0,45,278) | 0 | 3 | 3
  G2, Europe (n=0,45,278) | 0 | 37 | 254
  G2, Middle East (n=0,45,278) | 0 | 3 | 16
  G2, Latin America (n=0,45,278) | 0 | 2 | 5
  G3, Asia (n=1,83,490) | 0 | 17 | 88
  G3, Europe (n=1,83,490) | 1 | 62 | 369
  G3, Middle East (n=1,83,490) | 0 | 3 | 27
  G3, Latin America (n=1,83,490) | 0 | 1 | 6
  G4, Asia (n=0,30,230) | 0 | 0 | 0
  G4, Europe (n=0,30,230) | 0 | 16 | 112
  G4, Middle East (n=0,30,230) | 0 | 14 | 113
  G4, Latin America (n=0,30,230) | 0 | 0 | 5
  Other, Asia (n=1,7,49) | 1 | 2 | 13
  Other, Europe (n=1,7,49) | 0 | 2 | 15
  Other, Middle East (n=1,7,49) | 0 | 3 | 17
  Other, Latin America (n=1,7,49) | 0 | 0 | 4
  Total, Asia (n=11,377,2528) | 1 | 30 | 121
  Total, Europe (n=11,377,2528) | 8 | 284 | 1827
  Total, Middle East (n=11,377,2528) | 2 | 55 | 428
  Total, Latin America (n=11,377,2528) | 0 | 8 | 152
Statistical Analysis 1: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p = 0.0018, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.0425, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.9829, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.6700, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.7672, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p = 0.0067, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

74. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Region: Treatment-Experienced
Description: as for outcome 73
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Experienced: ITPA rs1127354 AA: Treatment-experienced participants with CHC with ITPA rs1127354 polymorphism 'AA' confirmed by blood sampling.
- Experienced: ITPA rs1127354 CA: Treatment-experienced participants with CHC with ITPA rs1127354 polymorphism 'CA' confirmed by blood sampling.
- Experienced: ITPA rs1127354 CC: Treatment-experienced participants with CHC with ITPA rs1127354 polymorphism 'CC' confirmed by blood sampling.
Arm/Group | Experienced: ITPA rs1127354 AA | Experienced: ITPA rs1127354 CA | Experienced: ITPA rs1127354 CC
Number analyzed (Participants) | 15 | 235 | 1449
participants
  G1, Asia (n=10,169,1057) | 2 | 27 | 67
  G1, Europe (n=10,169,1057) | 8 | 117 | 768
  G1, Middle East (n=10,169,1057) | 0 | 16 | 118
  G1, Latin America (n=10,169,1057) | 0 | 9 | 104
  G2, Asia (n=3,30,108) | 2 | 21 | 45
  G2, Europe (n=3,30,108) | 1 | 9 | 53
  G2, Middle East (n=3,30,108) | 0 | 0 | 5
  G2, Latin America (n=3,30,108) | 0 | 0 | 5
  G3, Asia (n=2,26,139) | 1 | 4 | 21
  G3, Europe (n=2,26,139) | 1 | 20 | 107
  G3, Middle East (n=2,26,139) | 0 | 0 | 3
  G3, Latin America (n=2,26,139) | 0 | 2 | 8
  G4, Asia (n=0,5,109) | 0 | 0 | 0
  G4, Europe (n=0,5,109) | 0 | 2 | 62
  G4, Middle East (n=0,5,109) | 0 | 3 | 45
  G4, Latin America (n=0,5,109) | 0 | 0 | 2
  Other, Asia (n=0,5,36) | 0 | 1 | 4
  Other, Europe (n=0,5,36) | 0 | 1 | 11
  Other, Middle East (n=0,5,36) | 0 | 3 | 18
  Other, Latin America (n=0,5,36) | 0 | 0 | 3
  Total, Asia (n=15,235,1449) | 5 | 53 | 137
  Total, Europe (n=15,235,1449) | 10 | 149 | 1001
  Total, Middle East (n=15,235,1449) | 0 | 22 | 189
  Total, Latin America (n=15,235,1449) | 0 | 11 | 122
Statistical Analysis 1: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p = 0.0003, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.1637, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.8579, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.6935, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.8124, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

75. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Region: Treatment-Naive
Description: as for outcome 73
Time Frame: Study Visit 1
Population: Core Analysis Population (Treatment-Naive); n = number of participants analyzed within each HCV RNA genotype category.
Measure: Number; unit: participants
Groups:
- Naive: ITPA rs7270101 AC: Treatment-naive participants with CHC with ITPA rs7270101 polymorphism 'AC' confirmed by blood sampling.
- Naive: ITPA rs7270101 AA: Treatment-naive participants with CHC with ITPA rs7270101 polymorphism 'AA' confirmed by blood sampling.
Arm/Group | Naive: ITPA rs7270101 CC | Naive: ITPA rs7270101 AC | Naive: ITPA rs7270101 AA
Number analyzed (Participants) | 36 | 491 | 2389
participants
  G1, Asia (n=17,300,1385) | 0 | 0 | 25
  G1, Europe (n=17,300,1385) | 14 | 230 | 1007
  G1, Middle East (n=17,300,1385) | 1 | 50 | 238
  G1, Latin America (n=17,300,1385) | 2 | 20 | 115
  G2, Asia (n=6,56,261) | 0 | 0 | 6
  G2, Europe (n=6,56,261) | 6 | 51 | 234
  G2, Middle East (n=6,56,261) | 0 | 3 | 16
  G2, Latin America (n=6,56,261) | 0 | 2 | 5
  G3, Asia (n=9,81,484) | 0 | 7 | 98
  G3, Europe (n=9,81,484) | 9 | 69 | 354
  G3, Middle East (n=9,81,484) | 0 | 4 | 26
  G3, Latin America (n=9,81,484) | 0 | 1 | 6
  G4, Asia (n=3,51,206) | 0 | 0 | 0
  G4, Europe (n=3,51,206) | 0 | 33 | 95
  G4, Middle East (n=3,51,206) | 3 | 16 | 108
  G4, Latin America (n=3,51,206) | 0 | 2 | 3
  Other, Asia (n=1,3,53) | 0 | 0 | 16
  Other, Europe (n=1,3,53) | 1 | 2 | 14
  Other, Middle East (n=1,3,53) | 0 | 1 | 19
  Other, Latin America (n=1,3,53) | 0 | 0 | 4
  Total, Asia (n=36,491,2389) | 0 | 7 | 145
  Total, Europe (n=36,491,2389) | 30 | 385 | 1704
  Total, Middle East (n=36,491,2389) | 4 | 74 | 407
  Total, Latin America (n=36,491,2389) | 2 | 25 | 133
Statistical Analysis 1: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p = 0.1834, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p = 0.8543, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.1485, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.0260, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; Other genotypes; Test type: Superiority or Other; p = 0.5317, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p = 0.0005, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

76. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Region: Treatment-Experienced
Description: as for outcome 73
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 18 | 270 | 1411
participants
  G1, Asia (n=14,214,1009) | 0 | 0 | 96
  G1, Europe (n=14,214,1009) | 13 | 175 | 706
  G1, Middle East (n=14,214,1009) | 0 | 21 | 113
  G1, Latin America (n=14,214,1009) | 1 | 18 | 94
  G2, Asia (n=1,9,130) | 0 | 0 | 67
  G2, Europe (n=1,9,130) | 0 | 8 | 55
  G2, Middle East (n=1,9,130) | 1 | 0 | 4
  G2, Latin America (n=1,9,130) | 0 | 1 | 4
  G3, Asia (n=2,18,147) | 0 | 0 | 26
  G3, Europe (n=2,18,147) | 2 | 16 | 110
  G3, Middle East (n=2,18,147) | 0 | 1 | 2
  G3, Latin America (n=2,18,147) | 0 | 1 | 9
  G4, Asia (n=1,22,91) | 0 | 0 | 0
  G4, Europe (n=1,22,91) | 1 | 16 | 47
  G4, Middle East (n=1,22,91) | 0 | 6 | 42
  G4, Latin America (n=1,22,91) | 0 | 0 | 2
  Other, Asia (n=0,7,34) | 0 | 0 | 5
  Other, Europe (n=0,7,34) | 0 | 3 | 9
  Other, Middle East (n=0,7,34) | 0 | 4 | 17
  Other, Latin America (n=0,7,34) | 0 | 0 | 3
  Total, Asia (n=18,270,1411) | 0 | 0 | 194
  Total, Europe (n=18,270,1411) | 16 | 218 | 927
  Total, Middle East (n=18,270,1411) | 1 | 32 | 178
  Total, Latin America (n=18,270,1411) | 1 | 20 | 112
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.4423, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 4: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.3824, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 5: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC; Other genotypes; Test type: Superiority or Other; p = 0.5246, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 6: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

77. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Country: Treatment-Naive (Table 1 of 2 [G1, G2, G3])
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype. HCV RNA genotype was obtained from medical records, and country of study site was documented during intake/enrollment.
Time Frame: Study Visit 1
Population: as for outcome 61
Measure: Number; unit: participants
Arm/Group | Naive: ITPA rs1127354 AA | Naive: ITPA rs1127354 CA | Naive: ITPA rs1127354 CC
Number analyzed (Participants) | 11 | 377 | 2528
participants
  G1, Argentina (n=9,212,1481) | 0 | 0 | 16
  G1, Belgium (n=9,212,1481) | 0 | 12 | 57
  G1, Chile (n=9,212,1481) | 0 | 1 | 17
  G1, Egypt (n=9,212,1481) | 0 | 0 | 0
  G1, Estonia (n=9,212,1481) | 0 | 11 | 114
  G1, France (n=9,212,1481) | 1 | 18 | 121
  G1, Germany (n=9,212,1481) | 2 | 12 | 86
  G1, Greece (n=9,212,1481) | 1 | 5 | 62
  G1, Italy (n=9,212,1481) | 2 | 45 | 280
  G1, Kuwait (n=9,212,1481) | 0 | 0 | 1
  G1, Latvia (n=9,212,1481) | 0 | 3 | 7
  G1, Lebanon (n=9,212,1481) | 0 | 1 | 21
  G1, Lithuania (n=9,212,1481) | 1 | 11 | 59
  G1, Macedonia (n=9,212,1481) | 0 | 6 | 25
  G1, Mexico (n=9,212,1481) | 0 | 0 | 20
  G1, Oman (n=9,212,1481) | 0 | 2 | 6
  G1, Pakistan (n=9,212,1481) | 0 | 2 | 7
  G1, Peru (n=9,212,1481) | 0 | 3 | 58
  G1, Portugal (n=9,212,1481) | 0 | 4 | 22
  G1, Qatar (n=9,212,1481) | 0 | 0 | 3
  G1, Romania (n=9,212,1481) | 0 | 32 | 183
  G1, Taiwan (n=9,212,1481) | 0 | 6 | 10
  G1, Turkey (n=9,212,1481) | 1 | 28 | 214
  G1, Slovakia (n=9,212,1481) | 0 | 5 | 23
  G1, Serbia (n=9,212,1481) | 0 | 2 | 11
  G1, Sweden (n=9,212,1481) | 0 | 1 | 13
  G1, Switzerland (n=9,212,1481) | 0 | 0 | 14
  G1, Syria (n=9,212,1481) | 1 | 0 | 1
  G1, United Arab Emirates (n=9,212,1481) | 0 | 1 | 9
  G1, Venezuela (n=9,212,1481) | 0 | 1 | 21
  G2, Argentina (n=0,45,278) | 0 | 0 | 0
  G2, Belgium (n=0,45,278) | 0 | 1 | 7
  G2, Chile (n=0,45,278) | 0 | 0 | 0
  G2, Egypt (n=0,45,278) | 0 | 0 | 0
  G2, Estonia (n=0,45,278) | 0 | 2 | 9
  G2, France (n=0,45,278) | 0 | 0 | 9
  G2, Germany (n=0,45,278) | 0 | 0 | 5
  G2, Greece (n=0,45,278) | 0 | 1 | 6
  G2, Italy (n=0,45,278) | 0 | 29 | 199
  G2, Kuwait (n=0,45,278) | 0 | 0 | 0
  G2, Latvia (n=0,45,278) | 0 | 0 | 1
  G2, Lebanon (n=0,45,278) | 0 | 1 | 1
  G2, Lithuania (n=0,45,278) | 0 | 3 | 12
  G2, Macedonia (n=0,45,278) | 0 | 0 | 0
  G2, Mexico (n=0,45,278) | 0 | 1 | 2
  G2, Oman (n=0,45,278) | 0 | 0 | 0
  G2, Pakistan (n=0,45,278) | 0 | 2 | 0
  G2, Peru (n=0,45,278) | 0 | 0 | 0
  G2, Portugal (n=0,45,278) | 0 | 0 | 1
  G2, Qatar (n=0,45,278) | 0 | 0 | 0
  G2, Romania (n=0,45,278) | 0 | 0 | 0
  G2, Taiwan (n=0,45,278) | 0 | 1 | 3
  G2, Turkey (n=0,45,278) | 0 | 2 | 15
  G2, Slovakia (n=0,45,278) | 0 | 0 | 0
  G2, Serbia (n=0,45,278) | 0 | 0 | 0
  G2, Sweden (n=0,45,278) | 0 | 1 | 3
  G2, Switzerland (n=0,45,278) | 0 | 0 | 2
  G2, Syria (n=0,45,278) | 0 | 0 | 0
  G2, United Arab Emirates (n=0,45,278) | 0 | 0 | 0
  G2, Venezuela (n=0,45,278) | 0 | 1 | 3
  G3, Argentina (n=1,83,490) | 0 | 0 | 1
  G3, Belgium (n=1,83,490) | 0 | 4 | 12
  G3, Chile (n=1,83,490) | 0 | 0 | 0
  G3, Egypt (n=1,83,490) | 0 | 0 | 0
  G3, Estonia (n=1,83,490) | 0 | 6 | 52
  G3, France (n=1,83,490) | 0 | 1 | 18
  G3, Germany (n=1,83,490) | 0 | 4 | 19
  G3, Greece (n=1,83,490) | 0 | 8 | 50
  G3, Italy (n=1,83,490) | 0 | 26 | 136
  G3, Kuwait (n=1,83,490) | 0 | 1 | 0
  G3, Latvia (n=1,83,490) | 0 | 0 | 0
  G3, Lebanon (n=1,83,490) | 0 | 0 | 9
  G3, Lithuania (n=1,83,490) | 0 | 5 | 26
  G3, Macedonia (n=1,83,490) | 0 | 3 | 12
  G3, Mexico (n=1,83,490) | 0 | 0 | 4
  G3, Oman (n=1,83,490) | 0 | 0 | 5
  G3, Pakistan (n=1,83,490) | 0 | 17 | 88
  G3, Peru (n=1,83,490) | 0 | 1 | 0
  G3, Portugal (n=1,83,490) | 0 | 2 | 7
  G3, Qatar (n=1,83,490) | 0 | 0 | 0
  G3, Romania (n=1,83,490) | 0 | 0 | 2
  G3, Taiwan (n=1,83,490) | 0 | 0 | 0
  G3, Turkey (n=1,83,490) | 0 | 2 | 11
  G3, Slovakia (n=1,83,490) | 0 | 1 | 10
  G3, Serbia (n=1,83,490) | 1 | 2 | 10
  G3, Sweden (n=1,83,490) | 0 | 0 | 11
  G3, Switzerland (n=1,83,490) | 0 | 0 | 4
  G3, Syria (n=1,83,490) | 0 | 0 | 0
  G3, United Arab Emirates (n=1,83,490) | 0 | 0 | 2
  G3, Venezuela (n=1,83,490) | 0 | 0 | 1
Statistical Analysis 1: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.1947, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.0226, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

78. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Country: Treatment-Naive (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 62
Measure: Number; unit: participants
Arm/Group | Naive: ITPA rs1127354 AA | Naive: ITPA rs1127354 CA | Naive: ITPA rs1127354 CC
Number analyzed (Participants) | 11 | 377 | 2528
participants
  G4, Argentina (n=0,30,230) | 0 | 0 | 4
  G4, Belgium (n=0,30,230) | 0 | 1 | 12
  G4, Chile (n=0,30,230) | 0 | 0 | 0
  G4, Egypt (n=0,30,230) | 0 | 4 | 54
  G4, Estonia (n=0,30,230) | 0 | 0 | 1
  G4, France (n=0,30,230) | 0 | 3 | 16
  G4, Germany (n=0,30,230) | 0 | 0 | 1
  G4, Greece (n=0,30,230) | 0 | 2 | 10
  G4, Italy (n=0,30,230) | 0 | 8 | 63
  G4, Kuwait (n=0,30,230) | 0 | 1 | 6
  G4, Latvia (n=0,30,230) | 0 | 0 | 0
  G4, Lebanon (n=0,30,230) | 0 | 1 | 23
  G4, Lithuania (n=0,30,230) | 0 | 0 | 0
  G4, Macedonia (n=0,30,230) | 0 | 0 | 0
  G4, Mexico (n=0,30,230) | 0 | 0 | 0
  G4, Oman (n=0,30,230) | 0 | 0 | 0
  G4, Pakistan (n=0,30,230) | 0 | 0 | 0
  G4, Peru (n=0,30,230) | 0 | 0 | 0
  G4, Portugal (n=0,30,230) | 0 | 0 | 6
  G4, Qatar (n=0,30,230) | 0 | 0 | 0
  G4, Romania (n=0,30,230) | 0 | 0 | 0
  G4, Taiwan (n=0,30,230) | 0 | 0 | 0
  G4, Turkey (n=0,30,230) | 0 | 4 | 6
  G4, Slovakia (n=0,30,230) | 0 | 0 | 0
  G4, Serbia (n=0,30,230) | 0 | 2 | 1
  G4, Sweden (n=0,30,230) | 0 | 0 | 0
  G4, Switzerland (n=0,30,230) | 0 | 0 | 2
  G4, Syria (n=0,30,230) | 0 | 2 | 16
  G4, United Arab Emirates (n=0,30,230) | 0 | 2 | 8
  G4, Venezuela (n=0,30,230) | 0 | 0 | 1
  Other, Argentina (n=1,7,49) | 0 | 0 | 0
  Other, Belgium (n=1,7,49) | 0 | 0 | 5
  Other, Chile (n=1,7,49) | 0 | 0 | 0
  Other, Egypt (n=1,7,49) | 0 | 0 | 0
  Other, Estonia (n=1,7,49) | 0 | 0 | 0
  Other, France (n=1,7,49) | 0 | 0 | 7
  Other, Germany (n=1,7,49) | 0 | 0 | 1
  Other, Greece (n=1,7,49) | 0 | 0 | 0
  Other, Italy (n=1,7,49) | 0 | 1 | 2
  Other, Kuwait (n=1,7,49) | 0 | 0 | 0
  Other, Latvia (n=1,7,49) | 0 | 0 | 0
  Other, Lebanon (n=1,7,49) | 0 | 1 | 0
  Other, Lithuania (n=1,7,49) | 0 | 0 | 0
  Other, Macedonia (n=1,7,49) | 0 | 0 | 0
  Other, Mexico (n=1,7,49) | 0 | 0 | 0
  Other, Oman (n=1,7,49) | 0 | 0 | 0
  Other, Pakistan (n=1,7,49) | 0 | 0 | 2
  Other, Peru (n=1,7,49) | 0 | 0 | 2
  Other, Portugal (n=1,7,49) | 0 | 0 | 0
  Other, Qatar (n=1,7,49) | 0 | 0 | 0
  Other, Romania (n=1,7,49) | 0 | 0 | 0
  Other, Taiwan (n=1,7,49) | 1 | 2 | 11
  Other, Turkey (n=1,7,49) | 0 | 2 | 17
  Other, Slovakia (n=1,7,49) | 0 | 0 | 0
  Other, Serbia (n=1,7,49) | 0 | 0 | 0
  Other, Sweden (n=1,7,49) | 0 | 0 | 0
  Other, Switzerland (n=1,7,49) | 0 | 1 | 0
  Other, Syria (n=1,7,49) | 0 | 0 | 0
  Other, United Arab Emirates (n=1,7,49) | 0 | 0 | 0
  Other, Venezuela (n=1,7,49) | 0 | 0 | 2
  Total, Argentina (n=11,377,2528) | 0 | 0 | 21
  Total, Belgium (n=11,377,2528) | 0 | 18 | 93
  Total, Chile (n=11,377,2528) | 0 | 1 | 17
  Total, Egypt (n=11,377,2528) | 0 | 4 | 54
  Total, Estonia (n=11,377,2528) | 0 | 19 | 176
  Total, France (n=11,377,2528) | 1 | 22 | 171
  Total, Germany (n=11,377,2528) | 2 | 16 | 112
  Total, Greece (n=11,377,2528) | 1 | 16 | 128
  Total, Italy (n=11,377,2528) | 2 | 109 | 680
  Total, Kuwait (n=11,377,2528) | 0 | 2 | 7
  Total, Latvia (n=11,377,2528) | 0 | 3 | 8
  Total, Lebanon (n=11,377,2528) | 0 | 4 | 54
  Total, Lithuania (n=11,377,2528) | 1 | 19 | 97
  Total, Macedonia (n=11,377,2528) | 0 | 9 | 37
  Total, Mexico (n=11,377,2528) | 0 | 1 | 26
  Total, Oman (n=11,377,2528) | 0 | 2 | 11
  Total, Pakistan (n=11,377,2528) | 0 | 21 | 97
  Total, Peru (n=11,377,2528) | 0 | 4 | 60
  Total, Portugal (n=11,377,2528) | 0 | 6 | 36
  Total, Qatar (n=11,377,2528) | 0 | 0 | 3
  Total, Romania (n=11,377,2528) | 0 | 32 | 185
  Total, Taiwan (n=11,377,2528) | 1 | 9 | 24
  Total, Turkey (n=11,377,2528) | 1 | 38 | 263
  Total, Slovakia (n=11,377,2528) | 0 | 6 | 33
  Total, Serbia (n=11,377,2528) | 1 | 6 | 22
  Total, Sweden (n=11,377,2528) | 0 | 2 | 27
  Total, Switzerland (n=11,377,2528) | 0 | 1 | 22
  Total, Syria (n=11,377,2528) | 1 | 2 | 17
  Total, United Arab Emirates (n=11,377,2528) | 0 | 3 | 19
  Total, Venezuela (n=11,377,2528) | 0 | 2 | 28
Statistical Analysis 1: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.1158, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.3675, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs1127354 AA vs Naive: ITPA rs1127354 CA vs Naive: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p = 0.0948, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

79. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Country: Treatment-Experienced (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 63
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs1127354 AA | Experienced: ITPA rs1127354 CA | Experienced: ITPA rs1127354 CC
Number analyzed (Participants) | 15 | 235 | 1449
participants
  G1, Argentina (n=10,169,1057) | 0 | 1 | 12
  G1, Belgium (n=10,169,1057) | 0 | 8 | 52
  G1, Chile (n=10,169,1057) | 0 | 1 | 25
  G1, Egypt (n=10,169,1057) | 0 | 0 | 1
  G1, Estonia (n=10,169,1057) | 1 | 0 | 6
  G1, France (n=10,169,1057) | 2 | 23 | 185
  G1, Germany (n=10,169,1057) | 1 | 8 | 60
  G1, Greece (n=10,169,1057) | 0 | 6 | 23
  G1, Italy (n=10,169,1057) | 3 | 23 | 177
  G1, Kuwait (n=10,169,1057) | 0 | 0 | 0
  G1, Latvia (n=10,169,1057) | 0 | 12 | 50
  G1, Lebanon (n=10,169,1057) | 0 | 2 | 18
  G1, Lithuania (n=10,169,1057) | 1 | 12 | 47
  G1, Macedonia (n=10,169,1057) | 0 | 0 | 0
  G1, Mexico (n=10,169,1057) | 0 | 3 | 24
  G1, Oman (n=10,169,1057) | 0 | 1 | 5
  G1, Pakistan (n=10,169,1057) | 0 | 1 | 3
  G1, Peru (n=10,169,1057) | 0 | 1 | 29
  G1, Portugal (n=10,169,1057) | 0 | 7 | 31
  G1, Qatar (n=10,169,1057) | 0 | 1 | 6
  G1, Romania (n=10,169,1057) | 0 | 13 | 114
  G1, Taiwan (n=10,169,1057) | 2 | 26 | 64
  G1, Turkey (n=10,169,1057) | 0 | 12 | 82
  G1, Slovakia (n=10,169,1057) | 0 | 2 | 15
  G1, Serbia (n=10,169,1057) | 0 | 0 | 0
  G1, Sweden (n=10,169,1057) | 0 | 1 | 2
  G1, Switzerland (n=10,169,1057) | 0 | 2 | 6
  G1, Syria (n=10,169,1057) | 0 | 0 | 0
  G1, United Arab Emirates (n=10,169,1057) | 0 | 0 | 6
  G1, Venezuela (n=10,169,1057) | 0 | 3 | 14
  G2, Argentina (n=3,30,108) | 0 | 0 | 0
  G2, Belgium (n=3,30,108) | 0 | 0 | 0
  G2, Chile (n=3,30,108) | 0 | 0 | 0
  G2, Egypt (n=3,30,108) | 0 | 0 | 0
  G2, Estonia (n=3,30,108) | 0 | 0 | 0
  G2, France (n=3,30,108) | 0 | 2 | 18
  G2, Germany (n=3,30,108) | 0 | 0 | 0
  G2, Greece (n=3,30,108) | 0 | 0 | 1
  G2, Italy (n=3,30,108) | 0 | 5 | 32
  G2, Kuwait (n=3,30,108) | 0 | 0 | 0
  G2, Latvia (n=3,30,108) | 0 | 0 | 2
  G2, Lebanon (n=3,30,108) | 0 | 0 | 0
  G2, Lithuania (n=3,30,108) | 1 | 2 | 0
  G2, Macedonia (n=3,30,108) | 0 | 0 | 0
  G2, Mexico (n=3,30,108) | 0 | 0 | 3
  G2, Oman (n=3,30,108) | 0 | 0 | 0
  G2, Pakistan (n=3,30,108) | 0 | 0 | 0
  G2, Peru (n=3,30,108) | 0 | 0 | 0
  G2, Portugal (n=3,30,108) | 0 | 0 | 0
  G2, Qatar (n=3,30,108) | 0 | 0 | 0
  G2, Romania (n=3,30,108) | 0 | 0 | 0
  G2, Taiwan (n=3,30,108) | 2 | 21 | 45
  G2, Turkey (n=3,30,108) | 0 | 0 | 5
  G2, Slovakia (n=3,30,108) | 0 | 0 | 0
  G2, Serbia (n=3,30,108) | 0 | 0 | 0
  G2, Sweden (n=3,30,108) | 0 | 0 | 0
  G2, Switzerland (n=3,30,108) | 0 | 0 | 0
  G2, Syria (n=3,30,10) | 0 | 0 | 0
  G2, United Arab Emirates (n=3,30,108) | 0 | 0 | 0
  G2, Venezuela (n=3,30,108) | 0 | 0 | 2
  G3, Argentina (n=2,26,139) | 0 | 1 | 3
  G3, Belgium (n=2,26,139) | 1 | 3 | 5
  G3, Chile (n=2,26,139) | 0 | 0 | 4
  G3, Egypt (n=2,26,139) | 0 | 0 | 0
  G3, Estonia (n=2,26,139) | 0 | 0 | 0
  G3, France (n=2,26,139) | 0 | 1 | 26
  G3, Germany (n=2,26,139) | 0 | 1 | 6
  G3, Greece (n=2,26,139) | 0 | 1 | 7
  G3, Italy (n=2,26,139) | 0 | 5 | 29
  G3, Kuwait (n=2,26,139) | 0 | 0 | 0
  G3, Latvia (n=2,26,139) | 0 | 0 | 0
  G3, Lebanon (n=2,26,139) | 0 | 0 | 1
  G3, Lithuania (n=2,26,139) | 0 | 5 | 15
  G3, Macedonia (n=2,26,139) | 0 | 0 | 1
  G3, Mexico (n=2,26,139) | 0 | 1 | 1
  G3, Oman (n=2,26,139) | 0 | 0 | 0
  G3, Pakistan (n=2,26,139) | 1 | 3 | 21
  G3, Peru (n=2,26,139) | 0 | 0 | 0
  G3, Portugal (n=2,26,139) | 0 | 4 | 14
  G3, Qatar (n=2,26,139) | 0 | 0 | 0
  G3, Romania (n=2,26,139) | 0 | 0 | 0
  G3, Taiwan (n=2,26,139) | 0 | 1 | 0
  G3, Turkey (n=2,26,139) | 0 | 0 | 1
  G3, Slovakia (n=2,26,139) | 0 | 0 | 3
  G3, Serbia (n=2,26,139) | 0 | 0 | 0
  G3, Sweden (n=2,26,139) | 0 | 0 | 1
  G3, Switzerland (n=2,26,139) | 0 | 0 | 0
  G3, Syria (n=2,26,139) | 0 | 0 | 0
  G3, United Arab Emirates (n=2,26,139) | 0 | 0 | 1
  G3, Venezuela (n=2,26,139) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p = 0.1236, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.0119, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.7472, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

80. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by HCV RNA Genotype and Country: Treatment-Experienced (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 64
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs1127354 AA | Experienced: ITPA rs1127354 CA | Experienced: ITPA rs1127354 CC
Number analyzed (Participants) | 15 | 235 | 1449
participants
  G4, Argentina (n=0,5,109) | 0 | 0 | 1
  G4, Belgium (n=0,5,109) | 0 | 1 | 10
  G4, Chile (n=0,5,109) | 0 | 0 | 1
  G4, Egypt (n=0,5,109) | 0 | 3 | 38
  G4, Estonia (n=0,5,109) | 0 | 0 | 0
  G4, France (n=0,5,109) | 0 | 0 | 22
  G4, Germany (n=0,5,109) | 0 | 0 | 3
  G4, Greece (n=0,5,109) | 0 | 0 | 4
  G4, Italy (n=0,5,109) | 0 | 1 | 13
  G4, Kuwait (n=0,5,109) | 0 | 0 | 0
  G4, Latvia (n=0,5,109) | 0 | 0 | 0
  G4, Lebanon (n=0,5,109) | 0 | 0 | 5
  G4, Lithuania (n=0,5,109) | 0 | 0 | 0
  G4, Macedonia (n=0,5,109) | 0 | 0 | 0
  G4, Mexico (n=0,5,109) | 0 | 0 | 0
  G4, Oman (n=0,5,109) | 0 | 0 | 0
  G4, Pakistan | 0 | 0 | 0
  G4, Peru (n=0,5,109) | 0 | 0 | 0
  G4, Portugal (n=0,5,109) | 0 | 0 | 10
  G4, Qatar (n=0,5,109) | 0 | 0 | 0
  G4, Romania (n=0,5,109) | 0 | 0 | 0
  G4, Taiwan (n=0,5,109) | 0 | 0 | 0
  G4, Turkey (n=0,5,109) | 0 | 0 | 1
  G4, Slovakia (n=0,5,109) | 0 | 0 | 0
  G4, Serbia (n=0,5,109) | 0 | 0 | 0
  G4, Sweden (n=0,5,109) | 0 | 0 | 0
  G4, Switzerland (n=0,5,109) | 0 | 0 | 0
  G4, Syria (n=0,5,109) | 0 | 0 | 0
  G4, United Arab Emirates (n=0,5,109) | 0 | 0 | 1
  G4, Venezuela (n=0,5,109) | 0 | 0 | 0
  Other, Argentina (n=0,5,36) | 0 | 0 | 0
  Other, Belgium (n=0,5,36) | 0 | 0 | 5
  Other, Chile (n=0,5,36) | 0 | 0 | 0
  Other, Egypt (n=0,5,36) | 0 | 0 | 0
  Other, Estonia (n=0,5,36) | 0 | 0 | 0
  Other, France (n=0,5,36) | 0 | 1 | 4
  Other, Germany (n=0,5,36) | 0 | 0 | 0
  Other, Greece (n=0,5,36) | 0 | 0 | 0
  Other, Italy (n=0,5,36) | 0 | 0 | 1
  Other, Kuwait (n=0,5,36) | 0 | 0 | 0
  Other, Latvia (n=0,5,36) | 0 | 0 | 0
  Other, Lebanon (n=0,5,36) | 0 | 0 | 0
  Other, Lithuania (n=0,5,36) | 0 | 0 | 0
  Other, Macedonia (n=0,5,36) | 0 | 0 | 0
  Other, Mexico (n=0,5,36) | 0 | 0 | 0
  Other, Oman (n=0,5,36) | 0 | 0 | 1
  Other, Pakistan (n=0,5,36) | 0 | 1 | 1
  Other, Peru (n=0,5,36) | 0 | 0 | 2
  Other, Portugal (n=0,5,36) | 0 | 0 | 1
  Other, Qatar (n=0,5,36) | 0 | 0 | 0
  Other, Romania (n=0,5,36) | 0 | 0 | 0
  Other, Taiwan (n=0,5,36) | 0 | 0 | 3
  Other, Turkey (n=0,5,36) | 0 | 3 | 17
  Other, Slovakia (n=0,5,36) | 0 | 0 | 0
  Other, Serbia (n=0,5,36) | 0 | 0 | 0
  Other, Sweden (n=0,5,36) | 0 | 0 | 0
  Other, Switzerland (n=0,5,36) | 0 | 0 | 0
  Other, Syria (n=0,5,36) | 0 | 0 | 0
  Other, United Arab Emirates (n=0,5,36) | 0 | 0 | 0
  Other, Venezuela (n=0,5,36) | 0 | 0 | 1
  Total, Argentina (n=15,235,1449) | 0 | 2 | 16
  Total, Belgium (n=15,235,1449) | 1 | 12 | 72
  Total, Chile (n=15,235,1449) | 0 | 1 | 30
  Total, Egypt (n=15,235,1449) | 0 | 3 | 39
  Total, Estonia (n=15,235,1449) | 1 | 0 | 6
  Total, France (n=15,235,1449) | 2 | 27 | 255
  Total, Germany (n=15,235,1449) | 1 | 9 | 69
  Total, Greece (n=15,235,1449) | 0 | 7 | 35
  Total, Italy (n=15,235,1449) | 3 | 34 | 252
  Total, Kuwait (n=15,235,1449) | 0 | 0 | 0
  Total, Latvia (n=15,235,1449) | 0 | 12 | 52
  Total, Lebanon (n=15,235,1449) | 0 | 2 | 24
  Total, Lithuania (n=15,235,1449) | 2 | 19 | 62
  Total, Macedonia (n=15,235,1449) | 0 | 0 | 1
  Total, Mexico (n=15,235,1449) | 0 | 4 | 28
  Total, Oman (n=15,235,1449) | 0 | 1 | 6
  Total, Pakistan (n=15,235,1449) | 1 | 5 | 25
  Total, Peru (n=15,235,1449) | 0 | 1 | 31
  Total, Portugal (n=15,235,1449) | 0 | 11 | 56
  Total, Qatar (n=15,235,1449) | 0 | 1 | 6
  Total, Romania (n=15,235,1449) | 0 | 13 | 114
  Total, Taiwan (n=15,235,1449) | 4 | 48 | 112
  Total, Turkey (n=15,235,1449) | 0 | 15 | 106
  Total, Slovakia (n=15,235,1449) | 0 | 2 | 18
  Total, Serbia (n=15,235,1449) | 0 | 0 | 0
  Total, Sweden (n=15,235,1449) | 0 | 1 | 3
  Total, Switzerland (n=15,235,1449) | 0 | 2 | 6
  Total, Syria (n=15,235,1449) | 0 | 0 | 0
  Total, United Arab Emirates (n=15,235,1449) | 0 | 0 | 8
  Total, Venezuela (n=15,235,1449) | 0 | 3 | 17
Statistical Analysis 1: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.9734, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.8303, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p = 0.0006, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

81. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Country: Treatment-Naive (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 61
Measure: Number; unit: participants
Arm/Group | Naive: ITPA rs7270101 CC | Naive: ITPA rs7270101 AC | Naive: ITPA rs7270101 AA
Number analyzed (Participants) | 36 | 491 | 2389
participants
  G1, Argentina (n=17,300,1385) | 0 | 4 | 12
  G1, Belgium (n=17,300,1385) | 0 | 10 | 59
  G1, Chile (n=17,300,1385) | 0 | 3 | 15
  G1, Egypt (n=17,300,1385) | 0 | 0 | 0
  G1, Estonia (n=17,300,1385) | 1 | 20 | 104
  G1, France (n=17,300,1385) | 1 | 29 | 110
  G1, Germany (n=17,300,1385) | 0 | 13 | 87
  G1, Greece (n=17,300,1385) | 0 | 7 | 61
  G1, Italy (n=17,300,1385) | 6 | 57 | 264
  G1, Kuwait (n=17,300,1385) | 0 | 0 | 1
  G1, Latvia (n=17,300,1385) | 0 | 4 | 6
  G1, Lebanon (n=17,300,1385) | 1 | 7 | 14
  G1, Lithuania (n=17,300,1385) | 0 | 16 | 55
  G1, Macedonia (n=17,300,1385) | 0 | 6 | 25
  G1, Mexico (n=17,300,1385) | 0 | 3 | 17
  G1, Oman (n=17,300,1385) | 0 | 0 | 8
  G1, Pakistan (n=17,300,1385) | 0 | 0 | 9
  G1, Peru (n=17,300,1385) | 0 | 3 | 58
  G1, Portugal (n=17,300,1385) | 0 | 8 | 18
  G1, Qatar (n=17,300,1385) | 0 | 0 | 3
  G1, Romania (n=17,300,1385) | 5 | 43 | 167
  G1, Taiwan (n=17,300,1385) | 0 | 0 | 16
  G1, Turkey (n=17,300,1385) | 0 | 41 | 202
  G1, Slovakia (n=17,300,1385) | 0 | 11 | 17
  G1, Serbia (n=17,300,1385) | 0 | 2 | 11
  G1, Sweden (n=17,300,1385) | 0 | 1 | 13
  G1, Switzerland (n=17,300,1385) | 1 | 3 | 10
  G1, Syria (n=17,300,1385) | 0 | 0 | 2
  G1, United Arab Emirates (n=17,300,1385) | 0 | 2 | 8
  G1, Venezuela (n=17,300,1385) | 2 | 7 | 13
  G2, Argentina (n=6,56,261) | 0 | 0 | 0
  G2, Belgium (n=6,56,261) | 0 | 1 | 7
  G2, Chile (n=6,56,261) | 0 | 0 | 0
  G2, Egypt (n=6,56,261) | 0 | 0 | 0
  G2, Estonia (n=6,56,261) | 0 | 2 | 9
  G2, France (n=6,56,261) | 0 | 3 | 6
  G2, Germany (n=6,56,261) | 0 | 1 | 4
  G2, Greece (n=6,56,261) | 0 | 1 | 6
  G2, Italy (n=6,56,261) | 6 | 40 | 182
  G2, Kuwait (n=6,56,261) | 0 | 0 | 0
  G2, Latvia (n=6,56,261) | 0 | 0 | 1
  G2, Lebanon (n=6,56,261) | 0 | 0 | 2
  G2, Lithuania (n=6,56,261) | 0 | 2 | 13
  G2, Macedonia (n=6,56,261) | 0 | 0 | 0
  G2, Mexico (n=6,56,261) | 0 | 1 | 2
  G2, Oman (n=6,56,261) | 0 | 0 | 0
  G2, Pakistan (n=6,56,261) | 0 | 0 | 2
  G2, Peru (n=6,56,261) | 0 | 0 | 0
  G2, Portugal (n=6,56,261) | 0 | 0 | 1
  G2, Qatar (n=6,56,261) | 0 | 0 | 0
  G2, Romania (n=6,56,261) | 0 | 0 | 0
  G2, Taiwan (n=6,56,261) | 0 | 0 | 4
  G2, Turkey (n=6,56,261) | 0 | 3 | 14
  G2, Slovakia (n=6,56,261) | 0 | 0 | 0
  G2, Serbia (n=6,56,261) | 0 | 0 | 0
  G2, Sweden (n=6,56,261) | 0 | 0 | 4
  G2, Switzerland (n=6,56,261) | 0 | 1 | 1
  G2, Syria (n=6,56,261) | 0 | 0 | 0
  G2, United Arab Emirates (n=6,56,261) | 0 | 0 | 0
  G2, Venezuela (n=6,56,261) | 0 | 1 | 3
  G3, Argentina (n=9,81,484) | 0 | 1 | 0
  G3, Belgium (n=9,81,484) | 0 | 4 | 12
  G3, Chile (n=9,81,484) | 0 | 0 | 0
  G3, Egypt (n=9,81,484) | 0 | 0 | 0
  G3, Estonia (n=9,81,484) | 1 | 11 | 46
  G3, France (n=9,81,484) | 0 | 2 | 17
  G3, Germany (n=9,81,484) | 2 | 1 | 20
  G3, Greece (n=9,81,484) | 1 | 7 | 50
  G3, Italy (n=9,81,484) | 4 | 21 | 137
  G3, Kuwait (n=9,81,484) | 0 | 0 | 1
  G3, Latvia (n=9,81,484) | 0 | 0 | 0
  G3, Lebanon (n=9,81,484) | 0 | 3 | 6
  G3, Lithuania (n=9,81,484) | 1 | 8 | 22
  G3, Macedonia (n=9,81,484) | 0 | 4 | 11
  G3, Mexico (n=9,81,484) | 0 | 0 | 4
  G3, Oman (n=9,81,484) | 0 | 1 | 4
  G3, Pakistan (n=9,81,484) | 0 | 7 | 98
  G3, Peru (n=9,81,484) | 0 | 0 | 1
  G3, Portugal (n=9,81,484) | 0 | 3 | 6
  G3, Qatar (n=9,81,484) | 0 | 0 | 0
  G3, Romania (n=9,81,484) | 0 | 0 | 2
  G3, Taiwan (n=9,81,484) | 0 | 0 | 0
  G3, Turkey (n=9,81,484) | 0 | 0 | 13
  G3, Slovakia (n=9,81,484) | 0 | 3 | 8
  G3, Serbia (n=9,81,484) | 0 | 4 | 9
  G3, Sweden (n=9,81,484) | 0 | 1 | 10
  G3, Switzerland (n=9,81,484) | 0 | 0 | 4
  G3, Syria (n=9,81,484) | 0 | 0 | 0
  G3, United Arab Emirates (n=9,81,484) | 0 | 0 | 2
  G3, Venezuela (n=9,81,484) | 0 | 0 | 1
Statistical Analysis 1: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p = 0.0065, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p = 0.9999, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.3472, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

82. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Country: Treatment-Naive (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 62
Measure: Number; unit: participants
Arm/Group | Naive: ITPA rs7270101 CC | Naive: ITPA rs7270101 AC | Naive: ITPA rs7270101 AA
Number analyzed (Participants) | 36 | 491 | 2389
participants
  G4, Argentina (n=3,51,206) | 0 | 1 | 3
  G4, Belgium (n=3,51,206) | 0 | 1 | 12
  G4, Chile (n=3,51,206) | 2 | 9 | 47
  G4, Egypt (n=3,51,206) | 0 | 0 | 0
  G4, Estonia (n=3,51,206) | 0 | 0 | 1
  G4, France (n=3,51,206) | 0 | 4 | 15
  G4, Germany (n=3,51,206) | 0 | 1 | 0
  G4, Greece (n=3,51,206) | 0 | 3 | 9
  G4, Italy (n=3,51,206) | 0 | 20 | 51
  G4, Kuwait (n=3,51,206) | 0 | 0 | 7
  G4, Latvia (n=3,51,206) | 0 | 0 | 0
  G4, Lebanon (n=3,51,206) | 1 | 4 | 19
  G4, Lithuania (n=3,51,206) | 0 | 0 | 0
  G4, Macedonia (n=3,51,206) | 0 | 0 | 0
  G4, Mexico (n=3,51,206) | 0 | 0 | 0
  G4, Oman (n=3,51,206) | 0 | 0 | 0
  G4, Pakistan (n=3,51,206) | 0 | 0 | 0
  G4, Peru (n=3,51,206) | 0 | 0 | 0
  G4, Portugal (n=3,51,206) | 0 | 4 | 2
  G4, Qatar (n=3,51,206) | 0 | 0 | 0
  G4, Romania (n=3,51,206) | 0 | 0 | 0
  G4, Taiwan (n=3,51,206) | 0 | 0 | 0
  G4, Turkey (n=3,51,206) | 0 | 0 | 10
  G4, Slovakia (n=3,51,206) | 0 | 0 | 0
  G4, Serbia (n=3,51,206) | 0 | 0 | 3
  G4, Sweden (n=3,51,206) | 0 | 0 | 0
  G4, Switzerland (n=3,51,206) | 0 | 0 | 2
  G4, Syria (n=3,51,206) | 0 | 3 | 15
  G4, United Arab Emirates (n=3,51,206) | 0 | 0 | 10
  G4, Venezuela (n=3,51,206) | 0 | 1 | 0
  Other, Argentina (n=1,3,53) | 0 | 0 | 0
  Other, Belgium (n=1,3,53) | 1 | 1 | 3
  Other, Chile (n=1,3,53) | 0 | 0 | 0
  Other, Egypt (n=1,3,53) | 0 | 0 | 0
  Other, Estonia (n=1,3,53) | 0 | 0 | 0
  Other, France (n=1,3,53) | 0 | 1 | 6
  Other, Germany (n=1,3,53) | 0 | 0 | 1
  Other, Greece (n=1,3,53) | 0 | 0 | 0
  Other, Italy (n=1,3,53) | 0 | 0 | 3
  Other, Kuwait (n=1,3,53) | 0 | 0 | 0
  Other, Latvia (n=1,3,53) | 0 | 0 | 0
  Other, Lebanon (n=1,3,53) | 0 | 0 | 1
  Other, Lithuania (n=1,3,53) | 0 | 0 | 0
  Other, Macedonia (n=1,3,53) | 0 | 0 | 0
  Other, Mexico (n=1,3,53) | 0 | 0 | 0
  Other, Oman (n=1,3,53) | 0 | 0 | 0
  Other, Pakistan (n=1,3,53) | 0 | 0 | 2
  Other, Peru (n=1,3,53) | 0 | 0 | 2
  Other, Portugal (n=1,3,53) | 0 | 0 | 0
  Other, Qatar (n=1,3,53) | 0 | 0 | 0
  Other, Romania (n=1,3,53) | 0 | 0 | 0
  Other, Taiwan (n=1,3,53) | 0 | 0 | 14
  Other, Turkey (n=1,3,53) | 0 | 1 | 18
  Other, Slovakia (n=1,3,53) | 0 | 0 | 0
  Other, Serbia (n=1,3,53) | 0 | 0 | 0
  Other, Sweden (n=1,3,53) | 0 | 0 | 0
  Other, Switzerland (n=1,3,53) | 0 | 0 | 1
  Other, Syria (n=1,3,53) | 0 | 0 | 0
  Other, United Arab Emirates (n=1,3,53) | 0 | 0 | 0
  Other, Venezuela (n=1,3,53) | 0 | 0 | 2
  Total, Argentina (n=36,491,2389) | 0 | 6 | 15
  Total, Belgium (n=36,491,2389) | 1 | 17 | 93
  Total, Chile (n=36,491,2389) | 0 | 3 | 15
  Total, Egypt (n=36,491,2389) | 2 | 9 | 47
  Total, Estonia (n=36,491,2389) | 2 | 33 | 160
  Total, France (n=36,491,2389) | 1 | 39 | 154
  Total, Germany (n=36,491,2389) | 2 | 16 | 112
  Total, Greece (n=36,491,2389) | 1 | 18 | 126
  Total, Italy (n=36,491,2389) | 16 | 138 | 637
  Total, Kuwait (n=36,491,2389) | 0 | 0 | 9
  Total, Latvia (n=36,491,2389) | 0 | 4 | 7
  Total, Lebanon (n=36,491,2389) | 2 | 14 | 42
  Total, Lithuania (n=36,491,2389) | 1 | 26 | 90
  Total, Macedonia (n=36,491,2389) | 0 | 10 | 36
  Total, Mexico (n=36,491,2389) | 0 | 4 | 23
  Total, Oman (n=36,491,2389) | 0 | 1 | 12
  Total, Pakistan (n=36,491,2389) | 0 | 7 | 111
  Total, Peru (n=36,491,2389) | 0 | 3 | 61
  Total, Portugal (n=36,491,2389) | 0 | 15 | 27
  Total, Qatar (n=36,491,2389) | 0 | 0 | 3
  Total, Romania (n=36,491,2389) | 5 | 43 | 169
  Total, Taiwan (n=36,491,2389) | 0 | 0 | 34
  Total, Turkey (n=36,491,2389) | 0 | 45 | 257
  Total, Slovakia (n=36,491,2389) | 0 | 14 | 25
  Total, Serbia (n=36,491,2389) | 0 | 6 | 23
  Total, Sweden (n=36,491,2389) | 0 | 2 | 27
  Total, Switzerland (n=36,491,2389) | 1 | 4 | 18
  Total, Syria (n=36,491,2389) | 0 | 3 | 17
  Total, United Arab Emirates (n=36,491,2389) | 0 | 2 | 20
  Total, Venezuela (n=36,491,2389) | 2 | 9 | 19
Statistical Analysis 1: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.2564, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; Other genotypes; Test type: Superiority or Other; p = 0.7361, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Naive: ITPA rs7270101 CC vs Naive: ITPA rs7270101 AC vs Naive: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

83. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Country: Treatment-Experienced (Table 1 of 2 [G1, G2, G3])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 63
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 18 | 270 | 1411
participants
  G1, Argentina (n=14,214,1009) | 0 | 6 | 7
  G1, Belgium (n=14,214,1009) | 0 | 6 | 54
  G1, Chile (n=14,214,1009) | 0 | 4 | 22
  G1, Egypt (n=14,214,1009) | 0 | 0 | 1
  G1, Estonia (n=14,214,1009) | 0 | 0 | 7
  G1, France (n=14,214,1009) | 4 | 49 | 157
  G1, Germany (n=14,214,1009) | 0 | 19 | 50
  G1, Greece (n=14,214,1009) | 0 | 5 | 24
  G1, Italy (n=14,214,1009) | 4 | 41 | 158
  G1, Kuwait (n=14,214,1009) | 0 | 0 | 0
  G1, Latvia (n=14,214,1009) | 0 | 11 | 51
  G1, Lebanon (n=14,214,1009) | 0 | 2 | 18
  G1, Lithuania (n=14,214,1009) | 3 | 9 | 48
  G1, Macedonia (n=14,214,1009) | 0 | 0 | 0
  G1, Mexico (n=14,214,1009) | 0 | 3 | 24
  G1, Oman (n=14,214,1009) | 0 | 0 | 6
  G1, Pakistan (n=14,214,1009) | 0 | 0 | 4
  G1, Peru (n=14,214,1009) | 0 | 2 | 28
  G1, Portugal (n=14,214,1009) | 1 | 11 | 26
  G1, Qatar (n=14,214,1009) | 0 | 2 | 5
  G1, Romania (n=14,214,1009) | 1 | 20 | 107
  G1, Taiwan (n=14,214,1009) | 0 | 0 | 92
  G1, Turkey (n=14,214,1009) | 0 | 16 | 78
  G1, Slovakia (n=14,214,1009) | 0 | 3 | 14
  G1, Serbia (n=14,214,1009) | 0 | 0 | 0
  G1, Sweden (n=14,214,1009) | 0 | 0 | 3
  G1, Switzerland (n=14,214,1009) | 0 | 1 | 7
  G1, Syria (n=14,214,1009) | 0 | 0 | 0
  G1, United Arab Emirates (n=14,214,1009) | 0 | 1 | 5
  G1, Venezuela (n=14,214,1009) | 1 | 3 | 13
  G2, Argentina (n=1,9,130) | 0 | 0 | 0
  G2, Belgium (n=1,9,130) | 0 | 0 | 0
  G2, Chile (n=1,9,130) | 0 | 0 | 0
  G2, Egypt (n=1,9,130) | 0 | 0 | 0
  G2, Estonia (n=1,9,130) | 0 | 0 | 0
  G2, France (n=1,9,130) | 0 | 3 | 17
  G2, Germany (n=1,9,130) | 0 | 0 | 0
  G2, Greece (n=1,9,130) | 0 | 1 | 0
  G2, Italy (n=1,9,130) | 0 | 2 | 35
  G2, Kuwait (n=1,9,130) | 0 | 0 | 0
  G2, Latvia (n=1,9,130) | 0 | 0 | 2
  G2, Lebanon (n=1,9,130) | 0 | 0 | 0
  G2, Lithuania (n=1,9,130) | 0 | 2 | 1
  G2, Macedonia (n=1,9,130) | 0 | 0 | 0
  G2, Mexico (n=1,9,130) | 0 | 0 | 3
  G2, Oman (n=1,9,130) | 0 | 0 | 0
  G2, Pakistan (n=1,9,130) | 0 | 0 | 0
  G2, Peru (n=1,9,130) | 0 | 0 | 0
  G2, Portugal (n=1,9,130) | 0 | 0 | 0
  G2, Qatar (n=1,9,130) | 0 | 0 | 0
  G2, Romania (n=1,9,130) | 0 | 0 | 0
  G2, Taiwan (n=1,9,130) | 0 | 0 | 67
  G2, Turkey (n=1,9,130) | 1 | 0 | 4
  G2, Slovakia (n=1,9,130) | 0 | 0 | 0
  G2, Serbia (n=1,9,130) | 0 | 0 | 0
  G2, Sweden (n=1,9,130) | 0 | 0 | 0
  G2, Switzerland (n=1,9,130) | 0 | 0 | 0
  G2, Syria (n=1,9,130) | 0 | 0 | 0
  G2, United Arab Emirates (n=1,9,130) | 0 | 0 | 0
  G2, Venezuela (n=1,9,130) | 0 | 1 | 1
  G3, Argentina (n=2,18,147) | 0 | 1 | 3
  G3, Belgium (n=2,18,147) | 0 | 1 | 8
  G3, Chile (n=2,18,147) | 0 | 0 | 4
  G3, Egypt (n=2,18,147) | 0 | 0 | 0
  G3, Estonia (n=2,18,147) | 0 | 0 | 0
  G3, France (n=2,18,147) | 1 | 3 | 23
  G3, Germany (n=2,18,147) | 0 | 1 | 6
  G3, Greece (n=2,18,147) | 0 | 1 | 7
  G3, Italy (n=2,18,147) | 1 | 4 | 29
  G3, Kuwait (n=2,18,147) | 0 | 0 | 0
  G3, Latvia (n=2,18,147) | 0 | 0 | 0
  G3, Lebanon (n=2,18,147) | 0 | 1 | 0
  G3, Lithuania (n=2,18,147) | 0 | 2 | 18
  G3, Macedonia (n=2,18,147) | 0 | 0 | 1
  G3, Mexico (n=2,18,147) | 0 | 0 | 2
  G3, Oman (n=2,18,147) | 0 | 0 | 0
  G3, Pakistan (n=2,18,147) | 0 | 0 | 25
  G3, Peru (n=2,18,147) | 0 | 0 | 0
  G3, Portugal (n=2,18,147) | 0 | 3 | 15
  G3, Qatar (n=2,18,147) | 0 | 0 | 0
  G3, Romania (n=2,18,147) | 0 | 0 | 0
  G3, Taiwan (n=2,18,147) | 0 | 0 | 1
  G3, Turkey (n=2,18,147) | 0 | 0 | 1
  G3, Slovakia (n=2,18,147) | 0 | 1 | 2
  G3, Serbia (n=2,18,147) | 0 | 0 | 0
  G3, Sweden (n=2,18,147) | 0 | 0 | 1
  G3, Switzerland (n=2,18,147) | 0 | 0 | 0
  G3, Syria (n=2,18,147) | 0 | 0 | 0
  G3, United Arab Emirates (n=2,18,147) | 0 | 0 | 1
  G3, Venezuela (n=2,18,147) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p = 0.0097, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p < 0.0001, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.9778, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

84. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by HCV RNA Genotype and Country: Treatment-Experienced (Table 2 of 2 [G4, Other, Total])
Description: as for outcome 77
Time Frame: Study Visit 1
Population: as for outcome 64
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 18 | 270 | 1411
participants
  G4, Argentina (n=1,22,91) | 0 | 0 | 1
  G4, Belgium (n=1,22,91) | 0 | 3 | 8
  G4, Chile (n=1,22,91) | 0 | 0 | 1
  G4, Egypt (n=1,22,91) | 0 | 5 | 36
  G4, Estonia (n=1,22,91) | 0 | 0 | 0
  G4, France (n=1,22,91) | 0 | 7 | 15
  G4, Germany (n=1,22,91) | 0 | 1 | 2
  G4, Greece (n=1,22,91) | 1 | 1 | 2
  G4, Italy (n=1,22,91) | 0 | 2 | 12
  G4, Kuwait (n=1,22,91) | 0 | 0 | 0
  G4, Latvia (n=1,22,91) | 0 | 0 | 0
  G4, Lebanon (n=1,22,91) | 0 | 0 | 5
  G4, Lithuania (n=1,22,91) | 0 | 0 | 0
  G4, Macedonia (n=1,22,91) | 0 | 0 | 0
  G4, Mexico (n=1,22,91) | 0 | 0 | 0
  G4, Oman (n=1,22,91) | 0 | 0 | 0
  G4, Pakistan (n=1,22,91) | 0 | 0 | 0
  G4, Peru (n=1,22,91) | 0 | 0 | 0
  G4, Portugal (n=1,22,91) | 0 | 2 | 8
  G4, Qatar (n=1,22,91) | 0 | 0 | 0
  G4, Romania (n=1,22,91) | 0 | 0 | 0
  G4, Taiwan (n=1,22,91) | 0 | 0 | 0
  G4, Turkey (n=1,22,91) | 0 | 0 | 1
  G4, Slovakia (n=1,22,91) | 0 | 0 | 0
  G4, Serbia (n=1,22,91) | 0 | 0 | 0
  G4, Sweden (n=1,22,91) | 0 | 0 | 0
  G4, Switzerland (n=1,22,91) | 0 | 0 | 0
  G4, Syria (n=1,22,91) | 0 | 0 | 0
  G4, United Arab Emirates (n=1,22,91) | 0 | 1 | 0
  G4, Venezuela (n=1,22,91) | 0 | 0 | 0
  Other, Argentina (n=0,7,34) | 0 | 0 | 0
  Other, Belgium (n=0,7,34) | 0 | 3 | 2
  Other, Chile (n=0,7,34) | 0 | 0 | 0
  Other, Egypt (n=0,7,34) | 0 | 0 | 0
  Other, Estonia (n=0,7,34) | 0 | 0 | 0
  Other, France (n=0,7,34) | 0 | 0 | 5
  Other, Germany (n=0,7,34) | 0 | 0 | 0
  Other, Greece (n=0,7,34) | 0 | 0 | 0
  Other, Italy (n=0,7,34) | 0 | 0 | 1
  Other, Kuwait (n=0,7,34) | 0 | 0 | 0
  Other, Latvia (n=0,7,34) | 0 | 0 | 0
  Other, Lebanon (n=0,7,34) | 0 | 0 | 0
  Other, Lithuania (n=0,7,34) | 0 | 0 | 0
  Other, Macedonia (n=0,7,34) | 0 | 0 | 0
  Other, Mexico (n=0,7,34) | 0 | 0 | 0
  Other, Oman (n=0,7,34) | 0 | 1 | 0
  Other, Pakistan (n=0,7,34) | 0 | 0 | 2
  Other, Peru (n=0,7,34) | 0 | 0 | 2
  Other, Portugal (n=0,7,34) | 0 | 0 | 1
  Other, Qatar (n=0,7,34) | 0 | 0 | 0
  Other, Romania (n=0,7,34) | 0 | 0 | 0
  Other, Taiwan (n=0,7,34) | 0 | 0 | 3
  Other, Turkey (n=0,7,34) | 0 | 3 | 17
  Other, Slovakia (n=0,7,34) | 0 | 0 | 0
  Other, Serbia (n=0,7,34) | 0 | 0 | 0
  Other, Sweden (n=0,7,34) | 0 | 0 | 0
  Other, Switzerland (n=0,7,34) | 0 | 0 | 0
  Other, Syria (n=0,7,34) | 0 | 0 | 0
  Other, United Arab Emirates (n=0,7,34) | 0 | 0 | 0
  Other, Venezuela (n=0,7,34) | 0 | 0 | 1
  Total, Argentina (n=18,270,1411) | 0 | 7 | 11
  Total, Belgium (n=18,270,1411) | 0 | 13 | 72
  Total, Chile (n=18,270,1411) | 0 | 4 | 27
  Total, Egypt (n=18,270,1411) | 0 | 5 | 37
  Total, Estonia (n=18,270,1411) | 0 | 0 | 7
  Total, France (n=18,270,1411) | 5 | 62 | 217
  Total, Germany (n=18,270,1411) | 0 | 21 | 58
  Total, Greece (n=18,270,1411) | 1 | 8 | 33
  Total, Italy (n=18,270,1411) | 5 | 49 | 235
  Total, Kuwait (n=18,270,1411) | 0 | 0 | 0
  Total, Latvia (n=18,270,1411) | 0 | 11 | 53
  Total, Lebanon (n=18,270,1411) | 0 | 3 | 23
  Total, Lithuania (n=18,270,1411) | 3 | 13 | 67
  Total, Macedonia (n=18,270,1411) | 0 | 0 | 1
  Total, Mexico (n=18,270,1411) | 0 | 3 | 29
  Total, Oman (n=18,270,1411) | 0 | 1 | 6
  Total, Pakistan (n=18,270,1411) | 0 | 0 | 31
  Total, Peru (n=18,270,1411) | 0 | 2 | 30
  Total, Portugal (n=18,270,1411) | 1 | 16 | 50
  Total, Qatar (n=18,270,1411) | 0 | 2 | 5
  Total, Romania (n=18,270,1411) | 1 | 20 | 107
  Total, Taiwan (n=18,270,1411) | 0 | 0 | 163
  Total, Turkey (n=18,270,1411) | 1 | 19 | 101
  Total, Slovakia (n=18,270,1411) | 0 | 4 | 16
  Total, Serbia (n=18,270,1411) | 0 | 0 | 0
  Total, Sweden (n=18,270,1411) | 0 | 0 | 4
  Total, Switzerland (n=18,270,1411) | 0 | 1 | 7
  Total, Syria (n=18,270,1411) | 0 | 0 | 0
  Total, United Arab Emirates (n=18,270,1411) | 0 | 2 | 6
  Total, Venezuela (n=18,270,1411) | 1 | 4 | 15
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.0151, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 2: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Other genotypes; Test type: Superiority or Other; p = 0.1052, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest
Statistical Analysis 3: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p = 0.0007, Chi-squared — Pearson Chi-Square Test for differences in the ITPA distribution between the nominal categories of interest

85. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Type of Virological Response in the First 12 Weeks of Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and virological response to prior treatment were obtained from medical records. Virological response types within the first 12 weeks of treatment included rapid virological response (RVR), complete early virological response (cEVR), and partial early virological response (pEVR). RVR was defined as an undetectable HCV RNA level within the first 4 weeks, cEVR as an undetectable level within the first 12 weeks, and pEVR as a 2-log drop from Baseline to 12 weeks. Undetectable viral loads include those below the lower limit of detection (LLOD) for the assay performed, which may vary from site to site. Response categories were mutually exclusive, meaning participants could only achieve cEVR/pEVR in the absence of RVR. Participants achieving neither RVR nor cEVR/pEVR were recorded as 'none of the above.'
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 346 | 705 | 227
participants
  G1, RVR | 41 | 37 | 13
  G1, cEVR | 117 | 199 | 44
  G1, pEVR | 27 | 147 | 62
  G1, None of above | 41 | 184 | 73
  G2, RVR | 46 | 13 | 2
  G2, cEVR | 9 | 7 | 4
  G2, pEVR | 2 | 2 | 1
  G2, None of above | 4 | 5 | 1
  G3, RVR | 20 | 10 | 5
  G3, cEVR | 10 | 27 | 6
  G3, pEVR | 2 | 7 | 0
  G3, None of above | 7 | 13 | 1
  G4, RVR | 11 | 6 | 2
  G4, cEVR | 4 | 17 | 4
  G4, pEVR | 0 | 11 | 5
  G4, None of above | 5 | 20 | 4
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0012, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.1717, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0253, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

86. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Type of Virological Response in the First 12 Weeks of Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and virological response to prior treatment were obtained from medical records. Virological response types within the first 12 weeks of treatment included RVR, cEVR, and pEVR. RVR was defined as an undetectable HCV RNA level within the first 4 weeks, cEVR as an undetectable level within the first 12 weeks, and pEVR as a 2-log drop from Baseline to 12 weeks. Undetectable viral loads include those below the LLOD for the assay performed, which may vary from site to site. Response categories were mutually exclusive, meaning participants could only achieve cEVR/pEVR in the absence of RVR. Participants achieving neither RVR nor cEVR/pEVR were recorded as 'none of the above.'
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 630 | 556 | 92
participants
  G1, RVR | 59 | 23 | 9
  G1, cEVR | 205 | 140 | 15
  G1, pEVR | 88 | 128 | 20
  G1, None of above | 92 | 170 | 36
  G2, RVR | 50 | 9 | 2
  G2, cEVR | 11 | 6 | 3
  G2, pEVR | 3 | 2 | 0
  G2, None of above | 7 | 2 | 1
  G3, RVR | 23 | 9 | 3
  G3, cEVR | 23 | 18 | 2
  G3, pEVR | 3 | 6 | 0
  G3, None of above | 10 | 10 | 1
  G4, RVR | 17 | 2 | 0
  G4, cEVR | 13 | 12 | 0
  G4, pEVR | 11 | 5 | 0
  G4, None of above | 15 | 14 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0330, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.1595, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.0412, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

87. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Type of Virological Response at End of Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and virological response to prior treatment were obtained from medical records. Virological response types at the end of treatment included undetectable and detectable HCV RNA level. Undetectable viral loads include those below the LLOD for the assay performed, which may vary from site to site.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 412 | 773 | 244
participants
  G1, Undetectable | 194 | 297 | 79
  G1, Detectable | 62 | 313 | 125
  G2, Undetectable | 73 | 24 | 8
  G2, Detectable | 5 | 9 | 1
  G3, Undetectable | 43 | 48 | 15
  G3, Detectable | 11 | 21 | 1
  G4, Undetectable | 16 | 29 | 8
  G4, Detectable | 8 | 32 | 7
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0421, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.7658, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.2950, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

88. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Type of Virological Response at End of Treatment and HCV RNA Genotype
Description: as for outcome 87
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 718 | 614 | 97
participants
  G1, Undetectable | 326 | 222 | 22
  G1, Detectable | 161 | 279 | 60
  G2, Undetectable | 82 | 18 | 5
  G2, Detectable | 8 | 6 | 1
  G3, Undetectable | 59 | 39 | 8
  G3, Detectable | 18 | 14 | 1
  G4, Undetectable | 37 | 16 | 0
  G4, Detectable | 27 | 20 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0827, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.7817, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.1986, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three IL28B genotype categories

89. Secondary Outcome: Number of Participants With IL28B Genotype rs12979860 by Overall Virological Response Type and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and virological response to prior treatment were obtained from medical records. Overall virological response types included sustained virological response (SVR), relapse, and breakthrough. SVR was defined as undetectable HCV RNA level at 24 weeks post-treatment, relapse as an undetectable level at end of treatment with a detectable level at the last post-treatment measurement, and breakthrough as an undetectable level at 1 or more treatment measurements with a detectable level at end of treatment. Undetectable viral loads include those below the LLOD for the assay performed, which may vary from site to site. Response categories were mutually exclusive. Participants with detectable HCV RNA level at 12 or more treatment measurements and who did not meet SVR criteria were considered nonresponders, and those with insufficient treatment response data were recorded as 'none of the above.'
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs12979860 CC | Experienced: IL28B rs12979860 TC | Experienced: IL28B rs12979860 TT
Number analyzed (Participants) | 474 | 891 | 290
participants
  G1, SVR | 99 | 72 | 14
  G1, Relapse | 95 | 221 | 63
  G1, Breakthrough | 20 | 63 | 24
  G1, Nonresponder | 43 | 253 | 92
  G1, None of above | 37 | 94 | 45
  G2, SVR | 61 | 11 | 3
  G2, Relapse | 15 | 13 | 4
  G2, Breakthrough | 1 | 2 | 0
  G2, Nonresponder | 2 | 7 | 1
  G2, None of above | 13 | 5 | 3
  G3, SVR | 23 | 19 | 4
  G3, Relapse | 19 | 24 | 8
  G3, Breakthrough | 1 | 5 | 1
  G3, Nonresponder | 10 | 15 | 1
  G3, None of above | 9 | 21 | 6
  G4, SVR | 8 | 17 | 4
  G4, Relapse | 6 | 13 | 3
  G4, Breakthrough | 4 | 8 | 1
  G4, Nonresponder | 4 | 21 | 5
  G4, None of above | 4 | 7 | 8
Statistical Analysis 1: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G2; Test type: Superiority or Other; p = 0.0002, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G3; Test type: Superiority or Other; p = 0.0394, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs12979860 CC vs Experienced: IL28B rs12979860 TC vs Experienced: IL28B rs12979860 TT; G4; Test type: Superiority or Other; p = 0.0493, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

90. Secondary Outcome: Number of Participants With IL28B Genotype rs8099917 by Overall Virological Response Type and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine IL28B genotype. HCV RNA genotype and virological response to prior treatment were obtained from medical records. Overall virological response types included SVR, relapse, and breakthrough. SVR was defined as undetectable HCV RNA level at 24 weeks post-treatment, relapse as an undetectable level at end of treatment with a detectable level at the last post-treatment measurement, and breakthrough as an undetectable level at 1 or more treatment measurements with a detectable level at end of treatment. Undetectable viral loads include those below the LLOD for the assay performed, which may vary from site to site. Response categories were mutually exclusive. Participants with detectable HCV RNA level at 12 or more treatment measurements and who did not meet SVR criteria were considered nonresponders, and those with insufficient treatment response data were recorded as 'none of the above.'
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: IL28B rs8099917 TT | Experienced: IL28B rs8099917 TG | Experienced: IL28B rs8099917 GG
Number analyzed (Participants) | 831 | 709 | 115
participants
  G1, SVR | 133 | 46 | 6
  G1, Relapse | 194 | 168 | 17
  G1, Breakthrough | 42 | 49 | 16
  G1, Nonresponder | 115 | 232 | 41
  G1, None of above | 78 | 79 | 19
  G2, SVR | 64 | 9 | 2
  G2, Relapse | 20 | 10 | 2
  G2, Breakthrough | 2 | 1 | 0
  G2, Nonresponder | 4 | 5 | 1
  G2, None of above | 17 | 2 | 2
  G3, SVR | 29 | 15 | 2
  G3, Relapse | 27 | 21 | 3
  G3, Breakthrough | 3 | 3 | 1
  G3, Nonresponder | 14 | 12 | 0
  G3, None of above | 19 | 14 | 3
  G4, SVR | 21 | 8 | 0
  G4, Relapse | 14 | 8 | 0
  G4, Breakthrough | 8 | 5 | 0
  G4, Nonresponder | 16 | 14 | 0
  G4, None of above | 11 | 8 | 0
Statistical Analysis 1: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G1; Test type: Superiority or Other; p < 0.0001, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 2: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G2; Test type: Superiority or Other; p = 0.0196, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 3: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G3; Test type: Superiority or Other; p = 0.3268, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories
Statistical Analysis 4: Comparison: Experienced: IL28B rs8099917 TT vs Experienced: IL28B rs8099917 TG vs Experienced: IL28B rs8099917 GG; G4; Test type: Superiority or Other; p = 0.1667, Jonckheere-Terpstra Test — Jonckheere-Terpstra Test for a trend of an ordinal variable across the three IL28B genotype categories

91. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by Incidence of Hemoglobin Drop During Prior Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype. HCV RNA genotype and hematology data were obtained from medical records. Participants with a history of a hemoglobin level less than 10 grams per deciliter (g/dL) or a drop of more than 3 g/dL at any time during prior treatment for CHC were recorded as 'yes' for this finding.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs1127354 AA | Experienced: ITPA rs1127354 CA | Experienced: ITPA rs1127354 CC
Number analyzed (Participants) | 14 | 185 | 1112
participants
  G1, Yes (n=9,133,810) | 2 | 35 | 322
  G1, No (n=9,133,810) | 7 | 98 | 488
  G2, Yes (n=3,27,89) | 2 | 9 | 42
  G2, No (n=3,27,89) | 1 | 18 | 47
  G3, Yes (n=2,20,105) | 0 | 1 | 33
  G3, No (n=2,20,105) | 2 | 19 | 72
  G4, Yes (n=0,2,85) | 0 | 0 | 36
  G4, No (n=0,2,85) | 0 | 2 | 49
  Other, Yes (n=0,3,23) | 0 | 1 | 15
  Other, No (n=0,3,23) | 0 | 2 | 8
  Total, Yes (n=14,185,1112) | 4 | 46 | 448
  Total, No (n=14,185,1112) | 10 | 139 | 664
Statistical Analysis 1: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p = 0.0021, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 2: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.5319, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 3: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.0114, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 4: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.2293, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 5: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.2857, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 6: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p = 0.0001, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories

92. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by Incidence of Hemoglobin Drop During Prior Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype. HCV RNA genotype and hematology data were obtained from medical records. Participants with a history of a hemoglobin level less than 10 g/dL or a drop of more than 3 g/dL at any time during prior treatment for CHC were recorded as 'yes' for this finding.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 13 | 205 | 1092
participants
  G1, Yes (n=10,159,783) | 1 | 49 | 309
  G1, No (n=10,159,783) | 9 | 110 | 474
  G2, Yes (n=0,8,110) | 0 | 1 | 52
  G2, No (n=0,8,110) | 0 | 7 | 58
  G3, Yes (n=2,14,111) | 0 | 3 | 31
  G3, No (n=2,14,111) | 2 | 11 | 80
  G4, Yes (n=1,19,67) | 0 | 3 | 33
  G4, No (n=1,19,67) | 1 | 16 | 34
  Other, Yes (n=0,5,21) | 0 | 2 | 14
  Other, No (n=0,5,21) | 0 | 3 | 7
  Total, Yes (n=13,205,1092) | 1 | 58 | 439
  Total, No (n=13,205,1092) | 12 | 147 | 653
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p = 0.0081, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 2: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p = 0.0563, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 3: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.3516, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 4: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.0064, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 5: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Other genotypes; Test type: Superiority or Other; p = 0.2707, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 6: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p < 0.0001, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories

93. Secondary Outcome: Number of Participants With ITPA Genotype rs1127354 by Erythropoietin Use During Prior Treatment and HCV RNA Genotype
Description: Participants underwent blood sampling at the Study Visit to determine ITPA genotype. HCV RNA genotype was obtained from medical records. Past medication use was obtained from medical records and/or participant interview at the Study Visit. Participants with a history of erythropoietin use during prior treatment for CHC were recorded as 'yes' for this finding.
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs1127354 AA | Experienced: ITPA rs1127354 CA | Experienced: ITPA rs1127354 CC
Number analyzed (Participants) | 15 | 225 | 1388
participants
  G1, Yes (n=10,162,1016) | 1 | 8 | 103
  G1, No (n=10,162,1016) | 9 | 154 | 913
  G2, Yes (n=3,30,105) | 0 | 4 | 14
  G2, No (n=3,30,105) | 3 | 26 | 91
  G3, Yes (n=2,24,137) | 0 | 0 | 4
  G3, No (n=2,24,137) | 2 | 24 | 133
  G4, Yes (n=0,5,106) | 0 | 1 | 18
  G4, No (n=0,5,106) | 0 | 4 | 88
  Other, Yes (n=0,4,24) | 0 | 0 | 3
  Other, No (n=0,4,24) | 0 | 4 | 21
  Total, Yes (n=15,225,1388) | 1 | 13 | 142
  Total, No (n=15,225,1388) | 14 | 212 | 1246
Statistical Analysis 1: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G1; Test type: Superiority or Other; p = 0.0634, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 2: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G2; Test type: Superiority or Other; p = 0.7176, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 3: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G3; Test type: Superiority or Other; p = 0.3944, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 4: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; G4; Test type: Superiority or Other; p = 0.8610, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 5: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Other genotypes; Test type: Superiority or Other; p = 0.4543, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 6: Comparison: Experienced: ITPA rs1127354 AA vs Experienced: ITPA rs1127354 CA vs Experienced: ITPA rs1127354 CC; Total genotypes; Test type: Superiority or Other; p = 0.0406, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories

94. Secondary Outcome: Number of Participants With ITPA Genotype rs7270101 by Erythropoietin Use During Prior Treatment and HCV RNA Genotype
Description: as for outcome 93
Time Frame: Study Visit 1
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Experienced: ITPA rs7270101 CC | Experienced: ITPA rs7270101 AC | Experienced: ITPA rs7270101 AA
Number analyzed (Participants) | 17 | 257 | 1354
participants
  G1, Yes (n=14,206,969) | 2 | 19 | 91
  G1, No (n=14,206,969) | 12 | 187 | 878
  G2, Yes (n=0,9,128) | 0 | 0 | 17
  G2, No (n=0,9,128) | 0 | 9 | 111
  G3, Yes (n=2,17,144) | 0 | 0 | 4
  G3, No (n=2,17,144) | 2 | 17 | 140
  G4, Yes (n=1,20,90) | 0 | 2 | 17
  G4, No (n=1,20,90) | 1 | 18 | 73
  Other, Yes (n=0,5,23) | 0 | 0 | 3
  Other, No (n=0,5,23) | 0 | 5 | 20
  Total, Yes (n=17,257,1354) | 2 | 21 | 132
  Total, No (n=17,257,1354) | 15 | 236 | 1222
Statistical Analysis 1: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G1; Test type: Superiority or Other; p = 0.8234, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 2: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G2; Test type: Superiority or Other; p = 0.2427, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 3: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G3; Test type: Superiority or Other; p = 0.4805, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 4: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; G4; Test type: Superiority or Other; p = 0.2901, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 5: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Other genotypes; Test type: Superiority or Other; p = 0.3927, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories
Statistical Analysis 6: Comparison: Experienced: ITPA rs7270101 CC vs Experienced: ITPA rs7270101 AC vs Experienced: ITPA rs7270101 AA; Total genotypes; Test type: Superiority or Other; p = 0.5769, Cochran-Armitage Trend Test — Cochran-Armitage Trend Test for a trend in binomial proportions across the three ITPA genotype categories

ADVERSE EVENTS:
Time Frame: Study Visit 1
Description: Safety Population: Of the 4766 participants enrolled, 33 did not undergo blood sampling and were thus excluded from the safety analysis. Only serious adverse events caused by a protocol-mandated intervention during the single study visit (Study Visit 1) were assessed; nonserious adverse events were not documented in the course of the study.
Arm/Group | Participants With CHC
Serious Adverse Events (participants affected / at risk) | 0/4733
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.